

# **Clinical Trial Protocol**

| | Document Number: | c39145241-04 |
|---|---|---|
| EudraCT No. | 2022-001091-34 | |
| BI Trial No. | 1305-0014 (FIBRONEER <sup>TM</sup> – IPF) | |
| BI Investigational<br>Medicinal Product | BI 1015550 | |
| Title | A double blind, randomized, placeb<br>the efficacy and safety of BI 101555<br>patients with Idiopathic Pulmonary | 50 over at least 52 weeks in |
| Lay Title | A study to find out whether BI 1015 in people with Idiopathic Pulmonary | |
| Clinical Phase | Phase III | |
| Clinical Trial Leader | Tel: Fax: | |
| Investigator | Phone: Fax | x: |
| Current Version and<br>Date | Version 4.0, 20 Sep 2023 | |
| Original Protocol<br>Date | Version 1.0, 13 Jun 2022 | |
| | Dronwigtory confidential information | <u> </u> |

Proprietary confidential information.

© 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Company name | Boehringer Ingelheim |
|---|---|
| Original Protocol date | 13 Jun 2022 |
| Latest revision date | 20 Sep 2023 |
| BI Trial No. | 1305-0014 |
| Title of trial | A double blind, randomized, placebo-controlled trial evaluating the efficacy and safety of BI 1015550 over at least 52 weeks in patients with Idiopathic Pulmonary Fibrosis (IPF) |
| Investigator | Phone: Fax: |
| Trial sites | Multi-centre trial conducted in approximately 400 sites and in |
| | 45 countries |
| Clinical phase | Phase III |
| Trial rationale Benefit-risk assessment | The purpose of this trial is to evaluate the efficacy, safety, and tolerability of BI 1015550 9 mg bid and 18 mg bid compared to placebo in patients with IPF in addition to patient's standard of care over the course of at least 52 weeks. New treatments with better tolerability are needed for patients with IPF to further reduce the decline in lung function and improve quality of life. Based on its anti-inflammatory and antifibrotic properties and the preliminary clinical evidence described, BI 1015550 may provide an additional treatment option to patients with pulmonary fibrosis irrespective of concomitant treatment with standard of care. Patients with IPF who receive treatment with BI 1015550 have the |
| and ethical<br>considerations | potential benefit of slowing lung function decline, improving symptoms, and improving quality of life over a long-term period. |
| | The toxicology data support administration of BI 1015550 to women and men in the planned Phase III clinical trials in patients with IPF and other forms of progressive pulmonary fibrosis irrespective of background antifibrotic treatment, except for women who are pregnant or breastfeeding. |
| | Data from the Phase II trial 1305-0013 in patients with IPF indicated a beneficial treatment effect of 18 mg BI 1015550 bid, with the preservation of Forced Vital Capacity (FVC) over 12 weeks together with an acceptable safety and tolerability profile supporting further investigation in Phase III clinical trials as a treatment for IPF and other forms of progressive pulmonary fibrosis. |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Trial objectives | The primary objective is to demonstrate a reduction in lung function decline as measured by the change from baseline in FVC for BI 1015550 when compared to placebo in patients with IPF. |
|---|---|
| | The main secondary objective of the trial is to demonstrate BI 1015550's ability in reducing the occurrence of clinically meaningful events such as acute IPF exacerbation, hospitalization for respiratory cause or death over the duration of the trial when compared to placebo in patients with IPF. An additional secondary objective of the trial is to show an effect of BI 1015550 on symptoms and lung function. |
| Trial endpoints | The primary endpoint is the absolute change from baseline in FVC [mL] at Week 52. |
| | The key secondary endpoint in this trial is time to the first occurrence of any of the components of the composite endpoint:time to first acute IPF exacerbation, first hospitalization for respiratory cause, or death (whichever occurs first) over the duration of the trial. |
| Trial design | A multi-centre, multi-national, prospective, randomized, placebo-controlled, double blind clinical trial to investigate the efficacy and safety of BI 1015550 at a dose of 9 mg bid and 18 mg bid in patients with IPF over at least 52 weeks. |
| Total number of | Approximately 963 patients |
| patients randomized | 11 , 1 |
| Number of patients per treatment group | Approximately 321 patients in each active treatment group and in |
| | the placebo group. |
| Diagnosis,<br>main inclusion and<br>exclusion criteria | <ul> <li>Inclusion criteria:</li> <li>Patients ≥40 years old at the time of signed consent</li> <li>IPF diagnosis based on 2022 ATS/ERS/JRS/ALAT Guidelines [P22-03204]</li> </ul> |
| | • FVC ≥45% of predicted normal |
| | <ul> <li>DLCO ≥25% of predicted normal corrected for hemoglobin (Hb)</li> <li>On stable treatment with nintedanib or pirfenidone for at least 12 weeks or not on treatment with either nintedanib or pirfenidone for at least 8 weeks</li> <li>Exclusion criteria:</li> </ul> |
| | • Prebronchodilator FEV1/FVC < 0.7 |
| | Acute IPF exacerbation within 3 months and/or during the screening period |
| | • Treated with immunomodulatory medications (other than oral corticosteroids) or prednisone >15 mg/day or equivalent for respiratory or pulmonary reasons |
| | Active, unstable or uncontrolled vasculitis within 8 weeks |
| | Any suicidal behaviour in the past 2 years |
| | • Any suicidal ideation of type 4 or 5 on the C-SSRS in the past 3 months |
| Trial intervention and test product | BI 1015550 |

# **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Dose and mode of | 9 mg bid, oral |
|---|---|
| administration | - |
| | 18 mg bid, oral |
| Comparator product | Placebo |
| Dose and mode of | Matching, oral |
| administration | 1.1.1.1.20 |
| <b>Duration of treatment</b> | At least 52 weeks and up to approximately 130 weeks |
| Statistical methods | This trial's primary objective is to demonstrate the ability of |
| | BI 1015550 to reduce lung function decline based on FVC between |
| | baseline and at Week 52 when compared to placebo. |
| | Primary analysis for primary endpoint will be restricted maximum likelihood estimation based on a mixed-effect model for repeated measures (MMRM) analysis to compare change from baseline in FVC at Week 52 between treatment groups. This model will include discrete fixed effects for treatment at each visit, baseline intake of antifibrotic treatment at each visit, and continuous fixed effects for baseline FVC value at each visit. |
| | An interim analysis assessing futility of the 9 mg dose vs. placebo will be conducted after approximately 300 patients have reached the Week 12 primary endpoint assessment. If the 9 mg dose is considered futile, the patients will be re-assigned to the 18 mg dose. |
| | Once the last randomized patient completes the Week-52 assessment, the main analysis of the trial will be carried out by the sponsor, who will be unblinded to assess the benefit-risk of the two doses of BI 1015550 compared with placebo. Patients will remain on their randomized blinded treatment until the sponsor has reviewed the efficacy and safety data from the main analysis and communicated the end of the trial. Once this trial ends, a final analysis based on all data will be carried out. |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **FLOW CHART**

| Trial Periods | Screening | Treatment Period A | | | | | | | | | Treatment Period | | Follow<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 <sup>1</sup> | Every<br>12 weeks <sup>1</sup> | EOT <sup>2</sup> | EOS <sup>17</sup> |
| Week | Up<br>to -8 weeks<br>to -1 week* | 1 | 2 | 6 | 12 | 18 | 26 | 36 | 44 | 52 | | | |
| Day | to 1 week | 1 | 15 | 43 | 85 | 127 | 183 | 253 | 309 | 365 | | | EOT +7d |
| Time window (days) | | | ±3d | ±7d | ±7d | ±7d | ±7d | ±7d | ±7d | ±7d | ±14d | | +3d |
| Informed consent | X | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Review of | X | X | | | | | | | | | | | |
| eligibility criteria | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | |
| Smoking Status | X | | | | | | | | | | | | |
| L-PF | 71 | X | | | X | | X | X | X | X | X | X | |
| (symptoms/impact) <sup>3</sup> | | 21 | | | 21 | | 21 | 21 | 21 | 21 | 21 | 21 | |
| EQ-5D <sup>3</sup> | | X | | X | X | X | X | X | X | X | X | X | |
| HADS <sup>3</sup> | X | X | | | X | - 1 | X | X | X | X | X | 11 | X |
| PGIS <sup>3</sup> | Λ | X | | | X | | X | X | X | X | X | X | Λ |
| | v | | v | v | | v | X | X | | | | | v |
| C-SSRS <sup>4</sup> | X<br>X | X | X | X | X | X | X | X | X | X | X<br>X | X | X<br>X |
| Physical examination | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | 37 | | | | | | | | | | | | |
| Height | X | 7.7 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 |
| Weight | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SpO2 | | X | | | X | | X | | | X | | X | |
| 12-lead ECG | X | | | | X | | | | | X | | X | |
| Chest HRCT | X | | | | | | | | | | | | |
| central Review <sup>6</sup> | | | | | | | | | | | | | |
| Spirometry <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Optional home | | X | X | X | | X | | X | X | | X | | |
| spirometry <sup>8</sup> | | | | | | | | | | | | | |
| DLCO | X | X | | | X | | X | | | X | | X | |
| Laboratory test <sup>9</sup> | X | X | | X | X | | X | X | X | X | X | X | X |
| Vasculitis | | X | | | | | | | | X | | | |
| biomarkers | | | | | | | | | | | | | |
| storage <sup>10</sup> | | | | | | | | | | | | | |
| Pregnancy test <sup>11</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Infection testing <sup>12</sup> | X | | | | | | | | | X | | X | |
| PK Sampling <sup>13</sup> | | | X | X | X | | X | | | | | | |
| ILD biomarkers | | X | | X | X | | X | | | X | | X14 | |
| sampling | | | | | | | | | | | | | |
| DNA Banking | | X | | | | | | | | | | | |
| (optional) <sup>15</sup> | | | | | | | | | | | | | |
| Serum/Plasma<br>Banking | | X | | | X | | X | | | X | | | |
| (optional) <sup>15</sup> | | | | | | | | | | | | | |
| Health Care resource Utilization | | X | X | X | X | X | X | X | X | X | X | X | |
| All AEs/SAEs/ | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AESIs <sup>16</sup> Concomitant | X | X | X | X | X | X | X | X | X | X | X | X | X |
| therapy | ** | | | | | | | | | | | 21 | |
| Dispense trial drug | | X | | X | X | X | X | X | X | X | X<br>X | | |
| IRT | X | X | | X | X | X | X | X | X | X | X | X | 1 |
| Call/Notification | | | | | | | | | | | <u> </u> | | |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Trial Periods | Screening | | Treatment Period A | | | | | | | Treatmen | Follow | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | В | 3 | up |
| Administer trial | | X | X | X | X | X | X | X | X | X | X | X | |
| drugs | | | | | | | | | | | | | |
| Return trial drug | | | X | X | X | X | X | X | X | X | X | X | |
| Compliance check | | | X | X | X | X | X | X | X | X | X | X | |
| Completion of | | | | | | | | | | | | $X^{17}$ | X |
| patient participation | | | | | | | | | | | | | |
| Vital status data <sup>18</sup> | | | | | | | | | | X | | X | |

- Screening may be extended up to 12 weeks to account for possible missing eligibility results, administrative, or organisational reason.
- (<sup>1</sup>) Following completion of V10 patients will continue to have study visits every 12 weeks until the start of EoT visits is announced. The global study will be completed after all patients have performed the EoT visit and the EoS visit (if not continuing in the separate extension trial).
- (<sup>2</sup>) In case of premature discontinuation of trial medication, the EOT visit should only be done if the discontinuation is permanent, and a Follow-up (FU) visit is to be performed 7 days (+3 days) after end of treatment. If a patient discontinued the trial medication more than a week prior to the EOT visit, this FU visit is not required. A scheduled visit may be missed if EOT or FU visit occurs within 4 weeks prior to scheduled visits. After the premature EOT, every effort should be made to collect data until the end of the trial.
- $(^{3})$ Patient-reported outcomes collected either on paper questionnaires or as ePRO, at home within 3 days before the site visit or at the site visit. At the latest, the patients' questionnaires must be completed prior to the pulmonary function tests.
- (<sup>4</sup>) At Visit 1, the C-SSRS version to be used is the "screening/baseline" one. At all other visits, the version of C-SSRS to be used is the version "since last visit".
- Vital signs will be taken as one measurement at predose.
- (6)Send chest HRCT not older than 12 months for central review. If the patient does not have a HRCT within 12 months of Visit 1 or the available HRCT scan fails to meet the required image acquisition specification, a new HRCT can be performed and submitted provided the patient meets all other inclusion and no exclusion criteria. To perform a HRCT within the trial, all local regulatory requirements to perform an HRCT have to be met. In Germany, no HRCT will be performed as trial procedure; only historical HRCT will be submitted.
- $(^{7})$ Order of lung function measurements: 1. FVC followed by patient's rest; 2. DLCO: Two DLCO measurements will be performed approximately at the same time of the day, at least within the same half-day (morning vs. afternoon, reference time at Visit 2).
- (8)Assisted home spirometry will be offered at selected centres where every patient should have a training and measurement with the device ideally at Visits 2 or 3. If the requirement to use the iSpiro appears later in the trial, then this timepoint can be shifted. Remote measurement can be performed as per investigator's judgement but should not replace the on-site FVC measurement.
- $(^{9})$ Safety laboratory tests will be performed predose. This includes blood and urine collection. Of note, in case of a suspected vasculitis event, additional blood sampling is required. For details please see Section 5.2.3.
- Additional blood sample to be taken for storage and analysis in case of vasculitis adverse event during the trial.
- (11)Women of childbearing potential only. Serum pregnancy test to be performed at V1; urine dipstick pregnancy test to be performed at V2 and following visits (if positive, urine dipstick test to be followed by serum test for confirmation). More frequent pregnancy testing may be done if required.
- Infection testing includes HBV, HCV, HIV, and tuberculosis (Section <u>5.2.3.2</u>)
- $(^{13})$ PK samples to analyse BI 1015550 will be collected predose (before drug administration).
- (14)Only drawn if EOT is performed at 52 weeks (study completion phase).
- Collection of biobanking samples (plasma, serum, DNA) is optional and is not a prerequisite for participation in the trial. Only for patients who signed a separate informed consent. DNA sample will be taken at Visit 2 preferably or at any subsequent visit until EOT.
- Includes assessment of exacerbations, hospitalisations for respiratory cause, vasculitis, and diarrhoea
- Patients may be eligible to enter an extension trial if they complete this study on blinded treatment and meet the eligibility criteria for the extension trial. For patients who complete all study visits and roll over to extension trial, end of study is EOT. A follow-up visit (EOS) is only required for those who do not roll-over in the separate extension trial (or could not roll-over within a week of EOT visit) and if the last drug intake was less than 7 days before the EOT visit.
- $(^{18})$ Patients who discontinue trial treatment prematurely and have agreed to be contacted, should be called at least at the end of the 12-month observation period (52 weeks) and at the end of their scheduled trial participation to obtain their vital status information.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# TABLE OF CONTENTS

| TITLE | PAGE | I |
|---|---|---|
| CLINIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| <b>FLOW</b> | CHART | 5 |
| TABLE | OF CONTENTS | 7 |
| | VIATIONS AND DEFINITIONS | |
| 1. | INTRODUCTION. | |
| 1.1 | MEDICAL BACKGROUND. | |
| 1.1 | DRUG PROFILE | |
| 1.3 | RATIONALE FOR PERFORMING THE TRIAL | |
| 1.3 | BENEFIT - RISK ASSESSMENT | |
| 1.4.1 | Benefits | |
| 1.4.2 | Risks | |
| 1.4.3 | Discussion | |
| 2. | TRIAL OBJECTIVES AND ENDPOINTS | |
| 2.1 | MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS | |
| 2.1.1 | Main objectives | |
| 2.1.2 | Primary endpoint | |
| 2.1.3 | Key Secondary endpoint | |
| 2.1.4 | Secondary endpoints | |
| 3. | DESCRIPTION OF DESIGN AND TRIAL POPULATION | 27 |
| 3.1 | OVERALL TRIAL DESIGN | 27 |
| 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF | |
| | CONTROL GROUP(S) | |
| 3.3 | SELECTION OF TRIAL POPULATION | |
| 3.3.1 | Main diagnosis for trial entry | |
| 3.3.2 | Inclusion criteria | |
| 3.3.3 | Exclusion criteria | |
| 3.3.4 | Discontinuation of patients from treatment or assessments | |
| 3.3.4.1 | Discontinuation of trial treatment | |
| 3.3.4.2 | Withdrawal of consent to trial participation | |
| 3.3.4.3 | Discontinuation of the trial by the sponsor | 33 |
| 4. | TREATMENTS | |
| 4.1 | INVESTIGATIONAL TREATMENTS | |
| 4.1.1 | Identity of the Investigational Medicinal Products | |
| 4.1.2 | Selection of doses in the trial and dose modifications | |
| 4.1.3 | Method of assigning patients to treatment groups | |
| 4.1.4 | Drug assignment and administration of doses for each patient | 38 |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 4.1.5 | Blinding and procedures for unblinding | .39 |
|---|---|---|
| 4.1.5.1 | Blinding | .39 |
| 4.1.5.2 | Unblinding and breaking the code | .40 |
| 4.1.6 | Packaging, labelling, and re-supply | .40 |
| 4.1.7 | Storage conditions | |
| 4.1.8 | Drug accountability | .41 |
| 4.2 | OTHER TREATMENTS, EMERGENCY PROCEDURES, | |
| | RESTRICTIONS | |
| 4.2.1 | Other treatments and emergency procedures | |
| 4.2.2 | Restrictions | |
| 4.2.2.1 | Restrictions regarding concomitant treatment | |
| 4.2.2.2 | Restrictions on diet and lifestyle | |
| 4.2.2.3 | Contraception requirements | |
| 4.3 | TREATMENT COMPLIANCE | |
| 5. | ASSESSMENTS | .45 |
| 5.1 | ASSESSMENT OF EFFICACY | .45 |
| 5.1.1 | FVC | .45 |
| 5.1.2 | Exacerbation of IPF | .46 |
| 5.1.3 | Time to death | .47 |
| 5.1.4 | Hospitalization due to respiratory cause | |
| 5.1.5 | Patient-Reported Outcome Questionnaires | |
| 5.1.5.1 | Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (L-PF) | |
| 5.1.5.2 | EuroQol 5-Dimensional quality of life Questionnaire (EQ-5D) | |
| 5.1.5.3 | Patient's Global Impression of Severity (PGIS) of Cough, Shortness of Breath and Fatigue | |
| 5.1.6 | DLCO | .49 |
| 5.2 | ASSESSMENT OF SAFETY | .50 |
| 5.2.1 | Physical examination | .50 |
| 5.2.2 | Vital signs | .50 |
| 5.2.3 | Safety laboratory parameters | .50 |
| 5.2.3.1 | Routine safety lab tests | |
| 5.2.3.2 | Infection serology | . 52 |
| 5.2.3.3 | Immunological vasculitis markers | . 53 |
| 5.2.4 | Electrocardiogram | |
| 5.2.5 | Other Safety parameters | |
| 5.2.5.1 | Suicidal risk (C-SSRS) | |
| 5.2.5.2 | Depression and anxiety | |
| 5.2.6 | Assessment of adverse events | |
| 5.2.6.1 | Definitions of AEs | |
| 5.2.6.1.1 | Adverse event | |
| 5.2.6.1.2 | Serious adverse event | |
| 5.2.6.1.3 | AEs considered "Always Serious" | |
| 5.2.6.1.4 | Adverse events of special interest | |
| 5.2.6.1.5 | Intensity (severity) of AEs | |
| 5.2.6.1.6 | Causal relationship of AEs. | . 58 |
| 5.2.6.2 | Adverse event collection and reporting | |
| 5.2.6.2.1 | AE Collection | .58 |


| Proprietary confidential | information © 2023 Bo | oehringer Ingelheim In | nternational GmbH ( | or one or more of its | affiliated companies |
|---|---|---|---|---|---|

| 5.2.6.2.2 | AE reporting to the sponsor and timelines | |
|---|---|---|
| 5.2.6.2.3<br>5.2.6.3 | Pregnancy Independent safety monitoring and adverse events with additional information | l |
| | collection | 60 |
| 5.3 | DRUG CONCENTRATION MEASUREMENTS AND | |
| <b>7</b> 0 1 | PHARMACOKINETICS | |
| 5.3.1 | Assessment of pharmacokinetics | |
| 5.3.2 | Methods of sample collection | 61 |
| 5.4 | ASSESSMENT OF BIOMARKERS | 61 |
| 5.4.1 | Pharmacodynamics biomarkers | |
| 5.4.1.1 | Methods and timing of sample collection | |
| 5.5 | BIOBANKING | |
| 5.5.1 | Methods and timing of sample collection | |
| 5.6 | OTHER ASSESSMENTS. | |
| 5.6.1 | Chest HRCT assessment | |
| 5.6.2 | Health care resource utilization (HCRU) | 63 |
| <b>5.7</b> | APPROPRIATENESS OF MEASUREMENTS | 63 |
| 6. | INVESTIGATIONAL PLAN | 64 |
| 6.1 | VISIT SCHEDULE | 64 |
| 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | |
| 6.2.1 | Screening period. | |
| 6.2.2 | Treatment periods | |
| 6.2.2.1 | Conduct of a regular site visit | 66 |
| 6.2.2.2 | Conduct of a fallback visit (remote/home visit) | 67 |
| 6.2.2.3 | End of treatment visit | 68 |
| 6.2.3 | Follow-up period and trial completion | 68 |
| 7. | STATISTICAL METHODS AND DETERMINATION OF SAMPLE | (0 |
| 7.1 | NULL AND ALTERNATIVE HYPOTHESES | |
| 7.1 | PLANNED ANALYSES. | |
| 7.2.1 | General considerations | |
| 7.2.2 | Handling of intercurrent events | |
| 7.2.3 | Primary objective analyses | |
| 7.2.3.1 | Sensitivity Analyses. | |
| 7.2.3.2 | Subgroup Analyses | 74 |
| 7.2.3.3 | Supplementary Analyses | 75 |
| 7.2.4 | Secondary objective analyses | 75 |
| 7.2.4.1 | Analysis of key secondary endpoint | |
| 7.2.4.2 | Analysis of other secondary endpoints | 75 |
| 7.2.5 | Further objective analyses. | |
| 7.2.6 | Safety analyses | |
| 7.2.7 | Other Analyses | |
| 7.2.7.1 | Pharmacokinetic Methods | |
| <b>7.2.8</b> | Interim analyses | |
| 7.3 | HANDLING OF MISSING DATA | 78 |


| Proprietary | y confidential | linformation | © 2023 Bo | ehringer l | Ingelheim | International | GmbH or | one or mor | e of its | affiliated | companies |
|---|---|---|---|---|---|---|---|---|---|---|---|

| 7.3.1 | Efficacy endpoints | |
|---|---|---|
| 7.3.2 | Safety endpoints | |
| 7.4 | RANDOMIZATION | |
| 7.5 | DETERMINATION OF SAMPLE SIZE | 80 |
| 8. | INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE | 85 |
| 8.1 | TRIAL APPROVAL, PATIENT INFORMATION, INFORMED | |
| 0.3 | CONSENT DATA QUALITY ASSURANCE | 85<br>00 |
| 8.2<br>8.3 | RECORDS | |
| 8.3.1 | Source documents | |
| 8.3.2 | Direct access to source data and documents | |
| 8.3.3 | Storage period of records | |
| 8.4 | EXPEDITED REPORTING OF ADVERSE EVENTS | |
| | STATEMENT OF CONFIDENTIALITY AND PATIENT PRIVACY | |
| 8.5 | | 88 |
| 8.5.1 | Collection, storage and future use of biological samples and | 00 |
| 0.6 | corresponding dataTRIAL MILESTONES. | |
| 8.6 | ADMINISTRATIVE STRUCTURE OF THE TRIAL | |
| 8.7 | | |
| 9. | REFERENCES | |
| 9.1 | PUBLISHED REFERENCES | 91 |
| 9.2 | UNPUBLISHED REFERENCES | 92 |
| 10. | APPENDICES | 93 |
| 10.1 | SPIROMETRY: BRONCHODILATOR WASHOUT | |
| | RECOMMENDATIONS | |
| 10.2 | PATIENT-REPORTED OUTCOMES | 94 |
| 10.2.1 | Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (LPF) | 0.4 |
| 10.2.2 | EuroQol 5-Dimensional quality of life Questionnaire (EQ-5D) | 94<br>107 |
| 10.2.2 | Hospital Anxiety and Depression Scale (HADS) | |
| 10.2.3 | | 10 / |
| 10.2.4 | Patient's Global Impression of Severity (PGIS) for Cough, Shortness of Breath, and Fatigue | 100 |
| 10.3 | COLUMBIA SUICIDAL SEVERITY RATING SCALE (C-SSRS) | 100<br>100 |
| 10.3 | | |
| | Visit 1 – Screening/baseline version | |
| 10.3.2 | C-SSRS – since last visit RESTRICTED MEDICATIONS TABLES | |
| 10.4 | | |
| 10.4.1 | Strong CYP3A4 inhibitors | |
| 10.4.2 | Equivalent doses of corticosteroids | |
| 10.4.3 | Restricted PDE inhibitors | |
| 10.5 | OPPORTUNISTIC INFECTIONS | |
| 10.6 | ELIGIBILITY CONFIRMATION OF IPF DIAGNOSIS | |
| 10.7 | TRIAL PARTICIPANT FEEDBACK | 120 |
| 11. | DESCRIPTION OF GLOBAL AMENDMENT(S) | 122 |
| 11.1 | GLOBAL AMENDMENT 1 | 122 |

| <b>Boehringer Ingelheim</b> |
|-----------------------------|
| BI Trial No.: 1305-0014 |
| c39145241-04 |

11.3

20 Sep 2023

| c3914524 | <b>41-04</b> | Clinical Trial Protocol | |
|---|---|---|---|
| Propriet | ary confidential in | formation © 2023 Boehringer Ingelheim International GmbH or | one or more of its affiliated companies |
| 11.2 | GLOBA | L AMENDMENT 2 | 125 |

BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ABBREVIATIONS AND DEFINITIONS

ADME Absorption, Distribution, Metabolism, Excretion

AE Adverse Event

AESI Adverse Event of Special Interest

AF Antifibrotic

ALAT Latin American Thoracic Association

ALT Alanine Aminotransferase
AMP Auxiliary Medicinal Products

ANCA Antineutrophil cytoplasmic antibodies

AP Alkaline phosphatase

aPTT Activated partial thromboplastin time

AST Aspartate aminotransferase ATS American Thoracic Society

AUC Area under the Curve

AZA Azathioprine

BI Boehringer Ingelheim

bid bis in die (twice daily dosing)

BMI Body Mass Index
CA Competent Authority

Cancer Antigen

cAMP Cyclic Adenosine Monophosphate

CI Confidence Interval CK Creatine kinase

CKD-EPI Chronic Kidney Disease - Epidemiology Collaboration

C<sub>max</sub> Maximum Plasma ConcentrationC<sub>min</sub> Minimum Plasma Concentration

C<sub>pre,ss</sub> Predose Concentration of Analyte in Plasma at Steady State

(e)COA (electronic) Clinical Outcome Assessment

COVID-19 Coronavirus Disease 2019
CRA Clinical Research Associate
(e)CRF (electronic) Case Report Form
CRO Contract Research Organization

CRP C-Reactive Protein

C-SSRS Columbia-Suicide Severity Rating Scale

CT Computed tomography

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol
CTR Clinical Trial Report

BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

CYP Cytochrome P450
DBL Database Lock

DILI Drug Induced Liver Injury

DLCO Diffusing Capacity (of Lung) for Carbon Monoxide

DMC Data Monitoring Committee
DNA Deoxyribonucleic Acid
ECG Electrocardiogram

eDC Electronic Data Capture

EDMS Electronic Document Management System

EDTA Ethylenediaminetetraacetic Acid eGFR Estimated glomerular filtration rate

EOS End of Study (corresponds with End of Trial)

EOT End of Treatment

ePRO Electronic Patient-Reported Outcome

EQ-5D EuroQol 5 Dimensional Quality of Life Questionnaire

ERS European Respiratory Society

ES Entered Set
EU European Union

EudraCT European Union Drug Regulating Authorities Clinical Trials Database

EuroQol European Quality of Life Group

FAS Full Analysis Set

FDA Food and Drug Administration

FEV1 Forced Expiratory Volume in 1 second

FU Follow-up

FVC Forced vital capacity

GBM Glomerular Basement Membrane

GCP Good Clinical Practice

GGT Gammaglutamyl transferase

GLI Global Lung Initiative

gMean Geometric Mean

GMP Good Manufacturing Practice

HA Health Authority

HADS Hospital Anxiety and Depression Scale

Hb Hemoglobin

HBV/HCV Hepatitis B or C Virus

HCRU Health Care Resource Utilization HIV Human Immunodeficiency Virus

HPLC-MS/MS High Performance Liquid Chromatography with Tandem Mass

Spectrometry

BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

HR Hazard Ratio

HRCT High-resolution Computed Tomography

i.v. Intravenous

IB Investigator's Brochure

IC<sub>50</sub> mean half-maximal inhibition

ICF Informed Consent Form

ICH International Council on Harmonisation of Technical Requirements for

Pharmaceuticals for Human Use

IDMS Isotope Dilution-mass Spectrometry

IEC Independent Ethics Committee

IFN-γ Interferon gamma

IGRA Interferon-Gamma Release Assay

IL Interleukin

ILD Interstitial Lung Disease

IMP Investigational Medical Product
INN International Non-Proprietary Name

INR International Normalized RatioIPD Important Protocol DeviationIPF Idiopathic Pulmonary Fibrosis

IRB Institutional Review Board

IRT Interactive Response Technology

ISF Investigator Site File

ISO International Organization for Standardization

iSpiro Handheld spirometer IUD Intrauterine Device

IUS Intrauterine Hormone-releasing System
IXRS Interactive Voice/Web Response Software

JRS Japanese Respiratory Society
LABA Long Acting Beta Agonist

LAMA Long Acting Muscarinic Antagonist

LOAEL Lowest Observed Adverse Effect Level

L-PF Living with Fibrosis Symptoms and Impact Questionnaire

LPLT Last patient last treatment
LPLV Last patient last visit
LPS Lipopolysaccharide

LTFU Lost To Follow Up

MACE Major Adverse Cardiovascular Event

MAR Missing At Random

MCH Mean Corpuscular Hemoglobin

BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

MCHC Mean Corpuscular Hemoglobin Concentration

MCV Mean Corpuscular Volume

MedDRA Medical Dictionary for Drug Regulatory Activities

mmHg Millimeters Mercury

MMRM Mixed-model repeated measures

MRD Multiple Rising Dose

mRNA Messenger Ribonucleic Acid miRNA Micro Ribonucleic Acid

MTX Methotrexate

NICE National Institute for Health and Care Excellence

NOAEL No observed adverse effect level

OC Oral contraceptive
OPU Operative Unit
p.o. per os (oral)

PCR Polymerase Chain Reaction
PDE Phosphodiesterase enzyme
PDE4B Phosphodiesterase 4B

PDE4i Phosphodiesterase inhibitor

PF Pulmonary Fibrosis

PF-ILD Progressive Fibrosing Interstitial Lung Disease

PFT Pulmonary Function Test

PGIS Patient's Global Impression of Severity

PGx Pharmacogenomics
PK Pharmacokinetics

PK/PD Pharmacokinetics/Pharmacodynamics

PPD Purified Protein Derivative PRO Patient-Reported Outcome

PT Preferred Term

Prothrombin Time

PV Pharmacovigilance RA Regulatory Authority

RBC Red blood cells

RDW Red Cell Distribution Width
REML Restricted maximum likelihood

REP Residual effect period RMP Risk Management Plan

RNA Ribonucleic Acid RS Randomized Set

SABA Short Acting Beta Agonist

BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

SAE Serious Adverse Event

SAMA Short-acting muscarinic antagonist

SARS-CoV-2 Severe Acute Respiratory Syndrome Coronavirus-2

SC Steering Committee SD Standard Deviation

SMC Safety Monitoring Committee SMQ Standardized MedDRA Queries

SoC Standard of Care

SOP Standard Operating Procedure

SpO2 Oxygen Saturation SRD Single Rising Dose

SUSAR Suspected Unexpected Serious Adverse Reactions

 $t_{1/2}$  Half-life time TB Tuberculosis

TBLC Transbronchial lung cryobiopsy

t<sub>max</sub> Timepoint of maximum plasma concentration

TMF Trial Master File

TNF-α Tumor Necrosis Factor alpha

TS Treated Set

TSAP Trial Statistical Analysis Plan

UGT Uridine Diphosphoglucuronosyl Transferase

UIP Usual interstitial pneumonia

ULN Upper limit of normal

US United States

V Visit vs. Versus

vWF von Willebrand Factor
WBC White blood cells

WHO World Health Organisation

WOCBP Woman of childbearing potential

**Clinical Trial Protocol** 

c39145241-04  Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. INTRODUCTION

BI 1015550, a preferential inhibitor of the phosphodiesterase 4B (PDE4B) isoenzyme which hydrolyzes and inactivates cyclic adenosine monophosphate (cAMP), is being developed by Boehringer Ingelheim (BI) for the treatment of idiopathic pulmonary fibrosis (IPF) and other forms of progressive pulmonary fibrosis.

#### 1.1 MEDICAL BACKGROUND

IPF and other progressive fibrosing interstitial lung diseases (PF-ILDs) share common pathophysiologic characteristics; alveolar epithelial cell injury and subsequent dysregulated repair, characterized by excessive deposition of extracellular matrix and loss of normal parenchymal architecture and lung function [P11-07084]. In IPF, fibroblasts exhibit unregulated proliferation and differentiate into myofibroblasts. The latter is considered the hallmark cell in the development and establishment of lung fibrosis [P12-03241]. Several growth factors are implicated in the proliferation, migration and transdifferentiation of the fibroblast and myofibroblast pool in pulmonary fibrosis.

As of date, nintedanib and pirfenidone are the only drugs registered for the treatment of IPF and recommended in the recent ATS/ERS/JRS/ALAT Clinical Practice Guideline for the Treatment of Idiopathic Pulmonary Fibrosis [P15-07362, R18-2794]. Nintedanib is also approved in the US, the European Union and many other countries for the treatment of other fibrosing ILDs with progressive phenotype. Despite the availability of these drugs, the medical need remains high in these devastating diseases.

#### 1.2 **DRUG PROFILE**

BI 1015550 is an oral preferential inhibitor of the PDE4B with broad anti-inflammatory and antifibrotic activities. Based on its mode of action, BI 1015550 is hypothesised to have complementary activity to current therapies in IPF and other forms of progressive pulmonary fibrosis. BI 1015550 shows a mean half-maximal inhibition (IC<sub>50</sub>) at 10 nM, with a nine-fold selectivity over phosphodiesterase 4D (PDE4 D; mean IC<sub>50</sub> 91 nM) without relevant known interaction with other targets (78 receptors and 42 enzymes tested at the very high concentration of 10 000 nM). In-vitro anti-inflammatory activity has been confirmed for TNF-α (IC<sub>50</sub>: 12 nM) and IL-2 release (IC<sub>50</sub>: 5 nM) from purified human peripheral blood mononuclear cells.



#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In the human ADME (mass balance) study, the total recovery of [<sup>14</sup>C]BI 1015550-related material was on average 95% of the administered dose with 58% excreted in faeces and 36% excreted in urine where 12% was excreted unchanged as parent compound.

#### **Drug-Drug Interaction:**

BI 1015550 is mainly metabolized by CYP3A with minor contributions from UGTs. Administration of BI 1015550 together with a strong CYP3A4 inhibitor increased AUC of BI 1015550 2.2-fold and  $C_{max}$  1.3-fold. In a clinical drug-drug interaction study with midazolam (sensitive CYP3A4 substrate), BI 1015550 was not shown to have a clinically relevant CYP3A induction.

Results from the Phase II trial 1305-0013 in patients with IPF showed that pre- and post-dose concentration levels of BI 1015550 were similar between patients treated with nintedanib and those not treated with any antifibrotic, suggesting nintedanib did not impact the exposure of BI 1015550. However, a 35-50% lower exposure was observed in IPF patients on background treatment with pirfenidone. Clinical relevance of this level of decrease in BI 1015550 exposure is unclear based on the limited data and will further be evaluated in a separate drug-drug interaction trial.

#### Residual Effect Period

The Residual Effect Period (REP) of BI 1015550 is \_\_\_\_\_. This is the period after the last dose with measurable drug levels and/or pharmacodynamic effects still likely to be present.

### Data from non-clinical toxicology studies

The toxicity profile for BI 1015550 has been assessed in safety pharmacology studies, genetic toxicity studies, and repeat dose toxicity studies in the rat, minipig, and monkeys of up to 26, 39, and 39 weeks, respectively. In addition, a fertility and early embryonic development (rat) and embryo-fetal development toxicity studies (rat and rabbit) were conducted. Decreased mating, fertility, and pregnancy indices were observed in male and female rats at a dose level that also caused evidence of severe toxicity in both sexes. In rats but not in rabbits fetal loss was increased. Teratogenicity and fetotoxicity was not observed. In long-term toxicity studies in rats (26 weeks), minipig (39 weeks) and monkeys (39 weeks) there was no microscopic evidence of changes in female reproductive organs or on male spermatogenesis. A sporadic menstrual cycle prolongation was observed in the 39-week study in female monkeys receiving ≥10 mg/kg/day, i.e., at approximately 4-fold human exposure at 18 mg bid. Vasculopathy and mortality secondary to vasculopathy are the primary findings defining the NOAEL and LOAEL in the rat and minipig, respectively. In contrast, vascular changes were not observed in 13-week and 39-week monkey studies at 30 mg/kg/day, supporting the decreased sensitivity of primates to PDE4i-induced vascular changes. Vasculopathy is a well characterized class-effect pathology associated with PDE4 inhibitors [R10-1559] and has not been demonstrated in humans administered marketed PDE4i apremilast and roflumilast.

#### Data from clinical studies

Treatment with BI 1015550 at 18 mg twice daily in a Phase II proof-of-concept trial preserved lung function in patients with IPF over a period of 12 weeks, either as a monotherapy or on top of approved antifibrotic standard of care (nintedanib or pirfenidone). BI 1015550 showed acceptable safety and tolerability in the overall study population and in the subgroups of patients without or with background antifibrotic treatment.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In this trial 97 patients were exposed to BI 1015550 and 50 patients to placebo. The most frequently reported AEs were gastrointestinal disorders (32.0% in the BI 1015550 group, 24.0% in the placebo group). Diarrhea was the most common AE, with a higher frequency in the BI 1015550 group (23.7%) than in the placebo group (12.0%) and diarrhea was also the most common event leading to treatment discontinuation (3 patients, all in the BI 1015550 group and all on background treatment with nintedanib). However, the majority of diarrhea events were mild in intensity.

AEs leading to discontinuation of trial treatment were only observed in the BI 1015550 treatment group. Apart from the mentioned 3 patients with diarrhoea and 2 patients with COVID-19, all events occurred in single patients without any pattern or cluster. Serious adverse events were reported in 10.0% of patients in the placebo group and 6.2% of patients in the BI 1015550 treatment group. There were two events with fatal outcome in the BI 1015550 treatment group, one patient with COVID-19 pneumonia and one patient with suspected IPF exacerbation and suspected vasculitis (the diagnosis of vasculitis could not be confirmed by the sponsor nor the independent external data monitoring committee). Risk factors were present in both fatal events.

There were no clinically relevant changes in vital signs (including body weight) and/or ECG parameters (including QTc) observed. No changes in the C-SSRS and no AEs of suicidal ideation or behaviour were reported during trial treatment.

The primary endpoint for efficacy in this trial was met, with a relevant treatment effect in favour of BI 1015550 on the change from baseline in FVC at 12 weeks in patients with IPF. Treatment with BI 1015550 preserved FVC irrespective of background antifibrotic treatment, in contrast to the placebo groups in which a marked decline in FVC was observed. (non-AF stratum:  $-95.62 \pm 30.75$  mL under placebo vs.  $6.10 \pm 22.90$  mL with BI 1015550; AF stratum:  $-77.70 \pm 23.60$  mL under placebo vs.  $2.72 \pm 18.13$  mL).

Overall, in Phase Ic and II trials in patients with IPF, BI 1015550 at a dose of 18 mg bid for up to 12 weeks showed acceptable safety and tolerability, both in patients without or with background antifibrotic treatment (nintedanib or pirfenidone).

For a more detailed description of the BI 1015550 profile, please refer to the Investigator's Brochure (IB) current version [c02094779].

### 1.3 RATIONALE FOR PERFORMING THE TRIAL

The purpose of this trial is to evaluate the efficacy, safety, and tolerability of BI 1015550 9 mg bid and 18 mg bid compared to placebo in patients with IPF in addition to patient's standard of care. This trial's primary objective is to demonstrate the ability of BI 1015550 to reduce lung function decline based on Forced Vital Capacity (FVC) between baseline and Week 52 when compared to placebo.

Efficacy and safety of BI 105550 will be assessed in patients with IPF both on approved antifibrotic therapy (i.e. nintedanib or pirfenidone) (AF group) or not on an antifibrotic background therapy (non-AF group).

Despite the availability of nintedanib and pirfenidone as antifibrotic therapies, there remains a high unmet medical need for more efficacious and better tolerated treatments for patients


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

living with IPF. Currently available treatments reduce the decline in FVC compared to placebo, but do not completely stop the deterioration of lung function over time; patients still experience worsening of symptoms and quality of life or experience exacerbations of their disease. Mortality remains high in this patient population. Suboptimal tolerability with current treatment options is an unmet need that can impact patient's ability to remain on standard of care.

Based on its anti-inflammatory and antifibrotic properties and the preliminary clinical evidence described, BI 1015550 may provide an additional treatment option to patients with pulmonary fibrosis irrespective of concomitant treatment with currently approved antifibrotics as standard of care.

#### 1.4 BENEFIT - RISK ASSESSMENT

#### 1.4.1 Benefits

IPF and other progressive fibrosing ILDs are serious debilitating conditions characterised by worsening symptoms and quality of life, progressive loss of lung function, ultimately resulting in respiratory failure, and early death. At the same time, the currently approved antifibrotic treatments have limitations: they do not impact symptoms and cannot stop or reverse fibrosis, i.e. the disease trajectory.

Data from the Phase II trial 1305-0013 in patients with IPF indicated a beneficial treatment effect of 18 mg BI 1015550 bid, with the preservation of FVC over 12 weeks together with an acceptable safety and tolerability profile supporting further investigation in Phase III clinical trials as a treatment for IPF and other forms of progressive pulmonary fibrosis. Patients with IPF who receive treatment with BI 1015550 have the potential benefit of slowing lung function decline, improving symptoms, and improving quality of life over a long-term period.

#### 1.4.2 **Risks**

There are no identified risks (side effects) for BI 1015550, based on the toxicology program or any clinical trials conducted for this product to date. Vasculitis and foetal loss are considered as important potential risks based only on nonclinical findings.

Apart from risks related to trial procedures, the risks shown in <u>Table 1.4.2: 1</u> below are hypothetical in nature; these are derived from general safety considerations of immunomodulatory drugs and from nonclinical and clinical data of compounds with a comparable mode of action. For clinical data including adverse events reported during clinical trials with BI 1015550 please refer to Section 1.2.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 1.4.2: 1 Overview of trial related risks

| Possible or known risks of clinical relevance for this trial | Summary of data, rationale for the risk | Mitigation strategy |
|---|---|---|
| Pharmacokinetic interaction with strong CYP3A4 inhibitors | <ul> <li>CYP450 3A4 is regarded as the major enzyme responsible for BI 1015550 metabolism in human hepatocytes and predicted to contribute to ~70% of its hepatic metabolism.</li> <li>In a drug-drug interaction trial, the strong CYP3A4 inhibitor itraconazole increased the exposure to BI 1015550 by 1.3-fold (Cmax) and 2.2-fold (AUC).</li> </ul> | Potent CYP3A inhibitors are restricted medication. If short-term treatment with potent CYP3A4 inhibitor is needed, trial medication needs to be paused |
| Vasculitis | <ul> <li>Vasculopathy is an established nonclinical toxicity of PDE4 inhibitors.</li> <li>Vasculitis has been shown in both the rats and minipigs following oral administration of BI 1015550 but not in 13- or 39-week studies in monkeys.</li> <li>Vasculitis is listed as an important potential risk in the RMP for the marketed PDE4- inhibitor apremilast.</li> <li>In marketed PDE4 inhibitors, vasculitis has not been identified as an adverse drug reaction in humans</li> </ul> | Active vasculitis (unstable or uncontrolled) is an exclusion criterion. Vasculitis assessment as part of AE questioning Close clinical monitoring for AEs of vasculitis Assessment of (suspected) vasculitis events by independent adjudication and data monitoring committee. Treatment interruption in case of any vasculitis adverse event. Restart only if not BI 1015550 related and considered acceptable by the investigator |
| Weight decrease in<br>underweight patients<br>(BMI <18.5 kg/m <sup>2</sup> ) | For the marketed PDE4-inhibitors apremilast and roflumilast weight loss in underweight patients is an identified important risk. | <ul> <li>Body weight evaluated regularly during the trial.</li> <li>Patients who have a BMI &lt;18.5 kg/m², and subsequently experience unexplained and clinically significant weight loss (&gt;10%) will be discontinued from trial treatment.</li> </ul> |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Possible or known<br>risks of clinical<br>relevance for this<br>trial | Summary of data, rationale for the risk | Mitigation strategy |
|---|---|---|
| Psychiatric disorders: Depression and anxiety Suicidality | <ul> <li>For the marketed PDE4 inhibitors depression is listed as a side effect. They are associated with increased risk of depression with some patients reporting suicidal ideation and/or attempts, with some reported cases of completed suicide.</li> <li>High incidence of depression in the ILD population per se.</li> <li>In IPF patients treated with 18 mg BI 1015550 bid for up to 12 weeks, no on-treatment events of suicidal ideation or behavior and no events of depression or anxiety were reported</li> </ul> | <ul> <li>Acute or chronic severe depression defined as Hospital Anxiety and Depression Scale (HADS) subscore &gt;14 at screening will be excluded</li> <li>Any suicidal behavior in the past 2 years and any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 3 months or at Visit 1 are exclusion criteria.</li> <li>Prospective monitoring for depression and anxiety will be performed using the HADS and the C-SSRS</li> <li>Patient's withdrawal criteria in case of new-onset severe depression defined as HADS subscore &gt;14 and/or suicidal behavior or any suicidal ideation of type 4 or 5 in the C-SSRS.</li> </ul> |
| Severe Infections including, serious, opportunistic and Mycobacterium tuberculosis infections | <ul> <li>Inhibition of the immune response due to the anti-inflammatory mode of action of BI 1015550 potentially increases the risk of infections, including COVID-19</li> <li>Serious infections were balanced between placebo and BI 1015550 in Phase II trial</li> <li>Nasopharyngitis was more frequently reported under treatment with BI 1015550 in Phase I trials and the numbers were very small</li> </ul> | <ul> <li>Screening procedures for infections are defined for this trial. Patients with any relevant chronic or acute infections including human immunodeficiency virus (HIV), viral hepatitis or active tuberculosis are excluded from the trial.</li> <li>Treatment of infections should be initiated promptly according to standards of care.</li> <li>Treatment interruption in case of severe acute infection until the patient has recovered based on the investigator's medical judgement</li> </ul> |
| MACE and tachyarhythmia | <ul> <li>Important potential risk for marketed PDE4 inhibitor apremilast</li> <li>In nonclinical studies with BI 1015550 no adverse cardiovascular findings detected</li> <li>In clinical trials with BI 1015550 no relevant findings were observed</li> </ul> | These risks will be addressed by careful safety monitoring and safety measures such as close clinical monitoring for AEs regular monitoring of vital signs and ECG assessments Adjudication committee for MACE events in Phase III |

 Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Possible or known risks of clinical relevance for this trial | Summary of data, rationale for the risk | Mitigation strategy |
|---|---|---|
| Malignancies | Inhibition of the immune response with an immunomodulatory drug may potentially impair immune defences and thus theoretically decrease immune defense against malignancies. | <ul> <li>Patients with a recent history of malignancy within 5 years will be excluded from participation in this trial except patients with appropriately treated basal cell carcinoma or in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix</li> <li>In case of occurrence of malignant neoplasm other than appropriately treated basal cell carcinoma or in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix, the investigator should discontinue trial treatment</li> <li>Diagnostics and treatment have to be initiated according to local standard of care.</li> </ul> |
| Gastrointestinal<br>disorders (e.g.<br>diarrhoea, nausea,<br>vomiting, abdominal<br>pain) | <ul> <li>Vomiting and diarrhea are important dose-limiting side effects of marketed oral PDE-4 inhibitors.</li> <li>Diarrhoea was the most frequently reported adverse event in Phase II with the majority of events being of mild intensity.</li> <li>Gastrointestinal disorders are very common or common side effect of the approved antifibrotics.</li> </ul> | <ul> <li>Increased awareness of symptoms.</li> <li>Careful monitoring of hydration in patients with diarrhoea recommended.</li> <li>Management strategies as described in approved labels of antifibrotics have to be followed.</li> <li>Symptomatic treatment, e.g. loperamide, if required</li> <li>Treatment interruption if needed</li> </ul> |
| Reproductive toxicity: • Fetal loss • Decreased fertility | <ul> <li>No teratogenicity was seen in 2 species in preclinical studies and exposure with BI 1015550 via the semen is expected to be very low.</li> <li>In rats, male and female fertility was potentially reduced. Long term toxicity studies with BI 1015550 in rat and monkey showed no microscopic evidence of changes in female reproductive organs or male spermatogenesis. For another PDE4 inhibitor with comparable nonclinical findings, clinical data showed no effect on male fertility and sperm in humans.</li> <li>In monkeys, a sporadic prolongation in menstrual cycles was observed at approximately ≥4-fold human exposure at 18 mg BI 1015550 bid.</li> <li>Fetal loss was increased in female rats treated with BI 1015550.</li> </ul> | <ul> <li>Women of childbearing potential (WOCBP) need to use a highly effective method of contraception. WOCBP taking oral contraceptives (OCs) also have to ensure the use of one barrier method during sexual intercourse with their partner, e.g., condom to account for the risk of potentially reduced efficacy of the OCs in the event of severe vomiting and diarrhea</li> <li>In case of vomiting or diarrhea, instructions in the label of the OC should be followed</li> <li>In case of prolonged (&gt;48h) or repeated vomiting/diarrhea, the use of an alternative highly effective contraceptive measure should be considered</li> <li>Regular pregnancy testing for WOCBP</li> <li>Treatment discontinuation in case of pregnancy</li> </ul> |

# **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Possible or known<br>risks of clinical<br>relevance for this<br>trial | Summary of data, rationale for the risk | Mitigation strategy |
|---|---|---|
| | General safety topics | |
| Drug-induced liver injury (DILI) | • Rare but severe event, standard topic of interest for products in development thus under constant surveillance by sponsors and regulators. | • Timely detection, evaluation, and follow-up of laboratory alterations in selected liver laboratory parameters to ensure patients' safety. |
| | Trial procedures | |
| Blood Sampling | • As with all blood sampling, there is a risk of mild pain, local irritation, or bruising (a black or blue mark) at the puncture site. Furthermore, there is a small risk of light-headedness and/or fainting. In rare cases, the puncture site can also become infected or nerves may be damaged, inducing long-lasting abnormal sensations (paraesthesia), impaired sensation of touch and persistent pain. | These risks will be addressed by careful safety monitoring and risk mitigation measures such as: close clinical monitoring for AEs selection of experienced sites and site staff |
| Chest HRCT | • The more radiation is received over the course of a life, the greater risk of having cancerous tumours or of inducing changes in genes. The changes in genes possibly could cause abnormalities or disease in future offspring. The radiation in this trial is not expected to greatly increase these risks, but the exact increase in such risks is not known. | <ul> <li>New HRCT measurement only required in case no historical record (not older than 12 months at the time of screening) is available or in case of insufficient quality.</li> <li>These risks will be addressed by careful safety monitoring and risk mitigation measures such as: <ul> <li>close clinical monitoring for AEs</li> <li>selection of experienced sites and site staff</li> </ul> </li> </ul> |
| Lung function<br>measurements<br>(Spirometry and<br>DLCO) | Risks and discomforts associated with<br>lung function testing may include<br>shortness of breath, dizziness, or<br>headache during the breathing tests. | These risks will be addressed by careful monitoring and risk mitigation measures such as: close clinical monitoring for AEs selection of experienced sites and site staff Training from vendor to conduct correct manoeuvre. |
| | Other risks | |
| Administration of<br>Placebo or<br>BI 1015550 | • If the patient is randomized to receive<br>a placebo or BI 1015550, the patient's<br>condition could get worse during the<br>course of the trial. | In an event of disease worsening,<br>treatment with standard of care is<br>always an option per physician<br>discretion for all randomized patients |


#### **Clinical Trial Protocol**

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1.4.3 Discussion

Treatment with BI 1015550 has the potential to provide significant benefit to patients with IPF and other progressive fibrosing ILDs by ultimately slowing lung function decline, improving symptoms and quality of life over a long-term period.

The obtained toxicology data support administration of BI 1015550 to women and men in the planned Phase III clinical trials in patients with IPF and other forms of progressive pulmonary fibrosis irrespective of background antifibrotic treatment, except for women who are pregnant or breastfeeding. Women of childbearing potential must use a highly effective method of contraception (for details please refer to Sections 3.3.2 and 4.2.2.3).

Data from the Phase II trial 1305-0013 in patients with IPF indicated a beneficial treatment effect of 18 mg BI 1015550 bid, with the preservation of FVC over 12 weeks together with an acceptable safety and tolerability profile supporting further investigation in Phase III clinical trials as a treatment for IPF and other forms of progressive pulmonary fibrosis. Based on the clinical and nonclinical data available to date, no risks (side effects) were identified. There are no listed events.

Considering the unmet medical need and anticipated benefit of BI 1015550, and the lack of compound or mechanism related safety signals, the benefit risk evaluation of BI 1015550 for the treatment of IPF and other progressive fibrosing ILDs is favourable.

## 2. TRIAL OBJECTIVES AND ENDPOINTS

### 2.1 MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS

### 2.1.1 Main objectives

The trial will evaluate efficacy and safety of BI 1015550 9 mg and 18 mg bid compared to placebo in patients with IPF in addition to the patient's standard of care treatment.

The primary objective is to demonstrate a reduction in lung function decline as measured by the change from baseline in FVC for BI 1015550 when compared to placebo in patients with IPF.

The main secondary objective of the trial is to demonstrate BI 1015550's ability in reducing the occurrence of clinically meaningful events such as acute IPF exacerbation, hospitalization for respiratory cause or death over the duration of the trial when compared to placebo in patients with IPF. An additional secondary objective of the trial is to show an effect of BI 1015550 on symptoms and lung function.

### 2.1.2 Primary endpoint

The primary endpoint of the trial is the absolute change from baseline in Forced Vital Capacity (FVC) [mL] at Week 52.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2.1.3 Key Secondary endpoint

The key secondary endpoint in this trial is time to the first occurrence of any of the components of the composite endpoint: time to first acute IPF exacerbation, first hospitalization for respiratory cause, or death (whichever occurs first) over the duration of the trial.

# 2.1.4 Secondary endpoints

The secondary endpoints of the trial are:

- Time to first acute IPF exacerbation or death over the duration of the trial
- Time to hospitalization for respiratory cause or death over the duration of the trial
- Time to absolute decline in FVC % predicted of >10% from baseline or death over the duration of the trial
- Time to absolute decline in (DLCO) % predicted of >15% from baseline or death over the duration of the trial
- Time to death over the duration of the trial
- Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms Dyspnea domain score at Week 52
- Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms Cough domain score at Week 52
- Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms Fatigue domain score at Week 52
- Absolute change from baseline in FVC % predicted at Week 52
- Absolute change from baseline in DLCO % predicted at Week 52



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



## 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

### 3.1 OVERALL TRIAL DESIGN

This Phase III trial (1305-0014) is a multi-centre, multi-national, prospective, randomized, placebo-controlled, double blind clinical trial to investigate the efficacy and safety of BI 1015550 at a dose of 9 mg bid and 18 mg bid in patients with IPF over at least 52 weeks.

A total of approximately 963 patients will be randomized into the trial of which 321 patients will be in each active treatment group and in the placebo group.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

After signing the informed consent, the initial visit (Visit 1) will be conducted to determine eligibility. Eligible patients will enter the randomization visit (Visit 2) to allow collection of all clinical and safety information and review of all inclusion and exclusion criteria. Patients will be randomized in a 1:1:1 ratio into either BI 1015550 9 mg bid, BI 1015550 18 mg bid or placebo and then enter the treatment phase for at least 52 weeks.

Patient randomization will be stratified by the presence of background treatment with antifibrotics (AF group vs. non-AF group).

- *Non-AF group*: patients not treated with an approved antifibrotic medication (nintedanib or pirfenidone) in the last 8 weeks prior to enrolment, (e.g. patients previously treated with antifibrotics, but discontinued that treatment or patients never treated with antifibrotics before).
- *AF group*: patients on a stable treatment with an approved antifibrotic drug (e.g. nintedanib or pirfenidone) for at least 12 weeks at study entry, and are planned to stay on this background treatment after randomization.

The trial will be conducted in 2 parts. Treatment Period A of the trial will consist of Visits 2 through 10, until one year after randomization. Treatment Period B will begin following completion of the Week 52 visit (Visit 10); patients will continue treatment with blinded trial medication in Treatment Period B and have trial visits every 12 weeks. Assuming a respective recruitment period (about 18 months), first randomized patients may be on trial treatment for up to 130 weeks.

The main analysis of this study will be performed once the last randomized patient reaches the Week-52 visit (Visit 10 at the end of Part A). At that time, a first database lock (DBL1; Figure 3.1: 1) will occur and all data will be unblinded to the sponsor. Efficacy and safety analyses will be performed on the data from Part A of the trial to assess the benefit-risk of BI 1015550 over 52 weeks. In addition, data collected in Part B of the trial (after 52 weeks) and available at the time of data cut-off for the main analysis will be reported together with data from Part A (i.e. over the whole trial).

Trial 1305-0014 Part B, will continue until all patients have completed the EOT visit and the EOS visit as applicable. A final database lock (DBL2; Figure 3.1: 1) will then occur and a final analysis based on the data over the whole trial will be carried out.

Depending on the results of the evaluation based on DBL1 and determination of the BI 1015550 dose with the more favorable benefit-risk profile, patients receiving trial medication until the end of Part B will be eligible for open-label treatment with BI 1015550 in a separate extension trial.

After review of the efficacy and safety data available at DBL1, the sponsor will communicate the end of the trial and all patients still on blinded study treatment will perform an End of Treatment (EOT) visit and an End of Study (EOS) visit if applicable. The trial ends when all patients complete these visits. Details on follow-up and rollover to the extension trial are given in Section 6.2.3.

First patient

randomized

c39145241-04 



Figure 3.1: 1 Trial design overview at patient level (upper panel) and trial level (lower panel)

#### 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF **CONTROL GROUP(S)**

Last patient

randomized

This trial is a placebo-controlled, randomized, double-blind trial to provide the highest scientific rigor and is thus considered the most appropriate design. FVC measurement over time is a widely accepted clinical endpoint in the indication of the trial for the evaluation of treatment effects on lung function. FVC assessments are supported by clinically meaningful outcomes and patient-reported outcomes as secondary endpoints.

A placebo-controlled study design is considered justified in the trial, as it will be conducted in addition to the patient's standard of care at the time of enrollment:

- Patients who are on a stable treatment with antifibrotic treatment at the time of screening and randomization are planned to continue this background treatment during the trial.
- Patients without an AF background treatment at enrollment and randomization will be allowed to initiate a treatment with an approved antifibrotic agent in case of IPF progression and/or exacerbation after the first 12 weeks of treatment in the trial.

Stratification will be based on presence of AF background treatment and will facilitate the interpretation of the efficacy and safety data in patients that use BI 1015550 alone or in

Last patient

completes

52 weeks

DBL1

Main

analysis

Last patient

completes

trial

DBL2

Final

analysis

#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

addition to an antifibrotic agent. The expected proportion of the respective subgroups of patients with or without background antifibrotic treatment corresponds to the current treatment/prescription practices across the participating countries (70% vs. 30%), so that patients can be accepted to the trial without modification of the ongoing SoC treatment.

The minimum treatment period of 52 weeks is selected according to the respective guidance from the American and European Clinicians organisations on the investigation of treatment effects on FVC in IPF (2015 ATS/ERS/JRS/ALAT Guideline [P15-07362]), where based on the natural decline during disease progression, a minimal follow up of the effects of new drugs for 52 weeks is recommended. However, clinical endpoint data are needed to provide evidence of a clinically meaningful effect beyond a decreased decline of FVC. Based on the incidence rates of these clinically meaningful events included in the key secondary endpoint (IPF exacerbation, respiratory hospitalization, and death), the blinded treatment should be extended to a long-term treatment beyond 52 weeks. This is reflected with the continuation of study participation for up to 130 weeks with the additional Treatment Period B for patients that are recruited early in the trial. The additional data collected while patients remain on blinded treatment beyond 52 weeks will provide supportive long-term efficacy and safety data on the effect of BI 1015550 in a controlled manner. Due to the varying length of follow-up in Part B of the trial, the efficacy analyses incorporating data from Part A and Part B will focus on time-to-event endpoints.

This trial will include an option for participants and participant caregivers to complete anonymized questionnaires to provide feedback on their clinical trial experience. Providing this feedback is not required for trial participation, and information collected from these questionnaires will not be analyzed as part of the clinical data for the trial (see Section 10.7).

#### 3.3 SELECTION OF TRIAL POPULATION

Patients with IPF will be screened at approximately 400 sites to ensure randomization of about 963 patients, 321 in the active treatment arms and 321 in the placebo group.

During the recruitment period, the number of patients randomized with an approved background AF-treatment and without AF background treatment will be closely monitored. If necessary, recruitment of one group may be stopped in order to achieve sufficient representation of both groups.

Screening of patients for this trial is competitive, i.e. screening for the trial will stop at all sites once a sufficient number of patients has been screened. Investigators will be notified about screening completion and will then not be allowed to screen additional patients for this trial. Patients already in screening at this time will be allowed to continue to randomization if eligible.

A log of all patients enrolled into the trial (i.e. who have signed informed consent) will be maintained in the Investigator Site File (ISF) irrespective of whether they have been treated with investigational drug or not.

If retrospectively it is found that a patient has been randomized in error (did not meet all inclusion criteria or met one or more exclusion criteria), the sponsor or delegate should be

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

contacted immediately. Based on an individual benefit-risk assessment, a decision will be made whether continued trial participation is possible or not.

# 3.3.1 Main diagnosis for trial entry

Patients diagnosed with IPF who comply with trial requirements may qualify to participate in the trial. The diagnosis is based on (Appendix 10.6):

- The 2022 ATS/ERS/JRS/ALAT Guideline [P22-03204] as confirmed by the investigator based on chest HRCT scan taken within 12 months of Visit 1 and, if available, surgical lung biopsy or transbronchial lung cryobiopsy, and
- "UIP" or "Probable UIP" HRCT pattern consistent with the clinical diagnosis of IPF, as confirmed by central review prior to Visit 2.
  - O Patients with an "Indeterminate" HRCT finding are eligible if a clinical diagnosis of IPF can be confirmed locally based on (historical) surgical lung biopsy or cryobiopsy demonstrating a "UIP" or "Probable UIP" histopathology pattern. (Table 10.6: 1)
  - Patients with an "Alternative diagnosis" HRCT finding are eligible if a clinical diagnosis of IPF can be confirmed locally based on (historical) surgical lung biopsy or cryobiopsy demonstrating a "UIP" histopathology pattern. (<u>Table 10.6:</u> 1)

Please refer to Section <u>8.3.1</u> (Source Documents) for the documentation requirements pertaining to the inclusion and exclusion criteria.

### 3.3.2 Inclusion criteria

- 1. Patients  $\geq$ 40 years old at the time of signed informed consent.
- 2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
- 3. Diagnosis of IPF (Section 3.3.1)
- 4. Patients may be either:
  - on a stable therapy\* with nintedanib or pirfenidone for at least 12 weeks prior to Visit 1 and during screening and are planning to stay on this background treatment after randomization. Combination of nintedanib plus pirfenidone is not allowed. \*stable therapy is defined as the individually and general tolerated regimen of either nintedanib or pirfenidone (no dose changes) for at least 12 weeks.
  - o not on a treatment with nintedanib or pirfenidone for at least 8 weeks prior to Visit 1 and during the screening period (e.g. either AF-treatment naïve or previously discontinued) and do not plan to start or re-start antifibrotic treatment.
- 5. Forced Vital Capacity (FVC) ≥45% of predicted normal at Visit 1.
- 6. DLCO ≥25% of predicted normal corrected for hemoglobin (Hb) at Visit 1.
- 7. Women of childbearing potential (WOCBP)<sup>1</sup> must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OCs) also have to use one barrier method; please refer to Section 4.2.2.3.

<sup>&</sup>lt;sup>1</sup> A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.3 Exclusion criteria

- 1. Prebronchodilator FEV1/FVC < 0.7 at Visit 1
- 2. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
- 3. Acute IPF exacerbation within 3 months prior to Visit 1 and/or during the screening period (investigator-determined).
- 4. Relevant chronic or acute infections including human immunodeficiency virus (HIV) and viral hepatitis.
- 5. Confirmed infection with SARS-CoV-2 not fully recovered according to investigator judgement within the 4 weeks prior to randomization (Visit 2).
- 6. Major surgery (major according to the investigator's assessment) performed within 6 weeks prior to Visit 2 or planned during the trial period, e.g. hip replacement. Registration on lung transplantation list would not be considered as planned major surgery.
- 7. Any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1, except appropriately treated basal cell carcinoma of the skin, in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
- 8. AST or ALT >2.5 x ULN or total Bilirubin >1.5 x ULN at Visit 1.
- 9. eGFR ≤30 ml/min/1.73 m² at Visit 1. (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula or Japanese version of CKD-EPI for Japanese patients)
- 10. Patients with underlying liver cirrhosis (Child Pugh A, B or C hepatic impairment).
- 11. Cardiovascular diseases, any of the following:
  - a. Severe hypertension (uncontrolled under treatment ≥160/100 mmHg at multiple occasions) within 3 months of Visit 1
  - b. Myocardial infarction, stroke or transient ischemic attack within 6 months of Visit 1
  - c. Unstable cardiac angina within 6 months of Visit 1
- 12. Patients who are treated with immunomodulatory medications (other than oral corticosteroids) or prednisone >15 mg/day or equivalent for respiratory or pulmonary reasons.
- 13. Active vasculitis, unstable or uncontrolled within 8 weeks prior to Visit 1 or during the screening period.
- 14. Any suicidal behaviour in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
- 15. Any suicidal ideation of type 4 or 5 on the C-SSRS in the past 3 months or at Visit 1 and/or Visit 2 (i.e. active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, intent and plan).
- 16. Acute or chronic severe depression defined as HADS subscore >14 at Visit 1 and/or Visit 2.
- 17. Patients who must or wish to continue the intake of restricted medications (see Section 4.2.2.1) or any drug considered likely to interfere with the safe conduct of the trial. Please note: potent CYP3A4 inhibitors should not be taken 5 half-life times prior to Visit 1.
- 18. Patients treated with PDE1, PDE3, PDE4, PDE10 inhibitors, and non-selective PDE inhibitors within 30 days before Visit 1
- 19. Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant).


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 20. Inability to refrain from smoking on trial visit days.
- 21. History of allergy or hypersensitivity or contraindications to the class of drugs under study including known hypersensitivity to the drug or its excipients.
- 22. Patients with a significant disease or condition other than the ILD under study, which in the opinion of the investigator, may put the patient at risk because of participation, interfere with study procedures, or cause concern regarding the patient's ability to participate in the study.
- 23. Patients with active tuberculosis (TB).
- 24. Previous randomization in this trial or in trial 1305-0023.
- 25. Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s) or receiving other investigational treatment(s).
- 26. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
- 27. History of stem cell therapy for the treatment of pulmonary fibrosis.

# 3.3.4 Discontinuation of patients from treatment or assessments

Patients may discontinue trial treatment or withdraw consent to trial participation as a whole ("withdrawal of consent") with very different implications; please see Sections 3.3.4.1 and 3.3.4.2 below.

However, if the patient agrees, every effort should be made to keep randomized patients in the trial, even if continuing trial treatment is not possible. They should attend further trial visits to ensure their safety and to collect important trial data, e.g. FVC measurement at Week 52.

Measures to control the withdrawal rate include careful patient selection, appropriate explanation of the trial requirements and procedures prior to trial enrolment, as well as the explanation of the consequences of withdrawal.

The decision to discontinue trial treatment or withdraw consent to trial participation and the respective reason must be documented in the patient files and CRF. If applicable, consider the requirements for Adverse Event collection and reporting (please see Section 5.2.6.2).

#### 3.3.4.1 Discontinuation of trial treatment

The End of Treatment (EOT) visit activities will be performed when a patient discontinues trial medication **permanently**.

A premature Follow-up (FU) visit is to be performed 7 days (+3 days) after end of treatment. If the patient discontinued the trial medication more than a week prior to the EOT visit, this FU visit is not required.

Ideally, patients who permanently discontinue trial medication should attend all remaining visits after treatment discontinuation. For those patients who are unable to complete the scheduled visits, at least phone contacts should occur at the scheduled visit time points. Should that not be acceptable, a phone contact at 52 weeks after randomization and at the end of the planned observation period should occur to collect the most relevant information: vital status (please see Section <u>5.2.6.2.1</u>), adverse events, or last contact date in case of lost to

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

follow-up (LTFU). Every effort should be done to obtain the vital status information in case of LTFU. The number of LTFU patients should be limited. The need to obtain vital status information will be part of the patient information/informed consent procedure.

An individual patient will discontinue trial treatment permanently if:

- The patient wants to discontinue trial treatment. The patient will be asked to explain the reasons but has the right to refuse to answer.
- The patient has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both the investigator and sponsor representative, the safety of the patient cannot be guaranteed as he/she is not willing or able to adhere to the trial requirements in the future.
- The patient exhibits suicidality, in the clinical judgment of the investigator or according to the following criteria:
  - o any suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
  - o any suicidal ideation of type 4 or 5 in the C-SSRS (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
- In case of occurrence of malignant neoplasm other than appropriately treated basal cell carcinoma or in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
- The patient will undergo lung transplantation, with an assigned date of surgery.
- The patient becomes pregnant. For further details, please refer to Section <u>5.2.6.2.3</u>
- Patients with a BMI <18.5 kg/m<sup>2</sup> that experience an additional, unexplained and clinically significant (>10%) weight loss during trial treatment

An individual patient should discontinue trial treatment **temporarily** if:

- The patient has a new onset of severe depression as defined by a HADS subscore >14.
  - Re-introduction of IMP could be considered after the patient has recovered, individual benefit-risk evaluation by the investigator and exclusion of BI 1015550-induced depression
- The patient fulfills the AESI definition of hepatic injury.
  - Re-introduction of IMP could be considered after the patient has recovered, individual benefit-risk evaluation by the investigator and exclusion of BI 1015550-induced liver injury
- The patient has an event suspicious of vasculitis
  - If thorough evaluation does not confirm a causal relationship between trial medication and the event, treatment may be restarted based on the investigator's medical judgement.
- The patient needs to take concomitant medication that interferes with the safety of the investigational medicinal product or other trial treatment, e.g. CYP3A4 inhibitors as listed in Appendix 10.4.1,
  - Re-introduction of IMP could be considered at least 5 half-life times after the restricted medication has been stopped
- The patient has to stop trial treatment for medical reasons such as surgery, adverse events, other diseases.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For patients who temporarily pause the trial treatment due to specific adverse events (refer to Section 4.2.1) such as diarrhoea, severe infections, vasculitis, and concomitant medication related issues, every effort should be made to restart trial treatment if medically justified. The decision and associated reasoning for the restart of trial treatment should be documented in source data.

If new efficacy/safety information becomes available, Boehringer Ingelheim will review the benefit-risk-assessment and, if needed, pause or discontinue the trial treatment for all patients or take any other appropriate action to guarantee the safety of the trial patients or take any other appropriate action to guarantee the safety of the trial patients.

### 3.3.4.2 Withdrawal of consent to trial participation

Patients may withdraw their consent to trial participation at any time without the need to justify the decision.

If a patient wants to withdraw consent, the investigator should be involved in the discussion with the patient and explain the difference between trial treatment discontinuation and withdrawal of consent to trial participation, as well as explain the options for continued follow-up after trial treatment discontinuation, please see Section 3.3.4.1.

## 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site.
- 2. New efficacy or safety information invalidating the earlier positive benefit-risk assessment, please refer to Section 3.3.4.1.
- 3. Deviations from GCP, the trial protocol, or the contract impairing the appropriate conduct of the trial.

Further treatment and follow up of patients affected will occur as described in Section 3.3.4.1.

The investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the third reason).

### 4. TREATMENTS

#### 4.1 INVESTIGATIONAL TREATMENTS

The investigational product has been manufactured by BI Pharma GmbH & Co. KG.

### 4.1.1 Identity of the Investigational Medicinal Products

The characteristics of the test products are given below:

Clinical Trial Protocol


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Table 4.1.1: 1 BI 1015550 9 mg

| Substance: | BI 1015550 |
|-----------------------------|-------------------------------------------|
| Pharmaceutical formulation: | Film-coated tablets |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | 9 mg |
| Posology: | bid |
| Mode of administration: | Oral |

# Table 4.1.1: 2 BI 1015550 18 mg

| Substance: | BI 1015550 |
|-----------------------------|-------------------------------------------|
| Pharmaceutical formulation: | Film-coated tablets |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | 18 mg |
| Posology: | bid |
| Mode of administration: | Oral |

# Table 4.1.1: 3 Placebo matching BI 1015550 9 mg

| Substance: | Placebo matching in size, weight, colour and shape |
|---|---|
| | to BI 1015550 |
| Pharmaceutical formulation: | Film-coated tablets |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | NA |
| Posology: | bid |
| Mode of administration: | Oral |

# Table 4.1.1: 4 Placebo matching BI 1015550 18 mg

| Substance: | Placebo matching in size, weight, colour and shape |
|---|---|
| | to BI 1015550 |
| Pharmaceutical formulation: | Film-coated tablets |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | NA |
| Posology: | bid |
| Mode of administration: | Oral |

## 4.1.2 Selection of doses in the trial and dose modifications

Preclinical in vitro data and indirect target engagement data from Phase I trials support antifibrotic and anti-inflammatory activity of BI 1015550 at plasma concentrations related to the dose of 9 mg bid and 18 mg bid.


#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

target human PDE4B (10.3 nM). Furthermore, Phase I trials in healthy volunteers showed an indirect target engagement, using an ex vivo whole blood assay with an inhibition of LPS-stimulated TNF- $\alpha$  and IFN- $\gamma$  release (anti-inflammatory activity), starting at multiple doses of 6 mg bid.

In the Phase I trials, single doses up to 48 mg and multiple doses up to 18 mg bid with up to 12 weeks of treatment have been evaluated in healthy volunteers and patients with IPF. The maximum tolerated dose was not reached as BI 1015550 was well tolerated. The selected 18 mg dose was tested in a Phase Ic trial (1305-0012) in IPF patients not on background antifibrotic treatment, administered for 4 to 12 weeks. In the Phase II trial (1305-0013), BI 1015550 at 18 mg bid dose was evaluated vs. placebo over a course of 12 weeks in 147 IPF patients, of whom 74 were on a background treatment with antifibrotic (AF group) and 73 without antifibrotic background treatment (non-AF group). This trial showed substantial evidence of treatment benefit of BI 1015550 on FVC change from baseline at 12 weeks in both the AF and non-AF groups [c37065416]. Treatment of BI 1015550 at a dose of 18 mg bid demonstrated an acceptable safety and tolerability in IPF patients over 12 weeks.

In addition, based on population PK/PD analysis of Phase II study 1305-0013 in IPF patients, the FVC response did not change as a function of exposure within the exposure range observed for the BI 1015550 18 mg bid dose given over 12 weeks. This suggested that the maximum effect of BI 1015550 on FVC has been reached with the 18 mg bid dose [c37934954] consistent with the observed clinical stabilization of FVC over the treatment period.

Based on the simulated exposure, 9 mg bid dose provides a sufficient differentiation in the distribution of exposure compared to 18 mg bid dose, supporting that 9 mg and 18 mg bid doses provide wide ranges of plasma exposure to explore dose-response and exposure-response relationship.

IPF and other forms of progressive pulmonary fibrosis are serious debilitating conditions characterized by worsening symptoms and quality of life, progressive loss of lung function, ultimately resulting in respiratory failure, and early death. At the same time, the currently approved antifibrotic treatments have limitations: they do not impact symptoms and cannot stop or reverse fibrosis. Under these circumstances, the highest BI 1015550 dose that is considered safe and well-tolerated (18 mg bid) was selected for the Phase III trials to maximise the potential for efficacy of the treatment, i.e. to preserve lung function and quality of life of patients. In order to provide further dose-response and exposure-response data, a dose of 9 mg bid has been chosen based on available preclinical data on target engagement and simulated exposure assessments, so that both efficacy and safety with this lower dose can be investigated with an expected therapeutic effect. Based on the data from the Phase II trial, demonstrating a stabilization in FVC and an acceptable safety and tolerability profile, these doses seem to provide a reasonable benefit to risk ratio for the patient treatment in this Phase III trial.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4.1.3 Method of assigning patients to treatment groups

After the assessment of all inclusion and exclusion criteria, each eligible patient will be randomized in 1:1:1 ratio to either BI 1015550 9 mg bid, BI 1015550 18 mg bid, or placebo at Visit 2. Randomization (stratified by patient's background AF-treatment at baseline) will be conducted via Interactive Response Technology (IRT). The appropriate medication number(s) will be assigned and documented in the CRF. Note that the medication number is different from the patient number (the latter is generated already during screening via the IRT system).

# 4.1.4 Drug assignment and administration of doses for each patient

During Visit 2, after randomization the patient will begin treatment for at least 52 weeks. The treatment will be assigned by an IRT contact during Visits 2, 4, 5, 6, 7, 8, 9. Patients that are treated in Treatment Period B will be assigned treatment at Visit 10 and the respective visits of Treatment Period B (every 12 weeks). The patient will receive either active treatment at a dose of 9 mg, 18 mg, or placebo. The first dose of BI 1015550 or placebo will be administered to the patient at the end of Visit 2 (Day 1) under direct supervision of the investigator or designee. On the day of any further clinic visit, supervision of administration is not required but the treatment will preferably be administered to the patient during the visit.

Table 4.1.4: 1 Number of IMP kits dispensed at each visit

| Trial visits | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 Treatment Period B |
|---|---|---|---|---|---|---|---|---|---|
| Number of IMP kits dispensed | 2 | 0 | 2 | 2 | 3 | 3 | 3 | 3 | 4* 4 per visit |

<sup>\*</sup> IMP kits will only be dispensed in case Visit 10 is not replaced with the EOT visit.

The trial medication will consist of 2 tablets to be taken orally twice daily. The patient should swallow the trial medication in its entirety (without chewing) with a glass of water ( $\sim$ 250 mL), observing a 12-hour dose interval. The patient should ensure to take the trial medication at the same time every day ( $\pm$ 30 mins), ideally between 6:00 and 11:00 in the morning and between 18:00 and 23:00 in the evening. There are no specific requirements regarding the timing of doses in relation to meals.

If taken around the same time (approximately within an hour), patients on nintedanib or pirfenidone background should take trial medication first, followed by the antifibrotic background medication. A missed dose should be skipped if the time window to the next dose is less than 8 hours. The next dose should be taken as scheduled. If an episode of vomiting happens after medication intake, redose with trial medication is not advised.

After a temporary interruption, trial treatment may be restarted (Section 3.3.4.1).

The investigational product should only be dispensed to participating patients according to the protocol by authorised personnel as documented in the ISF.


c39145241-04

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4.1.5 Blinding and procedures for unblinding

### 4.1.5.1 Blinding

Patients, investigators, central reviewers, and everyone involved in trial conduct or analysis or with any other interest in this double-blind trial will remain blinded regarding the randomized treatment assignments until the database is declared ready for analysis according to the sponsor's SOPs.

At the main analysis database lock (DBL1; see Section 3.1), the sponsor will be unblinded to assess the benefit-risk of both doses of BI 1015550 vs placebo and select the dose with the more favorable benefit-risk profile for the open-label extension trial. Patients, investigators, and other site personnel will remain blinded to the randomized treatment assignment until the end of the trial.

The trial medication is identified by a medication code number and packaging is identical. The color, size, and shape of the respective 9 mg and 18 mg BI 1015550 and the matching placebo tablets will be indistinguishable. The access to the randomization code will be kept restricted until its release for analysis at DBL1. Further details regarding the timepoint of unblinding the database for analysis is documented in the TSAP.

The randomization codes will be provided to bioanalytics before DBL1 to exclude placebo or comparator samples from the PK analysis. Bioanalytics will not disclose the randomization code or the results of their measurements until DBL1.

A dedicated database snapshot (not a partial DBL) will be generated prior to DBL1, after all patients have completed the last PK visit (i.e. Week-26 visit), to allow for development and refinement of the population PK model (for "fast-track" PK analysis). Details of the analysis will be defined in the PK/PD analysis plan. In addition, the data will be used for front-loading of descriptive analysis for PK. Only personnel involved in the population PK and descriptive analyses will be granted access to the unblinded PK data before DBL1, whereas the trial team and all other functions not involved in the population PK and PK descriptive analyses will remain blinded (details will be provided in a separate logistics and access plan). The analysis plan for the population PK analysis will be finalized and signed prior to this dedicated database snapshot.

No formal interim report will be generated for the population PK analysis. The final PK and PK/PD analyses will be reported separately from the clinical trial report (CTR) after DBL1.

The external DMC will review unblinded data upon request and for the futility interim analysis as described in Section 7.2.8, and only under conditions that ensure that patients, investigators, everyone involved in trial conduct or analysis, and anyone with any other participation in this double-blind trial will remain blinded.

If the 9 mg dose is considered futile based on the respective interim analysis (see Section 7.2.8), the patients will be re-assigned to the 18 mg dose in a blinded manner and the 18 mg dose will be given at the next scheduled visit.

# c39145241-04 Clinical Trial Protocol

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


# 4.1.5.2 Unblinding and breaking the code

Emergency unblinding will be available to the investigator via IRT. It must only be used in an emergency situation when the identity of the trial drug must be known to the investigator in order to provide appropriate medical treatment or otherwise assure safety of trial participants. The reason for unblinding must be documented in the source documents and/or appropriate CRF page.

To avoid unblinding of the study team through drug safety reports which are to be unblinded as per regulatory requirements, a procedure will be maintained to keep codebreaking in these cases invisible to study team.

Due to the requirements to report Suspected Unexpected Serious Adverse Reactions (SUSARs), it may be necessary for a representative from BI's Pharmacovigilance group to access the randomization code for individual patients during trial conduct. The access to the code will only be given to authorised pharmacovigilance representatives for processing in the PV database system and not be shared further.

# 4.1.6 Packaging, labelling, and re-supply

The trial medication will be tablets containing 9 mg of BI 1015550, 18 mg of BI 1015550, or the respective matching placebo in a double-dummy design. Each trial medication kit is packaged in a child-resistant tamper-evident wallet containing 112 tablets of 9 mg or 18 mg BI 1015550 or the respective matching placebo. Wallets will cover 4 weeks of treatment.

Each wallet will be labelled with a multi-language booklet or country specific label according to the requirements of the participating countries.

The investigational medicinal products will be provided by BI or a designated CRO. They will be packaged and labelled in accordance with the principles of Good Manufacturing Practice (GMP). Re-supply to the sites will be managed via an IRT system, which will also monitor expiration dates of supplies available at the sites.

For details of packaging and the description of the label, refer to the ISF.

# 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area according to the recommended storage conditions on the medication label. A temperature log must be maintained for documentation.

If the storage conditions are found to be outside the specified range, the Clinical Research Associate (CRA, as provided in the list of contacts) must be contacted immediately.

All unused trial medication must be returned to the Sponsor or appointed Contract Research Organization (CRO). Receipt, usage, and return must be documented on the respective forms/IRT system. Account must be given for any discrepancies.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4.1.8 **Drug accountability**

The investigator or designee will receive the investigational drugs delivered by the sponsor or delegate when the following requirements are fulfilled:

- Approval of the clinical trial protocol by the IRB/ethics committee, HA/RA if applicable.
- Availability of a signed and dated clinical trial contract between the sponsor or delegate and the investigational site,
- Approval/notification of the regulatory authority, e.g. competent authority,
- Availability of the *curriculum vitae* of the Principal Investigator,
- Availability of a signed and dated clinical trial protocol,
- Availability of the proof of a medical license for the Principal Investigator,
- Availability of FDA Form 1572 (if applicable).

Investigational drugs are not allowed to be used outside the context of this protocol. They must not be forwarded to other investigators or clinics. Patients should be instructed to return unused investigational drug.

The investigator or designee must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each patient, and the return to the sponsor or warehouse / drug distribution centre or alternative disposal of unused products. If applicable, the sponsor or warehouse/drug distribution centre will maintain records of the disposal.

These records will include dates, quantities, batch/serial numbers, expiration ('use-by') dates, and the unique code numbers assigned to the investigational medicinal product and trial patients. The investigator or designee will maintain records that document adequately that the patients were provided the doses specified by the Clinical Trial Protocol (CTP) and reconcile all investigational medicinal products received from the sponsor. At the time of return to the sponsor and/or appointed CRO, the Investigator or designee must verify that all unused or partially used drug supplies have been returned by the clinical trial patient and that no remaining supplies are in the investigator's possession.

# 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

# 4.2.1 Other treatments and emergency procedures

There are no special emergency procedures to be followed.

Temporary treatment interruption is allowed to manage adverse events. All efforts should be made to re-start IMP after resolution of the adverse event according to the Investigator's assessment.

Please find management guidance for specific adverse events below:

### Diarrhea

Depending on the intensity of the events, the following management strategies are recommended:

• Counselling of patients, including potential diet modifications


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Monitor and maintain adequate hydration
- Treatment with loperamide or other antidiarrheal medications
- For patients on antifibrotic medication, management strategies (e.g., dose reduction and/or temporary interruption) as described in the respective prescribing information should be followed

Temporary interruption of trial treatment can be considered, and trial treatment may be restarted when the patient has recovered according to investigator's assessment.

# Severe infections (CTCAE >2), serious infections, opportunistic or mycobacterium tuberculosis infections

Treatment of the infection should be initiated promptly according to local standard of care. No further trial medication should be administered until the active infection has resolved and trial treatment may be restarted when the patient has recovered according to investigator's assessment.

#### Malignancies

In case of occurrence of malignant neoplasm other than appropriately treated basal cell carcinoma or in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix, the investigator should <u>permanently</u> discontinue trial treatment. Diagnostics and treatment must be initiated according to local standard of care.

# Vasculitis

In case of events suspicious for vasculitis, trial treatment will be discontinued. A thorough work-up has to be initiated including at least but not limited to

- appropriate imaging, including angiography
- biopsy if possible
- appropriate laboratory screening, including measurements of vasculitis markers at the central lab, see Section <u>5.2.3.3</u>. In addition, an analysis of the previously collected and stored samples (baseline and/or Visit 10 samples) will need to be requested and considered.
- thorough documentation of all reported symptoms

Referral to a vasculitis expert is recommended. If required, vasculitis treatment should be initiated according to standard of care. If thorough evaluation does not confirm a causal relationship between trial medication and the event, trial treatment may be restarted based on the investigator's medical judgement.

# New onset of severe depression or suicidality

In case of new onset of severe depression defined as HADS >14 or the patient exhibits any suicidal behaviour or serious suicidality ideation defined as type 4 or 5 in the C-SSRS interview, trial treatment has to be discontinued. Referral to a psychiatrist for further diagnoses and initiation of treatment is recommended.

In case of severe depression: If thorough evaluation does not confirm a causal relationship between trial medication and the event, and the patient has recovered, trial treatment may be restarted based on the investigator's medical judgement (in case of new-onset of suicidality treatment has to be permanently discontinued).

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.2.2 Restrictions

c39145241-04

# 4.2.2.1 Restrictions regarding concomitant treatment

# Treatment with antifibrotic medication (nintedanib, pirfenidone)

# AF group:

Patients who are on a stable dose of marketed antifibrotic treatment (nintedanib or pirfenidone) should plan to remain on this treatment for the duration of the trial. Interruption and/or dose reductions of the background antifibrotic medication are left at the discretion of the investigator, e.g. to manage side effects in line with the respective prescribing information. Combined treatment with nintedanib plus pirfenidone is not allowed.

# Non-AF group:

For patients not receiving nintedanib or pirfenidone in the 8 weeks prior to study entry, nintedanib and pirfenidone are restricted medications during the full duration of the blinded treatment period. Nintedanib or pirfenidone should not be initiated in the first 12 weeks of trial treatment. After that timeframe, initiation of nintedanib or pirfenidone is only allowed as rescue medication in case of disease worsening defined as disease under study progression and/or IPF exacerbation (by investigator judgement).

# Immunomodulatory treatment

Immunomodulatory medications (other than oral corticosteroids) or prednisone >15 mg/day or equivalent should not be started for respiratory indications during the screening or treatment period. However, prednisone >15 mg/day or equivalent can be prescribed during the treatment period in case of (suspected) acute IPF exacerbation.

# Other restricted concomitant medication

While enrolled in this trial, patients must not participate in another investigational drug or device trial or receive other investigational treatment(s).

Stem cell therapy for the treatment of pulmonary fibrosis is not allowed.

Treatment with non-selective PDE inhibitors as well as PDE4 inhibitors is not allowed.

Potent CYP3A4 inhibitors should not be administered during the screening and trial treatment periods. If short-term treatment with potent CYP3A4 inhibitor is needed (e.g., Paxlovid for the treatment of COVID-19; clarithromycin for antibiotic treatment), IMP should be temporarily discontinued (see Section 3.3.4.1 about conditions to re-introduce IMP). Non-exhaustive lists of potent CYP3A inhibitors and PDE inhibitors are provided in the Appendix 10.4.1.

c39145241-04


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.2.2.1: 1 Restrictions regarding concomitant treatment

| Medication | Prior to Study <sup>1</sup> | Screening Period | Treatment Period A and B | Follow up<br>period |
|---|---|---|---|---|
| Potent CYP3A inhibitors | Not permitted | Not permitted | Not permitted <sup>2</sup> | Permitted |
| Stem cell therapy for the treatment of pulmonary fibrosis | Not permitted | Not permitted | Not permitted | Not permitted |
| PDE4 and non-selective<br>PDE inhibitors | Not permitted | Not permitted | Not permitted | Not permitted |
| Immunomodulatory medications (other than oral steroids) or Prednisone >15mg/day or equivalent <sup>3</sup> used for respiratory/ pulmonary reasons | Permitted <sup>4</sup> | Not permitted | Not permitted <sup>5</sup> | Permitted |

- 1. Duration of restriction before screening see exclusion criteria Section 3.3.3
- 2. If any short-term treatment with potent CYP3A4 inhibitor is needed, IMP should be temporarily discontinued
- 3. Inhaled, intra-nasal, and topical corticosteroids are allowed
- 4. Referring to historical episodes of intake, permitted unless the treatment is ongoing at time of Visit 1
- 5. Prednisone >15 mg/day or equivalent can be prescribed during the treatment period in case of (suspected) acute IPF exacerbation.

# 4.2.2.2 Restrictions on diet and lifestyle

Patients should refrain from drinking grapefruit juice during the duration of the trial.

Patients should refrain from smoking or vigorous activity 1 hour before performing spirometry assessments.

# 4.2.2.3 Contraception requirements

Women of childbearing potential (WOCBP)<sup>2</sup> must use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly throughout the trial, and for a period of at least 7 days after last trial drug intake. A list of contraception methods meeting these criteria is provided below and in the patient information.

\_

<sup>&</sup>lt;sup>2</sup> A woman is considered of childbearing potential (WOCBP), i.e.fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Acceptable highly effective methods of contraception include:

- Non-oral hormonal methods of contraception associated with inhibition of ovulation:
  - o Intravaginal or transdermal combinations of estrogen and progestogen
  - o Injectable or implantable progestogen
- Oral hormonal contraceptives together with one barrier method (e.g. condom) to account for the risk of potentially reduced efficacy of the OCs in the event of severe vomiting and diarrhea. In case of vomiting or diarrhea, instructions in the label of the OC should be followed in addition. In case of prolonged (>48h) or repeated vomiting/diarrhea, the use of an alternative highly effective contraceptive measure should be considered
- Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion
- Vasectomised sexual partner with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate, provided that partner is the sole sexual partner of the study participant
- Complete abstinence from male-female sex when this is in line with the preferred and usual lifestyle of the study participant. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods; declaration of abstinence for the duration of exposure to study drug; and withdrawal are not acceptable.

#### 4.3 TREATMENT COMPLIANCE

Patients are requested to bring all remaining trial medication including empty package material with them when attending visits.

Based on tablet counts, treatment compliance will be calculated as shown in the formula below. Compliance will be verified by the CRA authorised by the sponsor or delegate.

Treatment compliance (%) =  $\frac{\text{Number of tablets actually taken} \times 100}{\text{Number of tablets which should have been taken as directed by the investigator}}$ 

If the number of doses taken is not between 80-120%, site staff will explain to the patient the importance of treatment compliance.

# 5. ASSESSMENTS

# 5.1 ASSESSMENT OF EFFICACY

#### 5.1.1 FVC

Spirometry measurements will be performed according to ATS/ERS 2019 guideline [R20-2419]. FVC will be assessed using standardised spirometry equipment which will be provided centrally with supplies of precalibrated disposable flow sensors. These sensors meet International Organization for Standardization (ISO) 26782 standards, but with a maximum


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

permissible accuracy error of  $\pm 2.5\%$ , in accordance with the American Thoracic Society (ATS)/European Respiratory Society (ERS) Technical Statement [R20-2419]. As such there is no need to conduct daily calibration prior to use. Only these spirometers are to be used for this trial. Spirometry performance will be centrally reviewed.

Spirometry will be conducted with the patient in a seated position. It is preferable that the same trained individual performs the PFTs for a given patient. The best of three efforts will be defined as the highest FVC obtained on any of three blows meeting the 2019 ATS/ERS criteria (with a maximum of eight attempts). Predicted normal values will be calculated according to GLI (Global Lung Initiative).

Efforts should be made to schedule the spirometric measurements at approximately the same time of the day, at least within the same half-day (morning vs. afternoon), with reference to baseline measurement (Visit 2). On days of study visits, patients should be encouraged to refrain from vigorous activity and smoking within 1 hour of pulmonary function testing. If treated with bronchodilators, washout according to Appendix 10.1 should be advised before spirometry and documented in the source documents.

Spirometry results will be electronically transmitted. To ensure the quality of the primary endpoint measurement, a central spirometry review is put in place to provide feedback to the investigational site and the CRA on the quality of the data received from the site. In case unacceptable results for FVC/FEV1 at V1 or FVC at V10 are obtained after the review, the patient must be reassessed.

Further instructions regarding FVC measurements will be provided in the ISF.

# Optional assisted home spirometry measurements

At selected sites with respective setup, assisted home spirometry can be conducted intermittently during the trial and as a fallback/contingency option.

For the assisted home spirometry, patients may be using a handheld spirometer (iSpiro) together with a mobile phone with the installed iSpiro App provided by site. Training of the patients on the use of the iSpiro device and App can be done at any visit, ideally at Visit 2 or Visit 3 together with a first recording. During the treatment phase, the iSpiro device and the respective phone with the App will be provided to the patient upon decision of the investigator in order to perform an assisted (via video call) home spirometry either at unscheduled visits or as a fallback solution if the patient is unable to get to the site for the scheduled visit.

These home spirometry measurements will not replace the onsite FVC measurement at Visit 2 (Day 1), Visit 5 (Week 12), Visit 7 (Week 26), Visit 10 (Week 52) and the visit for EOT; every effort should be made to obtain an onsite spirometry within the planned visit window.

#### **5.1.2** Exacerbation of IPF

The most recent definition of acute IPF exacerbation will be used [P16-06899].


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Such events will be defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality with all of the following:

- Acute worsening or development of dyspnea typically less than 1 month duration.
- Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with IPF.
- Deterioration not fully explained by cardiac failure or fluid overload.

This event must be reported as adverse event in the category "acute exacerbation of disease under investigation".

Events that are clinically considered to meet the definition of acute IPF exacerbation but fail to meet all diagnostic criteria above due to missing CT data must be reported as "suspected acute exacerbations of disease under investigation" (as long as this assessment persists). Both confirmed and suspected cases will be considered for the endpoint evaluation.

#### 5.1.3 Time to death

Time to death will be based either on the date of death on the AE report for patients with AEs leading to death or will be based on the information from the vital status assessment.

# 5.1.4 Hospitalization due to respiratory cause

Hospitalization due to respiratory cause will be collected on a specific non-elective hospitalization CRF page. The CRF page will capture the date of hospitalization, whether the non-elective hospitalization was due to respiratory cause, and the primary admission diagnosis.

# **5.1.5** Patient-Reported Outcome Questionnaires

The patient will complete patient-reported outcome (PRO) questionnaires preferably according to the prespecified order defined hereafter:

Questionnaires completed by patient:

- 1. Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (L-PF)
- 2. EuroQol 5-Dimensional quality of life Questionnaire (EQ-5D)
- 3. Hospital Anxiety and Depression Scale (HADS, Section <u>5.2.5.2</u>)
- 4. Patient's Global Impression of Severity (PGIS) for Cough, Shortness of Breath, and Fatigue

Patients may complete these questionnaires at site or at home if they so choose to. The questionnaires may be completed either on paper versions, with site provided tablet, a mobile phone provided centrally or via an App downloaded to patient's personal device.

Patients are asked to be in a quiet area/room prior to any other trial related examination and should complete these questionnaires without any help from or interpretation by other people. If the patient is too sick to complete the questionnaires him/herself but is able to reply verbally, a member of the study team should read the instructions, questions, and response options aloud to the patient and collect the patient's verbal response in as neutral and


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

unbiased a manner as possible. If this is not possible either, the questionnaires are not to be completed.

If done at home, patient should compile the questionnaire preferably the same half-day as the intended scheduled site visit (morning or afternoon) and within the last 3 days before the site visit.

For the compilation of paper questionnaires, the site personnel will check the patient questionnaires for completeness prior to the patient leaving the site, but the response to each item will not be tampered with, and a patient should not be influenced in any manner on how to respond to the question. Scores will be entered into the eCRF by the site-personnel. For patient-reported outcomes compiled on electronic devices, completeness and consistency checks will be programmed into the App and no further check by site personnel is needed. Data from these patient outcome reports will be electronically submitted.

# 5.1.5.1 Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (L-PF)

The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item questionnaire with two modules: 1) Symptoms (23 scored items plus 5 oxygen questions) and 2) Impacts (21 items). L-PF was developed with the input of patients with pulmonary fibrosis (PF) and thus is intended to capture perceptions specific to PF patients.

The Symptoms module yields three domain scores: 1) dyspnea, 2) cough, and 3) fatigue as well as a total Symptoms score. There are 5 additional questions pertaining to oxygen use at the end of the Symptoms module. The Impacts module yields a single Impacts score. Symptoms and Impacts scores are summed to yield a total L-PF score. Scoring is performed as a summary score, the mean of the dimension ratings multiplied by 100. For details, please refer to the TSAP.

The L-PF Symptoms and Impact Questionnaire (Appendix <u>10.2.1</u>) will be self-administered by the patient at visits indicated in the <u>flow chart</u>.

# 5.1.5.2 EuroQol 5-Dimensional quality of life Questionnaire (EQ-5D)

The EQ-5D was developed by the European Quality of Life Group (EuroQol Group) and is a standardized instrument for use as a measure of health outcomes [R96-2382]. The version used in this trial is the new five-level version (EQ-5D-5L).

The questionnaire essentially consists of 2 pages. The first page is the descriptive system with 5 questions to the patient's health state today. Each question captures one dimension of health (e.g. mobility, self-care) and has five levels to answer. The second page records the patient's self-rated health status of today on a vertical graduated (0 to 100) visual analogue scale.

The EQ-5D (Appendix 10.2.2) will be self- administered by the patient at visits indicated in the flow chart.

c39145241-04

 Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.1.5.3 Patient's Global Impression of Severity (PGIS) of Cough, Shortness of Breath and Fatigue

The PGIS questionnaire will ask the patient to think about their cough and reflect how it was in the past 7 days: "recall whether you have had a cough and if so, how frequently it has occurred, how severe it has been, and whether cough has affected how you feel and how you function in your daily life. Considering all these, please rate the severity of your cough over the last 7 days by placing a tic in the one box corresponding to your response: not present, very mild, mild, moderate, severe, and very severe."

The patient will be asked to think about shortness of breath and reflect on the last 7 days: "call to mind how severe it has been and whether shortness of breath has affected how you feel and how you function in your daily life. Considering all these, please rate the severity of your shortness of breath over the last 7 days by placing a tic in the one box corresponding to your response: not present, very mild, mild, moderate, severe, and very severe."

If applicable, the patient will be asked to complete the PGIS fatigue to assess the patient's severity of fatigue. The measure consists of 1 item/question asking patients to rate their severity of fatigue on a 5-point Likert scale ranging from "no symptoms" to "very severe" including a recall "over the past 24 hours".

The PGIS (Appendix 10.2.4) will be self- administered by the patient at visits indicated in the flow chart.

#### 5.1.6 **DLCO**

The site will use its own carbon monoxide diffusion capacity (DLCO) equipment and conduct all measurements with the same DLCO equipment in case that several devices are available at the site. Single-breath DLCO measurement will be carried out according to the ATS/ERS guideline on DLCO measurements [R06-2002]. Raw data (gas mixture, equation used for prediction of normal, further adjustments made if so) must be traced.

Two acceptable DLCO measurements and the corresponding alveolar volume will be taken at time points indicated in the flow chart. Both acceptable DLCO measurements will be recorded. Maneuvers will be demonstrated before beginning of the test, and the patient will be carefully instructed.

Predicted DLCO value will be corrected for hemoglobin (Hb). The site has to enter the unadjusted predicted DLCO result without Hb correction in the eCRF. This value will be adjusted for the most recent Hb value.

At Visit 1, the most recent Hb value (ideally on the same day) will be entered into the eCRF to correct the DLCO value. During subsequent visits, Hb values will be transferred from the central lab and corrections will be done automatically (not visible into the eCRF).

For predicted normal values, different sites may use different prediction formulas, based on the method used to measure DLCO. In any case, the calculation method used must be in compliance with the ATS/ERS guideline on DLCO measurements [R06-2002] and the prediction formula appropriate for that method.

#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Predicted DLCO corrected for Hb**, with Hb expressed in g·dL-1 [R06-2002], will be calculated in the eCRF as:

- Males: DLCO predicted for Hb = DLCO predicted  $\times [1.7\text{Hb} / (10.22 + \text{Hb})]$
- Females: DLCO predicted for Hb = DLCO predicted  $\times [1.7\text{Hb} / (9.38 + \text{Hb})]$

**Percent predicted DLCO corrected for Hb** (unit: %) at Visit 1 will be calculated in the eCRF with the following formula:

Percent predicted DLCO corrected for Hb = (Mean value of two DLCO measurements, expressed in mmol/min/kPa) / Predicted DLCO corrected for Hb) \* 100

For each patient, spirometry testing and DLCO should always start at approximately the same time of day. DLCO must be performed after spirometry on the same day.

#### 5.2 ASSESSMENT OF SAFETY

# 5.2.1 Physical examination

A physical examination will be performed at the time points specified in the <u>flow chart</u>. It includes at a minimum general appearance, neck, lungs, cardiovascular system, abdomen, extremities, and skin. Measurements of height and body weight will be performed at the time points specified in the flow chart. The results must be included in the source documents available at the site.

All abnormal findings at baseline will be recorded on the Baseline Condition eCRF page. New abnormal findings or worsening of baseline conditions detected at the subsequent physical examinations, if judged clinically relevant, will be recorded as adverse events on the appropriate eCRF page.

# 5.2.2 Vital signs

Vital signs will be evaluated at the time points specified in the <u>flow chart</u>, prior to blood sampling.

This includes systolic and diastolic blood pressure and pulse rate (electronically or by palpation count for 1 minute) in a seated position after 5 minutes of rest. Additionally, SpO2 will be measured via pulse oximetry.

The results must be included in the source documents available at the site.

# 5.2.3 Safety laboratory parameters

Safety laboratory parameters to be assessed are listed in <u>Table 5.2.3.1: 1</u>. For the sampling time points please see the flow chart.

All analyses will be performed by a central laboratory, the respective reference ranges will be provided in the ISF.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Patients do not have to be fasted for the blood sampling for the safety laboratory.

Instructions regarding sample collection, sample handling/processing and sample shipping are provided in the Laboratory Manual in the ISF.

The central laboratory will send reports to the investigator. It is the responsibility of the investigator to evaluate the laboratory reports. Clinically relevant abnormal findings as judged by the investigator will be reported as adverse events (please refer to Section 5.2.6).

In case the criteria for hepatic injury are fulfilled, a number of additional measures will be performed (please see Section <u>5.2.6.1.4</u> and the DILI Checklist provided in the eDC system). The amount of blood taken from the patient concerned will be increased due to this additional sampling.

The central laboratory will transfer the results of the analysis to the sponsor or delegate.

# 5.2.3.1 Routine safety lab tests

Table 5.2.3.1: 1 Safety laboratory tests

| Functional lab group | Test name |
|---|---|
| Hematology | Hematocrit |
| | Hemoglobin |
| | Red blood cells (RBC) |
| | White blood cells (WBC) |
| | Platelet count |
| | MCV |
| | MCH |
| | MCHC |
| | RDW |
| Automatic WBC differential | Neutrophiles total |
| (relative and absolute) | Lymphocytes total |
| | Eosinophiles |
| | Basophiles |
| | Monocytes |
| | Lymphocytes |
| Manual differential WBC (if automatic differential | Polymorphnuclear neutrophils (segs), band |
| WBC is abnormal) | neutrophils (stabs), eosinophils, basophils, |
| | monocytes, lymphocytes |
| Coagulation | Activated partial thromboplastin time (aPTT) |
| | Prothrombin Time (PT) |
| | INR |
| Enzymes | Aspartate aminotransferase (AST) |
| | Alanine aminotransferase (ALT) |
| | Alkaline phosphatase (AP) |
| | Gammaglutamyl transferase (GGT) |
| | Creatine kinase (CK) |
| | Lipase |
| | Amylase |
| Substrates | Glucose |
| | Creatinine |


**Clinical Trial Protocol** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Functional lab group | Test name |
|---|---|
| | Urea Nitrogen |
| | Uric Acid |
| | Total bilirubin |
| | Direct bilirubin |
| | Total protein |
| | Albumin |
| | Globulin |
| | Albumin / Globulin ratio |
| | C-Reactive Protein (CRP) |
| | Total cholesterol |
| Electrolytes | Calcium |
| | Sodium |
| | Potassium |
| | Chloride |
| | Phosphate |
| Serum Pregnancy test (only for female patients of childbearing potential) at screening (V1) and at any visit where urine pregnancy test is positive | Human Serum Chorionic Gonadotropin |
| Urinalysis (qualitative determination) | Urine nitrite |
| , | Urine protein |
| | Urine glucose |
| | Urine ketone |
| | Urine bilirubin |
| | Urine hemoglobin ( detects erythrocytes) |
| | Urine leukocyte esterase (detects leucocytes) |
| | Urine pH |
| | Specific gravity |
| Urine sediment (microscopic examination if | Only positive findings will be reported (e.g. presence |
| erythrocytes, leukocytes nitrite or protein are | of sediment bacteria, casts in sediment, squamous |
| abnormal in urine) | epithelial cells, erythrocytes, leukocytes) |
| Urine Pregnancy test (only for female patients of childbearing potential) at V2 and following visits | Human Chorionic Gonadotropin in the urine |

eGFR will be analyzed and calculated by the central laboratory at the same timepoints as other safety laboratory parameters (refer to <u>flow chart</u>). eGFR will be calculated by using the CKD-EPI formula and using the Jaffe assay for serum creatinine measurement, IDMS standardized.

#### 5.2.3.2 Infection serology

The following lab tests for infection serology will be performed as indicated in the flow chart:

- Hepatitis B surface antigen (qualitative) and Hepatitis B core antibody (qualitative)
- HBV-DNA PCR (quantitative), which should be conducted if Hepatitis B core antibody is positive and Hepatitis B surface antigen is negative
- Hepatitis C antibodies (qualitative), where a positive Hep C antibodies test result should be confirmed by PCR
- HIV-1 and HIV-2 antibody (qualitative)

c39145241-04

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• IGRA-T (e.g. QuantiFERON®-TB Gold IT Test, provided by central lab): If the first QuantiFERON®-TB-Gold Plus (or if applicable, T-Spot®) test result is undetermined, a retest should be performed.

If the retest QuantiFERON®-TB-Gold Plus test result is undetermined, a PPD skin test should be performed.

For specific countries (e.g. Japan): T-Spot® TB test may be performed at local labs instead of QuantiFERON®TB test

In case of positive TB test, further diagnostic work up to confirm/exclude the diagnosis of latent or active is needed (documentation on respective eCRF page).

# 5.2.3.3 Immunological vasculitis markers

At Visit 2, Visit 10 and in case of a suspected vasculitis an additional blood sample will be taken. It will be stored and analyzed for the following immunological vasculitis markers:

- MPO-ANCA
- PR3-ANCA
- IL-6
- antiglomerular basement membrane (GBM) antibodies
- anti-Clq antibodies (immune complex-associated small-vessel vasculitis)
- rheumatoid factor
- antinuclear antibodies
- complement C3, C4, CH 50, anti-C1q antibodies.

Due to stability matter during storage, ANCA markers (MPO-ANCA and PR3-ANCA) from Visit 2 and Visit 10 are analyzed upon receipt, but investigators will not receive these results as it could influence their judgement regarding a suspected vasculitis. The rest of the analysis of immunological vasculitis markers is performed if an unscheduled "Vasculitis event" is collected. In this situation, the site will receive the result for all vasculitis markers previously performed (from V2 and V10 if already done) and from the unscheduled "Vasculitis event" kit. These results are shared by the trial team to the site via the CRA.

# 5.2.4 Electrocardiogram

The 12-lead ECGs must be administered by a qualified technologist and results will be recorded as scheduled in the <u>flow chart</u>. The investigator or a designee will evaluate whether the ECG is normal or abnormal and assess clinical relevance. ECGs may be repeated for quality reasons and a repeated recording used for analysis.

Additional ECGs may be recorded for safety reasons. Dated and signed printouts of ECG with findings should be documented in patient's medical record.

Clinically relevant abnormal findings will be reported either as baseline condition (if identified at the screening visit) or otherwise as AEs and will be followed up and / or treated as medically appropriate.

c39145241-04

 Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.2.5 **Other Safety parameters**

#### 5.2.5.1 Suicidal risk (C-SSRS)

Prospective monitoring will be conducted throughout this trial using the Columbia-Suicide Severity Rating Scale (C-SSRS).

The C-SSRS is a semi-structured, investigator-rated interview, developed by clinical experts in cooperation with the FDA, assessing both suicidal behavior and suicidal ideation. It does not give a global score but provides some categorical and some severity information specifically for behaviour and ideation.

The C-SSRS has been widely used in large multinational clinical trials. The C-SSRS will be administered at the screening visit (using the 'screening/baseline' version) with the aim to exclude patient's suicidal ideation type 4 to 5 within the preceding 3 months or at Visit 1 or any suicidal behaviour in the past 2 years. The lifetime history of suicidal ideation and behaviour will also be recorded.

After Visit 1, the assessment 'since last visit' will be performed at each clinic visit ('since last visit' version).

Appendix 10.3 details how the C-SSRS will be assessed.

C-SSRS results will be reported in terms of AEs as described in Section 5.2.6.2.

#### 5.2.5.2 Depression and anxiety

Prospective monitoring using the Hospital Anxiety and Depression Scale (HADS).

This questionnaire is patient friendly and easy to use and takes less than 5 minutes for completion. The questionnaire comprises seven questions for anxiety and seven questions for depression that are scored separately. Cut-off scores are available for quantification: The HADS questionnaire has been validated in many languages, countries and settings including general practice and community settings and is one of the tools recommended by National Institute for Health and Care Excellence (NICE) for diagnosis of depression and anxiety and is included in the American Thoracic Society's list of patient-reported outcome measures for use in ILD [R22-1857, R22-1856]. The HADS (Appendix 10.2.3) will be self-administered.

#### 5.2.6 Assessment of adverse events

#### 5.2.6.1 Definitions of AEs

#### 5.2.6.1.1 Adverse event

An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether considered related or not.

The following should also be recorded as an AE in the CRF and BI SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination and laboratory test results, if they are judged clinically relevant by the investigator.

If such abnormalities already exist prior to trial inclusion, they will be considered as baseline conditions and should be collected in the eCRF only.

# Adverse event report for diarrhea events

In case of events of diarrhoea the following definitions should be followed: Diarrhoea is defined ≥3 loose/liquid stools per day (WHO definition) Diarrhoea episode = 2 diarrhoea episodes are separated by at least 7 days without any diarrhoea

# Adverse event report for depression and anxiety

AE reporting based on the Hospital Anxiety and Depression Scale (HADS): new onset of moderate depression, defined as HADS subscore of >10, has to be reported as AE; new onset of moderate anxiety, defined as HADS subscore of >10, has to be reported as AE. HADS subscore of  $\leq$ 10 should only be reported as an AE if clinically relevant. See Section 5.2.6.1.4 for reporting of AESI based on HADS.

#### 5.2.6.1.2 Serious adverse event

A serious adverse event (SAE) is defined as any AE, which fulfils at least one of the following criteria:

- results in death,
- is life-threatening, which refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe,
- requires inpatient hospitalisation or prolongation of existing hospitalisation
- results in persistent or significant disability or incapacity,
- is a congenital anomaly / birth defect,
- is deemed serious for any other reason if it is an important medical event when based on appropriate medical judgement which may jeopardise the patient and may require medial or surgical intervention to prevent one of the other outcomes listed in the above definitions. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse.

#### For Japan only:

An event that possibly leads to disability will be handled as 'deemed serious for any other reason' and, therefore, reported as an SAE.

c39145241-04


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5.2.6.1.3 AEs considered "Always Serious"

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as defined above.

The latest list of "Always Serious AEs" can be found in the eDC system. A copy of the latest list of "Always Serious AEs" will be provided upon request. These events should always be reported as SAEs as described in Section 5.2.6.1.2.

Every occurrence of cancer of new histology must be classified as a serious event regardless of the time since the discontinuation of the trial medication and must be reported as described in Section <u>5.2.6.1.2</u>, subsections "AE Collection" and "**AE reporting to sponsor and timelines**".

# SAE reporting in case of Suicidal Risk assessed by the C-SSRS

All C-SSRS reports of suicidal ideation type 4 and 5 and all reports of suicidal behavior must be reported as separate SAEs by the investigator.

For 'self-injurious behavior, no suicidal intent' (type 11) standard AE/SAE reporting rules are to be applied.

For each negative report (Suicidal ideation type 1, 2, or 3) after the start of the trial, the investigator is to decide based on clinical judgement whether it represents an adverse event (AE) as defined in the protocol, and if it is considered an AE then it must be reported accordingly.

# 5.2.6.1.4 Adverse events of special interest

The term adverse events of special interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.2.6.2.2.

The following are considered as AESIs:

- Potential severe DILI
- Vasculitis
- Severe infections (CTCAE >2), serious, opportunistic, or mycobacterium tuberculosis infections (refer to Appendix 10.5)
- New onset of severe depression, defined as HADS subscore >14
- New onset of severe anxiety, defined as HADS subscore >14

Management of specific AEs is described in Section <u>4.2.1</u>, specific additional procedures to be performed in case of a suspected AESI are described in this section:


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Potential Severe DILI

c39145241-04

A potential severe Drug Induced Liver Injury (DILI) that requires follow-up is defined by the following alterations of hepatic laboratory parameters:

- An elevation of AST (Aspartate Aminotransferase) and/or ALT (Alanine Aminotransferase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or in samples drawn within 30 days of each other, or
- ALT and/or AST elevations  $\geq$ 10-fold ULN.

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the "DILI checklist" provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the investigator should make sure these parameters are analyzed, if necessary, in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

For patients with abnormal aminotransaminase levels between >1 and <3 x ULN at baseline:

- An elevation of AST and / or ALT ≥3-fold the baseline value combined with an elevation of bilirubin ≥2-fold ULN or ≥2-fold the baseline value (if bilirubin is elevated at baseline), measured in the same blood sample, or in samples drawn within 30 days of each other; or;
- Aminotransferase elevations ≥5-fold the baseline value.

# Vasculitis events

In this trial protocol vasculitis is defined as any event term included in the MedDRA SMQ Vasculitis (broad). This includes clinical and pathological features related to primary or secondary vasculitis syndromes and involving any type, size, and location of blood vessels. The investigator should monitor for any signs and symptoms of vasculitis at all times and specifically as part of the AE questioning.

In case of (suspected) events of vasculitis, further work-up and management as outlined in Section 4.2.1 has to be followed, including biopsy, appropriate imaging/angiography, laboratory measures (e.g. additional lab sample for immunological and further inflammation markers). Details will be collected on a dedicated eCRF page and events will referred for adjudication to an independent adjudication committee.

# 5.2.6.1.5 Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on CTCAE grading (see ISF for grading of specific events)

- Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age appropriate instrumental activities of daily living

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living.
- Grade 4: Life-threatening consequences; urgent intervention indicated.
- Grade 5: Death related to AE.

# 5.2.6.1.6 Causal relationship of AEs

Medical judgement should be used to determine the relationship between the adverse event and the BI investigational compound, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the trial drug.
- The event is known to be caused by or attributed to the drug class.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the event is reproducible when the drug is re-introduced.
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is reduced).

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pretreatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the trial drug concerned).
- Continuation of the event despite the withdrawal of the medication, considering the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.
- There is an alternative explanation, e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned.
- Disappearance of the event even though the trial drug treatment continues or remains unchanged.

# 5.2.6.2 Adverse event collection and reporting

#### 5.2.6.2.1 AE Collection

The investigator shall maintain and keep detailed records of all AEs in the patient files.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following must be collected and documented on the appropriate CRF(s) by the investigator:

- From signing the informed consent onwards until the individual patient's end of trial (= the End of Trial (EOS) visit): all AEs (serious and non-serious) and all AESIs.
- After the individual patient's end of trial: the investigator does not need to actively monitor the patient for new AEs but should only report any occurrence of cancer and trial drug related SAEs and trial drug related AESIs of which the investigator may become aware of by any means of communication, e.g. phone call. Those AEs should be reported on the BI SAE form (see Section 5.2.6.2.2), but not on the CRF.

# Vital Status Data Collection

Patients who discontinue trial treatment prematurely, who agree to be contacted further but do not agree to physical visits, should be followed up as described in Section 3.3.4.1, withdrawal from trial treatment. From then on until the individual patient's end of the trial the investigator must any occurrence of cancer, report all deaths/fatal AEs regardless of relationship, and trial drug related SAEs and trial drug related AESIs the investigator becomes aware of.

# 5.2.6.2.2 AE reporting to the sponsor and timelines

The investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the AE or SAE eCRF pages to the sponsor's unique entry point within 24 hours of becoming aware of the event, the country specific process will be specified in the ISF. The same timeline applies if follow-up information becomes available. In specific occasions, the investigator could inform the sponsor upfront via telephone in addition.

With receipt of any further information to these events, a follow-up reports have to be provided. For follow-up information the same rules and timeline apply as for initial information. All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been assessed as "chronic" or "stable", or no further information can be obtained.

Should the eDC system not be available for more than 24 hours, reporting must occur via the BI paper SAE forms.

# 5.2.6.2.3 Pregnancy

In rare cases, pregnancy might occur in a clinical trial. Once a patient has been enrolled in the clinical trial and has taken trial medication, the investigator must report any drug exposure during pregnancy in a trial participant immediately (within 24 hours) by means of Part A of the Pregnancy Monitoring Form to the sponsor's unique entry point.

Similarly, potential drug exposure during pregnancy must be reported if a partner of a male trial participant becomes pregnant. This requires written consent of the pregnant partner.

#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Reporting and consenting must be in line with local regulations. The ISF will contain the trial specific information and consent for the pregnant partner.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Studies (Part B).

The ISF will contain the Pregnancy Monitoring Form for Clinical Studies (Part A and B).

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE and/or AESI, only the Pregnancy Monitoring Form for Clinical Studies and not the SAE form is to be completed. If there is an SAE and/or AESI associated with the pregnancy an SAE form must be completed in addition.

5.2.6.3 Independent safety monitoring and adverse events with additional information collection

An independent data monitoring committee (DMC) will conduct regular reviews of the trial safety data, as detailed in the DMC charter.

An independent adjudication committee will review all fatal cases (to review the primary cause of death). The independent adjudication committee will also review all adverse events categorized as major adverse cardiovascular events (MACE).

A separate independent adjudication committee will review all events categorized as vasculitis (SMQ vasculitis broad).

Before providing any copy of patients' source documents to the sponsor, the investigator must ensure that all patient identifiers (e.g. patient's name, initials, address, phone number, social security number) have properly been removed or redacted to ensure patient confidentiality.

Additional details (on top of standard AE and SAE reporting) will be collected in the eCRF for the adverse event 'Diarrhea/gastrointestinal events', the adverse events in the Standard MedDRA Query (SMQ) 'vasculitis' and in case of positive TB tests (see Section 5.2.3.2).

# 5.3 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

# **5.3.1** Assessment of pharmacokinetics

Cpre,ss (predose concentration of analyte in plasma at steady state) will be the main PK parameter determined in this study. Further PK parameters might be calculated as appropriate.

Date and clock time of PK sampling, the two preceding and the current drug administrations will be recorded in the CRFs. The actual sampling times will be used for determination of the PK parameters.

PK sampling will be performed predose at the time points indicated in the flow chart.


Clinical Trial Protocol

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5.3.2 Methods of sample collection

For quantification of drug plasma concentrations of BI 1015550, venous blood will be collected using a prelabeled EDTA (Ethylenediaminetetraacetic acid) containing blood drawing tube at the times indicated in the <u>flow chart</u>. Blood will be withdrawn by means of either an indwelling venous catheter or by venipuncture with a metal needle. A detailed description of sample collection and handling is provided in the Lab Manual in the ISF.

Plasma samples will be discarded at latest 6 months after the final clinical trial report has been signed.



### 5.4 ASSESSMENT OF BIOMARKERS

Biomarkers associated with ILD pathology will be explored in serum, plasma, and whole blood and will be correlated with clinical endpoints.

#### 5.4.1 Pharmacodynamics biomarkers

Effects of BI 1015550 treatment on several protein biomarkers such as, but not limited to, KL-6, MMP-7, SP-D, COMP, vWF, CA-125, and CA19-9 will be investigated. Further protein markers will be evaluated and correlated to clinical endpoints. In addition, effects of BI 1015550 treatment on the formation of

and others will be

evaluated and correlated to clinical endpoints.

Total mRNA expression levels in whole blood and miRNA levels in plasma will be evaluated to investigate the drug's mode of action or the pathology and course of the disease.

All biomarkers assessed in this trial are considered exploratory and qualified assays will be used according to the sponsor's procedures. Characteristics of the analytical methods for the analysis of plasma and serum biomarkers will be given in detail in the analytical report.

Genome-wide expression profiling will be performed by RNA sequencing including bioinformatics analysis. Further characteristics of the analytical method for the analysis will be given in detail in the analytical report.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Changes in serum and plasma biomarkers, and in gene expression (RNA) levels will be analyzed over time, pre- and post-treatment with BI 1015550.

All assessed biomarkers will either be analyzed at the sponsor or at a CRO. The results of biomarker analyses will be reported separately in biomarker reports.

# 5.4.1.1 Methods and timing of sample collection

Whole blood will be collected for the preparation of serum, plasma, and RNA expression analysis.

Overall about 75 mL blood will be taken for explorative biomarker assessment during the course of the trial.

Remaining samples may be used for method development and evaluation and will be stored for a maximum of 3 years after approval of the clinical trial report.

Details about sample collection and sample handling will be provided in the ISF. A detailed overview of biomarker sample collection visits is outlined in the flow chart.

A detailed description of biomarker sample collection and sample handling is provided in the ISF.

#### 5.5 BIOBANKING

Participation in biobanking is voluntary and not a prerequisite for participation in the trial. Biobanking will only occur after a separate biobanking informed consent has been given in accordance with local ethical and regulatory requirements. Any country not approving the biobanking will not participate in this process.

# 5.5.1 Methods and timing of sample collection

Detailed instructions on sampling, preparation, processing, shipment, and storage are provided in the laboratory manual. For sampling timepoints see <u>flow chart</u>.

Serum/plasma from the original whole blood sample will be stored at an external biobanking facility contracted by the sponsor.

The following samples will be banked:

Unspecified pharmacogenomics (PGx) samples (DNA banking):

An additional blood sample (approximately 8.5 mL) for DNA banking will be collected in PAXgene Blood DNA tube at Visit 2. The DNA banking sample, derived from the original blood sample, will be stored at Boehringer Ingelheim. The stored DNA may be retrospectively analyzed.

# c39145241-04 Clinical Trial Protocol


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# <u>Unspecified serum/plasma samples (serum/plasma banking):</u>

Whole blood will be collected for the preparation of serum and plasma for banking purposes. In total, a maximum of 74 mL of blood will be drawn for the purpose of serum/plasma banking.

#### 5.6 OTHER ASSESSMENTS

#### 5.6.1 Chest HRCT assessment

Screening chest HRCT will be used in all patients to determine study eligibility.

An historical HRCT can be used to determine eligibility, providing the scan was performed within the 12 months prior to screening. If a historical scan is not available, or an available scan fails to meet the required image acquisition specification, an HRCT may be performed after consent to determine eligibility.

All HRCT scans will be sent to a vendor for central review and confirmation of UIP or probable UIP HRCT pattern (for detailed specifications see Appendix 10.6) prior to randomization. Confirmation of eligibility must be available prior to randomization Visit 2.

If required, the HRCT scan should be performed as close to screening date as possible, preferably once eligibility is confirmed based on other parameters, to avoid unnecessary scans for patients who are found ineligible based on other criteria.

To perform a HRCT within the trial, all local regulatory requirements to perform an HRCT have to be met. In Germany, no HRCT will be performed as trial procedure; only historical HRCT will be submitted.

In addition to central reading of the HRCT scans, there is the intention to apply a computer scoring technology. If feasible, this technology will only be applied for scientific reasons and learnings and results will not be part of the clinical trial report. Determination of eligibility will, however, always be based on the central visual reading.

# 5.6.2 Health care resource utilization (HCRU)

For the purpose of a separate health economic analysis (such as cost-utility analysis), health care resource utilization (HCRU) data will be collected throughout the trial. Resource use data collected for calculating direct costs will include unscheduled hospitalizations, healthcare provider visits, and emergency room/intensive care unit use. Non-medical resource use data will include changes in work productivity.

The economic evaluation of the HCRU data will not be part of the clinical trial report.

# 5.7 APPROPRIATENESS OF MEASUREMENTS

All measurements conducted for primary and secondary endpoints are using standard methods. The pharmacokinetic parameters and measurements outlined in Section 5.3 are

#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

generally used as measurements to assess drug response. Measures conducted for exploratory endpoints might be new methodologies used in clinical trials but not yet validated for IPF.

# 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

The trial consists of 2 parts: Treatment Period A and B. Treatment Period A will consist of Visits 2 through 10, which will occur within one year of randomization. Following completion of the Week 52 visit (Visit 10), patients will continue to have trial visits every 12 weeks (Treatment Period B) until the end of the trial.

The trial will last the until last patient completes the EOT Visit and the Follow-up Visit as applicable (see <u>Figure 3.1: 1</u>).

After giving informed consent, the patient will be screened for inclusion (see Section 3.3.2) and exclusion criteria (see Section 3.3.3) for the trial at Visit 1 and Visit 2 (refer to flow chart Treatment Period A). Visit 2 can be performed once the results from central laboratory of Visit 1 and central chest HRCT review are obtained. If for any reason the screening phase for an individual patient lasts for more than 8 weeks, then the laboratory examination for Visit 1 has to be repeated before randomization. The screening phase must be no longer than 12 weeks.

The patient will be randomized at Visit 2 if all inclusion criteria (including positive HRCT review and acceptable spirometry measurements) and none of the exclusion criteria (lab exclusion criteria referring to Visit 1 results) are fulfilled.

The acceptable time windows for visits are provided in the flow chart. Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed prior to the trial drug administration (including predose values for PK and biomarkers).

If a patient misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

In the event of force majeure or other disruptive circumstances (e.g. pandemic, war) the execution of the investigational plan as per this clinical trial protocol may not be feasible. With the consent of the patient, the sponsor and investigator may agree on alternative, back-up or rescue methodology which may include but will not be limited to virtual trial participant visits and assessments, home healthcare nurse visits, direct-to-patient/direct-from-patient shipments of trial treatment or bio-sample pick up from the patient's home. The implementation of these measures will depend on patient's consent, operational feasibility, local law and regulations.

Based on a thorough assessment of the benefits and risks, some specific visits may be performed remotely, e.g. via telephone and/or internet-based means of communication, performance of assisted home spirometry and ePRO collection where applicable, or at the patient's home where a respective study nurse or home healthcare nurse service is feasible.

c39145241-04

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The visits may also be performed as a combination of home and remote visits, see descriptions of procedures in Section 6.2.2.2.

All deviations from the original schedule of visits and procedures will be documented and the implications considered for the analysis of the trial data.

# 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

In regards to the timing of the investigations/assessments, the following aspects should be adhered to:

- the patients' questionnaires (L-PF [symptoms/impact], EQ-5D-5L, HADS, PGIS) are to be completed preferably in the order of the <u>flow chart</u> before any other visit assessments or treatments, and if possible, before any interaction with the investigator or other members of the study team. Alternatively, the patient can complete them at home within 3 days before the site visit. At the latest, the patients' questionnaires must be completed prior to the pulmonary function tests.
- the C-SSRS interview should be done second, before any other procedure or assessment at the site
- for the pulmonary function tests: FVC (spirometry) must be performed before DLCO
- if several measurements including venipuncture are scheduled for the same time, venipuncture should be the last of the measurements due to its inconvenience to the patient and possible influence on physiological parameters.
- IRT call and IMP dosing/dispensing should always be done as the last procedure after all visit assessments, except at Visit 1 where the IRT call may be done earlier during the patient's visit.

# 6.2.1 Screening period

# Screening Period

After informed consent is obtained, inclusion and exclusion criteria should be checked according to flow chart.

- During the screening visit, demographics information will be collected. This includes: age on the day of informed consent (in years)
- Sex (male, female; to describe the patient's sex at birth),
- Gender identity (male, female, other; in order to describe how the subject self-identifies regardless of their genotypic or phenotypic sex)
- For women: childbearing potential (yes/no) in order to characterize the patient population and as a basis for contraception requirements
- Ethnicity and race in order to sufficiently characterize the patient population, to support possible subgroup analyses if needed unless not acceptable according to local regulations.

Patients will be asked to give informed consent to the DNA, plasma and serum banking samples (please note: the banking samples must not be taken prior to Visit 2). Participation is voluntary and is not a prerequisite for participation in the trial.

For information regarding laboratory tests, ECG, vital signs, height, body weight, and physical examination, SpO2, refer to Sections 5.2.1 to 5.2.4.

c39145241-04

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For information on spirometry (FEV1 and FVC) and DLCO refer to Sections 5.1.1 and 5.1.6.

For information on the patient-reported outcomes/questionnaires and specific safety related questionnaires refer to Sections 5.1.5 and 5.2.5.

For information on chest HRCT, refer to Section <u>5.6.1</u>.

### Re-screening:

If patients fail on specific exclusion criteria during the first screening visit, they may be rescreened under the following conditions:

- If the patient was treated and cured from the acute infection.
- If the patient was treated for depression and HADS values are <14, not earlier than 3 months after the first screening.
- Other reversible conditions after respective treatment or resolution

If a patient results in a screen failure the patient must be registered as a screen failure in IRT system. However, re-screening of a previously screen failed patient will be permitted once. Details of IRT procedures can be found in the IRT manual located in the Investigator Site File (ISF).

Re-screened patients will need to sign a new informed consent before any re-screening procedures and will be given a new unique patient number.

If a patient is re-screened and there are valid screening determinations from patient's previous participation in the trial, like for example safety labs, performed within 8 weeks prior to randomization (Visit 2), these do not need to be repeated.

If the Investigator believes that an ineligible laboratory test result is the result of an error or extenuating circumstance, then the test can be repeated once without the patient having to be re-screened.

# **6.2.2** Treatment periods

# 6.2.2.1 Conduct of a regular site visit

At the beginning of each visit during treatment phase, Investigator and site personnel should check the well-being of the patient as well as prepare all requirements for conduct of the visits that are necessary.

For information regarding laboratory tests, ECG, vital signs, height, body weight and physical examination, SpO2, refer to Sections <u>5.2.1</u> to <u>5.2.4</u>.

For information on spirometry (FEV1 and FVC) and DLCO refer to Sections <u>5.1.1</u> and <u>5.1.6</u>.

For information on the patient-reported outcomes/questionnaires and specific safety related questionnaires refer to Sections 5.1.5 and 5.2.5.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Each patient will receive the first dose of BI 1015550 or placebo at the end of Visit 2 (Day 1) under direct supervision of the investigator or designee. Patients will take trial medication twice daily (bid) orally from that timepoint onwards. On the day of any further clinic visit, supervision of administration is not required but trial medication will preferably be administered to the patient during the visit (as the last procedure, see Section 6.2).

The patient will have to bring back all IMP kits, used and unused at each on-site visit, including Visit 3. At Visit 3, the patient will have to bring back the IMP kits dispensed at Visit 2 to cover the trial medication intake until Visit 4.

FVC should be measured at approximately the same time of day, at least within the same half-day (morning or afternoon, with reference to the time at Visit 2).

# 6.2.2.2 Conduct of a fallback visit (remote/home visit)

If a patient is not able to travel to the site for a trial visit (Force majeur or physical disablement), remote visits (by phone or video call) should be performed instead. Especially for Visits 2, 5, 7, 10, and EOT, patients should be encouraged to perform a site visit as close as possible to the intended timepoint per <u>flow chart</u> including visit windows to perform an onsite spirometry.

Trial medication may be shipped from the site directly to the patient (if acceptable according to local laws and regulations).

The following assessments can be done remotely:

- Collect and assess adverse events, concomitant therapies, assess trial medication compliance.
- Specific data for investigator reported data: C-SSRS interview, evaluation of vasculitis symptoms and HCRU questions.
- Patient-reported outcomes: the patient questionnaires can be compiled electronically by the patient on the provided device or via the App on his own device. If paper questionnaires had been handed out at the last visit, the questionnaires should be answered on the day (or within 3 days) of the remote visit and sent back to the site thereafter.
- Assisted home spirometry: for sites with the respective setup, see Section <u>5.1.1</u> and the respective home spirometry manual.
- Urine dipstick pregnancy test performed by the patient at home

If home visits are possible (e.g. by a Home Healthcare Nurse or qualified site staff visiting the patient), the following assessments can be done at the patient's home:

- collection of blood and urine samples to be sent to the central lab or local lab
- vital signs
- trial medication compliance assessment
- dispensing of the next treatment kits, if possible

If blood and urine sampling for central lab at the patient's home is not possible, safety lab analyses including the routine safety lab tasks as per Table 5.2.3.1: 1 should be performed at

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

a local lab. The results of the lab tests must be transferred to the investigator who ensures medical review and documents a clinically relevant safety issue as an adverse event.

#### 6.2.2.3 End of treatment visit

As described in Section 3.1, after the confirmation of the benefit-risk evaluation for a potential start of the extension trial based on the main analysis, all patients still on blinded study treatment will perform an EOT visit.

For premature treatment discontinuations, follow instructions in Section <u>3.3.4.1</u>.

# 6.2.3 Follow-up period and trial completion

A follow up period of a minimum of 7 days (+3 days) after the end of treatment will be required. All patients will complete a visit at the end of the follow-up period for AE assessment, laboratory tests, recording of ECG and vital signs, and physical examination.

Patients may be eligible to enter an extension trial if they complete this study on blinded treatment and meet the eligibility criteria for the extension trial. For these patients, the last visit in this trial and the end of this trial is the EOT visit. For patients who do not roll over to the separate extension trial (or could not roll over within a week of the EOT visit), the follow-up visit is required as the regular EOS visit.

Patients prematurely discontinuing trial treatment permanently will perform the EOT visit at the time of permanent discontinuation and the follow-up visit 7 days (+3 days) later. As this is taking place before the end of study, the patients should perform all regular trial visits as indicated in Section 3.3.4.1. For these off-treatment visits, PK samples can be skipped.

The follow-up visit can be skipped if the treatment had been discontinued at least 7 days before the actual EOT visit or if the following regular visit after the end of treatment is planned at 7-21 days after the last dose was administered.

For patients who withdraw consent – at time of trial medication discontinuation, end of study is an EOT visit followed by a follow-up visit.

All abnormal values (including laboratory parameters) at the last study visit (EOS) that are judged clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. All (S)AEs persisting after individual patient's end of trial must be followed up until they have resolved, have been assessed as "chronic" or "stable", or no further information can be obtained.

If needed in the opinion of the investigator, after the EOS visit additional FU visits may be scheduled for continued safety monitoring.

The end of the trial is defined as the date of the last visit of the last patient in the whole trial ("Last Patient Completed").

c39145241-04  Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

As a default, a patient is considered to have completed the trial in case any of the following applies:

- Completion of planned follow-up period
- Lost to follow-up
- Refusal to be followed-up
- Death

#### 7. STATISTICAL METHODS AND DETERMINATION OF **SAMPLE SIZE**

This is a multi-centre, multi-national, prospective, randomized, placebo-controlled, double blind clinical trial to investigate the efficacy and safety of BI 1015550 at a dose of 9 mg bid and 18 mg bid, in patients with IPF. The eligible patients will be randomized to BI 1015550 9 mg bid, BI 1015550 18 mg bid and placebo in 1:1:1 ratio, stratified by intake of AF treatment at baseline.

The primary endpoint is the absolute change from baseline in FVC (mL) at Week 52. The primary endpoint will be analyzed using a mixed-effect model for repeated measures (MMRM) as detailed in Section 7.2.3.

The key secondary endpoint is time to the first occurrence of any of the components of the composite endpoint: time to first acute IPF exacerbation, first hospitalization for respiratory cause, or death. The key secondary endpoint will be analyzed using a Cox proportional hazards model as detailed in Section 7.2.4 with data from the whole trial, i.e. including data beyond 52 weeks.

#### 7.1 NULL AND ALTERNATIVE HYPOTHESES

Multiplicity adjusted analyses will be performed on the primary and key secondary endpoints. The graphical testing procedure [R16-4473] as depicted in Figure 7.1: 1 will be used to test the primary and key secondary endpoints for both dose levels. As the graphical testing procedure abides the closed test principle, it holds strong control of family-wise type I error rate at two-sided alpha level of 0.05.

Statistical hypotheses to be tested for the primary endpoint are:

- $H_{01}$ : there is no difference in the mean change from baseline in FVC in mL at Week 52 between BI 1015550 18 mg bid and placebo vs. H<sub>al</sub>: there is a difference in the mean change from baseline in FVC in mL at Week 52 between BI 1015550 18 mg bid and placebo.
- $H_{02}$ : there is no difference in the mean change from baseline in FVC in mL at Week 52 between BI 1015550 9 mg bid and placebo vs. H<sub>a2</sub>: there is a difference in the mean change from baseline in FVC in mL at Week 52 between BI 1015550 9 mg bid and placebo.

Statistical hypotheses to be tested for the key secondary endpoint are:

 $H_{03}$ : there is no difference in the time to first acute IPF exacerbation, first hospitalization for respiratory cause or death between BI 1015550 18 mg bid and Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

placebo vs.

 $H_{a3}$ : there is a difference in the time to first acute IPF exacerbation, first hospitalization for respiratory cause or death between BI 1015550 18 mg bid and placebo.

•  $H_{04}$ : there is no difference in the time to first acute IPF exacerbation, first hospitalization for respiratory cause or death between BI 1015550 9 mg bid and placebo vs.

 $H_{a4}$ : there is a difference in the time to first acute IPF exacerbation, first hospitalization for respiratory cause or death between BI 1015550 9 mg bid and placebo.

The hypothesis testing of the key secondary endpoint is based on data collected up to the main analysis (all data up to DBL1; see <u>Figure 3.1: 1</u>). A supplementary analysis of the key secondary endpoint using all data collected over the whole trial will be performed after DBL2.



Figure 7.1: 1 Graphical testing procedure for hypothesis testing strategy

The testing procedure will start from testing of  $H_{01}$  and  $H_{02}$  for the primary endpoint. 4% level of the alpha level will be initially allocated to the comparison between 18 mg bid and placebo. 1% level of the alpha level will be initially allocated to the comparison between the 9 mg bid arm and placebo. At this step, no alpha is reserved for tests of the key secondary endpoint.

- If neither  $H_{01}$  nor  $H_{02}$  is rejected, all  $\alpha$  is deemed as "spent" and no further testing will be performed.
- If at least one of  $H_{01}$  or  $H_{02}$  is rejected, the retained  $\alpha$  from the successful hypothesis will be propagated according to the weights on the arrows leaving that hypothesis as depicted by the Figure 7.1: 1.

Note that  $\epsilon$  is set to a negligible amount of 0.0001 at the start, to reflect the priority on hypotheses for 18 mg bid vs. placebo, namely  $H_{01}$  and  $H_{03}$ ! over the 9 mg bid vs. placebo"


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The testing process continues if there is at least one hypothesis in the procedure that can be rejected at its allocated  $\alpha$  level at that point. Each time a hypothesis is rejected, the graph is updated to reflect the reallocation of  $\alpha$ . This iterative process of updating the graph and reallocating  $\alpha$  is repeated until all hypotheses have been tested or when no remaining hypotheses can be rejected at their corresponding  $\alpha$  levels at that point.

The primary objective of the trial will be achieved if either  $H_{01}$  or  $H_{02}$  is rejected and this trial is considered positive.

If the 9 mg bid arm is considered futile at the futility interim, the remaining tests for 18 mg bid arm will be tested sequentially for primary and key secondary endpoint with  $\alpha$  level of 0.04 and 0.02 as depicted in Figure 7.1: 1.

No adjustment for multiplicity is planned beyond primary and key secondary objective analyses.

#### 7.2 PLANNED ANALYSES

#### 7.2.1 General considerations

All planned efficacy and safety analyses, including for the primary and key secondary endpoints will be carried out at DBL1 (Figure 3.1: 1) and the statistical hypotheses described in Section 7.1 will be tested. After DBL2, analyses of the efficacy endpoints defined as "over the duration of the trial" and all safety analyses will be repeated to include all data collected until the end of the trial.

The following analysis sets will be defined for statistical analyses:

Entered Set (ES): This patient set includes all patients who signed informed consent. The ES will be used for the analyses of patient disposition.

Randomized Set (RS): This patient set includes all entered and randomized patients. The RS will be used for the analyses of patient disposition.

Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug. The FAS will be used for baseline demographics and characteristics, protocol deviations, and all efficacy analyses, in which patients will be analyzed as their randomized treatment group.

Treated Set (TS): This patient set includes all randomized patients who received at least one dose of study drug. The TS will be used for all safety analyses, in which patients will be analyzed according to the actual treatment they received.

Data from patients who are screened but not randomized will be listed but not included in any summary statistics or inferential statistics. Definitions and handling of important protocol deviations (IPDs) will be included in the DV domain specifications and will be stored within the trial master file (TMF) in the electronic document management system (EDMS). All potential important protocol deviations will be discussed during trial oversight meetings and


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

report planning meetings. All final decisions concerning IPDs will be made before unblinding.

Further Analysis Sets will be defined in the TSAP, if needed.

# 7.2.2 Handling of intercurrent events

The expected intercurrent events of interest in this trial are:

- Change in background antifibrotic therapy after baseline
- Start of a restricted medication
- Treatment discontinuation
- Death
- Lung transplant

The strategies for handling intercurrent events in this trial are as follows:

Primary strategy for primary and key secondary objectives:

All intercurrent events except for death and lung transplant will be handled according to the treatment policy approach as defined in ICH E9 (R1). Use of the "treatment policy" approach disregards the intercurrent event and uses the value of the variable regardless of the occurrence of the intercurrent event (e.g., start of a restricted medication).

The intercurrent event of death will be primarily handled using a mixture of composite and hypothetical strategy as defined in ICH E9 (R1). Use of the "hypothetical approach" considers the effect of what would have happened if the intercurrent event did not occur. Use of the "composite approach" considers that a poor outcome will be expected. The intercurrent event of lung transplant will be primarily handled using a hypothetical strategy as defined in ICH E9 (R1).

Table 7.2.2: 1 Handling of intercurrent events as per ICH E9 (R1) within the different strategies

| Intercurrent event | Primary strategy for primary objective | Primary strategy for key secondary objective |
|---|---|---|
| Change of background antifibrotic therapy | Treatment policy | Treatment policy |
| Start of a restricted medication | Treatment policy | Treatment policy |
| Treatment discontinuation or interruption (any cause) | Treatment policy | Treatment policy |
Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Intercurrent event | Primary strategy for primary objective | Primary strategy for key secondary objective |
|---|---|---|
| Death | Hypothetical/<br>Composite | Composite (event) |
| Lung transplant | Hypothetical | Hypothetical (censored) |

Each analysis will reference the strategy for handling intercurrent events that it will be estimating. The estimand for each main analysis in this protocol is the combination of the relevant detailed clinical objective from Section 2.1 and this strategy.

The secondary strategy will handle change of background antifibrotic therapy and treatment discontinuation by a hypothetical approach. Remaining intercurrent events will be handled in the same way as the primary strategy.

Any intercurrent events that are not listed will be decided by blinded review based on the general principle outlined and secondary strategies will be documented in the TSAP.

### 7.2.3 Primary objective analyses

### Planned analyses for primary endpoint

The primary analysis is a restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) comparing the change from baseline in FVC at Week 52 between treatment groups. The analysis will include the fixed, categorical effects of treatment at each visit, baseline intake of AF treatment at each visit, and the fixed continuous effects of baseline FVC value at each visit. Visit will be treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The statistical model will be as follows:

$$y_{ijkm} = \beta_j S_i + \tau_{jk} + f_{jm} + e_{ij}$$
$$e_{ij} \sim N_Z(0, \Sigma)$$

- $y_{ijkm}$  = change from baseline in FVC value [mL] for patient i in intake of AF treatment at baseline stratum m at visit j receiving treatment k,
- $S_i$  = FVC baseline measurement (mL) of patient i, i = 1, 2, ...
- $\beta_i$  = coefficient of baseline effect at visit j
- $\tau_{jk}$  = the effect of treatment k at visit j, j = 1, ..., Z and k = 1, ..., Y,
- $f_{jm}$  = the effect of intake of AF treatment at baseline stratum m at visit j, m = 1,2. Intake of AF treatment at baseline is used as reported in the CRF ("No" as the class of reference, regardless of any mis-assignment to treatment based on identification of the wrong stratum in IXRS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

-  $e_{ij}$  = the random error associated with the  $j^{th}$  visit of the  $i^{th}$  patient. Errors are independent between patients.

 $\Sigma$  = an unstructured covariance matrix

The Kenward-Roger approximation will be used to estimate denominator degrees of freedom and adjust standard errors. Significance tests will be based on least-squares means using a two-sided  $\alpha$  according to the multiple testing strategy specified in Section 7.1. The primary treatment comparison will be the contrast between treatments at Week 52.

Baseline is defined as data collected at Visit 2 prior to administration of first dose of study medication, or screening data if Visit 2 data are missing.

The primary analysis will be performed on the FAS. Patients will be analyzed according to the stratum to which they belong (regardless of any mis-assignment to treatment based on identification of the wrong stratum), as such an error occurs before randomization and is therefore consistent with regulatory guidance.

A treatment policy estimand will be used for primary analysis (i.e., all available data from the FAS in each active treatment arm and the placebo arm within the first 52 weeks will be used, including baseline and data retrieved post treatment discontinuation for patients who prematurely discontinued randomized treatment and after use of antifibrotic (rescue) therapy for patients not on AF therapy).

### 7.2.3.1 Sensitivity Analyses

Sensitivity analysis will be performed to assess whether background therapy status influences the primary efficacy analysis. This will use the same primary analysis model with an additional covariate of antifibrotic treatment at baseline, treatment, and visit interaction.

MMRM analyses assume that data are missing at random (MAR). For the primary outcome, tipping point analyses will assess how robust the primary analysis is against deviations from the MAR assumption by imposing a penalty for missing data. The tipping point analysis for the longitudinal FVC data will be based on the Multiple Delta Adjustment Method. A delta adjustment, dependent on a shift parameter and the weeks between visits, will be added to each imputed value. Shift parameters will be selected by arm covering plausible and implausible cumulative changes of FVC values at Week 52.

Additional sensitivity analyses based on different missing data imputation scheme as detailed in Section <u>7.3.1</u> will be conducted.

On-treatment, while-compliant-to-protocol analyses and models with modified sets of covariates will be conducted as further sensitivity analyses.

Further details will be specified in the TSAP.

### 7.2.3.2 Subgroup Analyses

Subgroup analyses will include at least gender, age and antifibrotic treatment at baseline. A complete list of subgroup analyses will be specified in the TSAP.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.2.3.3 Supplementary Analyses

Further details will be specified in the TSAP.

### 7.2.4 Secondary objective analyses

### 7.2.4.1 Analysis of key secondary endpoint

The key secondary endpoint of time to first acute IPF exacerbation, first hospitalization for respiratory cause or death will be analyzed with a Cox proportional hazards model using data over the whole trial, i.e., including data beyond 52 weeks. The equality of the hazard rates will be tested by the Wald test for the treatment effect at a two-sided significance level deemed for test in each step as specified in Section 7.1. The model will include the treatment effect, intake of AF treatment, age (continuous), FVC % predicted and DLCO % predicted (corrected for hemoglobin) at baseline as covariates. Breslow's method for handling ties will be used. Kaplan-Meier plots by treatment group will be presented. In addition, percentage of patients with event at Week 52 will be presented both descriptively and by Kaplan-Meier estimates.

In general, for all time-to-event endpoint, the time to the event of interest will be computed as (event date – first drug intake date) +1. All events observed after first drug intake date until trial termination will be included in the analysis except for events occurring after a lung transplantation as outlined in Section 7.2.2. Patients who do not have an event during the trial period will be censored at the individual day of trial completion or the last day that the patient was known to be free of the event, whichever is earlier. The time to censoring will be computed as (individual day of trial completion or the last day known to be free of the event – first drug intake date) + 1. For patients who have more than one event during the trial, the time to the first event will be considered for the analysis.

Same as for the primary endpoint, the primary analysis will be performed on the FAS using a treatment policy estimand listed in Section 7.2.2.

On-treatment, while-compliant-to-protocol analyses and models with modified sets of covariates will be conducted as further sensitivity analyses. In addition, handling change of background antifibrotic therapy or treatment discontinuation will also be evaluated by hypothetical approach (censored) and composite approach (addition of antifibrotic therapy considered as event).

Further details will be specified in the TSAP.

### 7.2.4.2 Analysis of other secondary endpoints

Absolute change from baseline in the various Living with Pulmonary Fibrosis (L-PF) (domain) scores at Week 52 will be analyzed by a restricted maximum likelihood (REML) estimation based approach using a mixed-effect model with repeated measurements (MMRM) analysis comparing the change from baseline in respective L-PF (domain) Score at Week 52 between treatment groups. The analysis will include the fixed, categorical effects of treatment at each visit, intake of AF treatment at baseline, and the fixed continuous effects of baseline at each visit.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In general, for all time-to-event endpoints, the time to the event of interest will be computed as (event date – first drug intake date) +1. All events observed after first drug intake date until trial termination will be included in the analysis except for events occurring after a lung transplantation as outlined in Section 7.2.2. Patients who do not have an event during the trial period will be censored at the individual day of trial completion or the last day that the patient was known to be free of the event, whichever is earlier. The time to censoring will be computed as (individual day of trial completion or the last day known to be free of the event – first drug intake date) + 1. For patients who have more than one event during the trial, the time to the first event will be considered for the analysis.

Time to event secondary efficacy endpoints will be analyzed using a Cox proportional hazards model using data from the whole trial i.e. including data beyond 52 weeks. The equality of the hazard rates will be tested by the Wald test for the treatment effect at the two-sided 5% significance level. The model will include the treatment effect and intake of AF treatment, age (continuous), FVC % predicted and DLCO % predicted (corrected for hemoglobin) at baseline as covariates . Breslow's method for handling ties will be used. Kaplan-Meier plots by treatment group will be presented. In addition, percentage of patients with event at Week 52 will be presented both descriptively and by Kaplan-Meier estimates.

Any p-values presented for the other secondary endpoints will be considered nominal in nature and no adjustment for multiplicity will be made.

### 7.2.5 Further objective analyses

All further endpoints will be considered exploratory in nature. The analysis of further endpoints over 26 or 52 weeks will be performed with the same models and procedures as described for the primary and secondary endpoints.

Restricted maximum likelihood estimation based on a random slope and intercept model will be used to compare the adjusted annual rate of decline in FVC [mL/year] as measured over 52 weeks between treatment groups. This model will include fixed effects for time, treatment, baseline, intake of AF treatment at baseline, as well as treatment-by-time and baseline-by-time interactions. Random effects for time and intercept will be included for each patient.

Further time to event endpoints will be assessed using similar analysis models as respective secondary time to event endpoints (e.g. Cox regression models, Kaplan-Meier plots).

The annualized rate of hospitalization due to respiratory cause over the whole trial will be analyzed using negative binomial regression with logarithm of the exposure as an offset. The analyses will include the treatment effect, intake of AF treatment at baseline, and other key covariates of interest with more detail to be provided in the TSAP. The mean number of events per patient year by treatment arm, the rate ratio, and corresponding 95% confidence interval will be presented.

### 7.2.6 Safety analyses

All safety assessments described below will focus on data collected within the first 52 weeks and additional safety analyses will be repeated to include data over the whole trial.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Adverse events will be coded using the Medical Dictionary for Drug Regulatory Activities (MedDRA). Standard BI summary tables and listings will be produced. All adverse events with an onset between start of treatment and end of the REP, a period of 7 days after the last dose of trial medication, will be assigned to the on-treatment period for evaluation.

Kaplan-Meier plots will be produced for the time to premature treatment discontinuation and for the time to first treatment interruption.

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events, i.e. all adverse events occurring between start of treatment and end of the REP. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.

Frequency, severity, and causal relationship of adverse events will be tabulated by system organ class and preferred term after coding according to the current version of the Medical Dictionary for Drug Regulatory Activities (MedDRA) at database lock.

Laboratory data will be analyzed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be summarised. Treatment groups will be compared descriptively with regard to distribution parameters as well as with regard to frequency and percentage of patients with abnormal values or clinically relevant abnormal values.

Vital signs, physical examinations, or other safety-relevant data observed at screening, baseline, during the course of the trial and at the end-of-trial evaluation will be assessed with regard to possible changes compared to findings before start of treatment.

Summary tables will be produced for the adjudication results of MACE and deaths.

Further details will be specified in the TSAP

### 7.2.7 Other Analyses

### 7.2.7.1 Pharmacokinetic Methods

In the Clinical Trial Report, plasma concentrations of BI 1015550 will be tabulated with descriptive statistics. A population PK analysis may be performed on BI 1015550 plasma concentrations. If so, a separate population PK analysis plan will be written, and results will be reported separately.

### 7.2.8 Interim analyses

An interim analysis to assess futility of the 9 mg bid dose will be performed when approximately 300 patients (100 patients per arm) in the trial have completed 12 weeks of treatment taking also into account the safety data from trial 1305-0023. Specific details of timing of the interim, futility criteria and analysis plan will be detailed in the DMC charter or

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP as appropriate. The DMC will review the results and make a recommendation to the sponsor on continuation or stoppage of the 9 mg bid dose arm. If the 9 mg dose is considered futile, the patients on that treatment arm will be re-assigned to the 18 mg dose in a blinded manner (see Section 4.1.5.1) at their next scheduled visit.

Full details will be provided in the DMC charter.

### 7.3 HANDLING OF MISSING DATA

### 7.3.1 Efficacy endpoints

In the primary analysis of primary endpoint, missing data will not be imputed except for death, where a poor outcome will be assigned, see <u>Table 7.3.1: 1</u>. The mixed effect model will handle missing data based on a likelihood method under the "missing at random assumption".

A tipping point analysis is planned as sensitivity analysis, see Section <u>7.2.3.1</u>. The effect of missing data on the primary endpoint will be further investigated using other multiple imputation techniques.

These four subsets of patients will be used in sensitivity analyses to estimate the treatment effect under differing assumptions around the persistence of efficacy after withdrawal of trial medication.

- 1. Patients with an FVC result at Week 52 who received trial medication until Week 52.
- 2. Patients with an FVC result at Week 52 who prematurely discontinued trial medication prior to Week 52.
- 3. Patients without an FVC result at Week 52 who were alive at Week 52.
- 4. Patients without an FVC result at Week 52 who died prior to Week 52.

<u>Table 7.3.1: 1</u> describes the planned sensitivity analyses for handling missing primary endpoint data. Sensitivity analyses 1 and 2 will only be performed if there are at least 10 patients included in patient subset 2 in each treatment group.

Table 7.3.1: 1 Sensitivity analyses for handling missing primary endpoint data

| Analysis | Patient subset 3 but alive at Wee | | Patient subset 4: No FVC result but died Week 52 | |
|---|---|---|---|---|
| | Handling of missing FVC | Underlying assumption | Handling of missing FVC | Underlying assumption |
| Primary<br>analysis | Missing data<br>handled by<br>model | Missing data Assumes I handled by missing at 1 | | Patients who died before Week 52 would have expected a poor outcome |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Analysis | Patient subset 3 but alive at Wee | | Patient subset 4: No FVC result<br>but died Week 52 | |
|---|---|---|---|---|
| | Handling of missing FVC | Underlying assumption | Handling of missing FVC | Underlying assumption |
| | | patients who did not discontinue. | | |
| Sensitivity<br>analysis 1 | Retrieve dropout: based on the point estimates for drug and placebo in patient subset 2. | Patients without<br>a result would<br>have behaved<br>similarly to<br>discontinued<br>patients with a<br>result who are<br>in the same<br>treatment group | Impute based on 10 <sup>th</sup> percentile <sup>1</sup> of all observed values (change from baseline) in each treatment arm at each visit | Patients who died before Week 52 would have expected a poor outcome. |
| Sensitivity analysis 2 | Follow reference: based on the point estimates for all placebo patients in patient subset 1 & 2. | Patients without<br>a result would<br>have behaved<br>similarly to all<br>patients in the<br>placebo arm | | |

<sup>&</sup>lt;sup>1</sup> selected based on pooled INPULSIS I/II data to reflect a negative outcome, while retain estimation efficiency by avoiding extreme values.

In the analysis of all other continuous endpoints, missing data will not be imputed. The mixed effect model will handle missing data based on a likelihood method under the "missing at random assumption".

In the primary analysis of time-to-event endpoints, missing or incomplete data will be handled using standard survival analysis techniques (i.e. censoring), except for death which will be handled as event.

Additional details on the handling of missing data and sensitivity analysis will be specified in the TSAP prior to unblinding.

### 7.3.2 Safety endpoints

Missing or incomplete AE dates will be imputed according to BI standards. Other missing safety data will not be imputed.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.4 RANDOMIZATION

Patients will be parallel randomized in blocks to double-blind treatment. The randomization will be stratified by intake of AF treatment at baseline (Yes/No), within the IRT system. Approximately equal numbers of patients will be randomized to BI 101550 18 mg bid, BI 1015550 9 mg bid and placebo in a 1:1:1 ratio. For patients to be enrolled and randomized after a potential futility stop of the low dose level (9 mg; see Section 7.2.8), the randomization ratio will be 1:1 (BI 1015550 18 mg bid vs. Placebo).

BI will arrange for the randomization and the packaging and labelling of trial medication. The randomization list will be generated using a validated system, which involves a pseudorandom number generator so that the resulting treatment will be both reproducible and non-predictable. The block size will be documented in the Clinical Trial Report. Access to the codes will be controlled and documented.

### 7.5 DETERMINATION OF SAMPLE SIZE

Results from the Phase II trial 1305-0013 show substantial improvement of BI 1015550 over placebo in FVC change from baseline to Week 12. Given the uncertainty of whether a similar progressive patient population will be recruited in the current trial, for trial 1305-0014 in IPF patients, a target treatment effect of 110 mL in FVC decline at Week 52 compared to Placebo, as seen in the pooled INPULSIS trials is assumed for patients receiving BI 1015550 and not on antifibrotic background therapy.

No data on the treatment effect beyond 12 weeks on top of antifibrotics is available. However, the maximum treatment effect on top of antifibrotics is limited by the natural agerelated decline in FVC. Therefore, assuming FVC decline at 52 weeks is 110 mL in the placebo arm for patients on antifibrotic background therapy, a lower treatment effect of 65 mL is assumed for BI 1015550 in patients on background antifibrotic therapy. 70% of patients are expected to be on background antifibrotic treatment.

Additionally, 25% of Placebo patients not on antifibrotic treatment, are expected to initiate antifibrotic therapy on average at Week 26 and 12.5% of BI 1015550 patients not on AF treatment expected to switch AF treatment after 26 weeks. Under the linearity assumption of FVC decline assumed treatment effect at Week 52 in patients not on background treatment will be reduced by 12.5%. Based on all above-mentioned assumptions, a treatment effect of 74 mL for BI 1015550 vs. placebo in FVC change from baseline at Week 52 is expected for trial 1305-0014. A common adjusted standard deviation (SD) of FVC change of 280 mL is assumed based on estimates from INPULSIS trials.

An effective sample size of 310 patients per group, will detect a treatment effect of 74 mL with 91% power under two-sided alpha of 5% for one active BI 1015550 dose arm vs. placebo. With 310 patients per arm and a two-sided type I error rate of 0.05, a treatment effect size of 90, 65, 55, and 45 can be detected for each of the primary endpoint with 98%, 82%, 69%, and 52% power respectively.

Calculations were performed using R Version 4.0.2.

Boehringer Ingelheim BI Trial No.: 1305-0014 c39145241-04

20 Sep 2023


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Clinical Trial Protocol** 

For the key secondary endpoint time to first acute IPF exacerbation, first hospitalization for respiratory cause or death, assumptions for the power calculations are derived from the pivotal INPULSIS trials (1199-0032 and 1199-0034) and patients with UIP-like fibrotic pattern from the INBUILD trial (1199-0247). The proportion of Placebo patients with at least one event of the composite outcome observed until Week 52 was 17.5% for pooled INPULSIS patients and was estimated as 18.3% for patients with a UIP-like fibrotic pattern in INBUILD. In order to reflect potential differences in the trial population of 1305-0014, scenarios including 15%, 17.5%, and 20% are presented in the power calculations. As the treatment effect on the key secondary endpoint is unknown, the power was evaluated for hazard ratios in the range of 0.60 to 0.75 for the treatment effect of BI 1015550 vs. placebo over the duration of the trial. Accrual time for 1305-0014 is expected to be 15 to 18 months with a follow-up period of 12 months. Table 7.5: 1 provides power calculations for time to first acute IPF exacerbation, first hospitalization for respiratory cause or death on different combined scenarios. Power calculations assuming a 1:1:1 randomization for an effective sample size of 310 patients per arm with linear accrual rate have been performed based on a two-sided Log-rank test comparing BI 1015550 18 mg bid vs. placebo, with a significance level of 5%. No correction for dropouts has been incorporated into the power calculation for the key secondary endpoint.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.5: 1 Power evaluation for secondary endpoint based on a two-sided, two-sample Log-rank test with a significance level of 5% considering different effect sizes, event rates and accrual time

| 52 week event rate<br>for key secondary<br>endpoint (placebo) | Hazard Ratio | Accrual time in months | Expected number<br>of events/Local<br>Power <sup>1</sup> |
|---|---|---|---|
| 15% | 0.75 | 15 | 127/37% |
| 15% | 0.70 | 15 | 124/51% |
| 15% | 0.65 | 15 | 120/66% |
| 15% | 0.60 | 15 | 117/79% |
| 17.5% | 0.75 | 15 | 147/42% |
| 17.5% | 0.75 | 18 | 157/44% |
| 17.5% | 0.70 | 15 | 144/57% |
| 17.5% | 0.70 | 18 | 153/60% |
| 17.5% | 0.65 | 15 | 140/72 % |
| 17.5% | 0.65 | 18 | 149/75% |
| 17.5% | 0.60 | 15 | 136/85% |
| 17.5% | 0.60 | 18 | 144/87% |
| 20% | 0.75 | 15 | 167/46% |
| 20% | 0.70 | 15 | 163/62% |
| 20% | 0.65 | 15 | 159/77% |
| 20% | 0.60 | 15 | 154/89% |

numbers reflecting comparison between one active dose arm and placebo arm

Based on the range of plausible assumptions and hazard ratios considered, local power of the key secondary ranges from 37%-46% for a hazard ratio of 0.75 to around 79%-89% for a hazard ratio of 0.6 as often targeted in pivotal trials.

Calculations were performed using "rpact" package version 3.0.4 in R version 4.0.2.

As a graphical testing procedure is used for the hypothesis tests in this Phase III trial and the controlled one-sided type I error rate for each hypothesis test depends on the result of other endpoints, it is very complicated, if not impossible, to derive the mathematical formula for the power of each efficacy endpoints considered in the graphical testing procedure. As a result, we conducted simulations to approximate the power for each efficacy endpoint (i.e. the probability of rejecting each null hypothesis) using the graphical testing procedure under five different scenarios of the effect size for each efficacy endpoint and dose level with the proposed graph. 310 effective patients per arm, two-sided family-wide type I error rate of 0.05, and 0.4 correlation among efficacy endpoints. The probability of rejecting at least one dose in primary endpoint, namely  $H_{01}$  or  $H_{02}$ , as well as the probability of rejecting both primary and secondary endpoint for high dose are calculated.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Simulation results as presented in Table 7.5: 2 suggest that with 310 effective sample size per arm, there is at least 93% power to detect an effect size of 74 mL in FVC change from baseline at Week 52 for at least one dose is significant (Scenario #1). Regardless of effect size of the 9 mg bid arm, probability of detecting a significant FVC effect of 74 mL in the 18 mg bid arm is between 89% to 90%. Furthermore, if 18 mg bid arm has an effect of 74 mL in primary endpoint and HR of 0.6 in key secondary endpoint, the probability of rejecting both  $H_{01}$  and  $H_{03}$  is between 65% to 74% depending on relative effect size of the 9 mg bid arm. The simulation results also show a well controlled type-I error under the null hypothesis (Scenario #5) with the proposed testing strategy.

Additional simulation results, which are not displayed here, also show that the transition weight from  $H_{01}$  to  $H_{02}$  ranging from 0.5 to 0.7 does not impact the marginal power for the primary and key secondary efficacy endpoints much. Hence we choose 0.5 as the transition weight given desirable success probabilities of 88%-93% for primary endpoint and 65% to 74% for key secondary endpoint 18 mg bid arm under various conditions.

In summary with 310 effective patients per arm, simulation results show satisfactory operational characteristics of the proposed graphical testing procedure under Scenarios #1-5 which are considered plausible for this Phase III trial.

Table 7.5: 2 Multiplicity adjusted probabilities of success for each hypothesis and positive study under different scenarios of effect sizes from simulations.

| | 18 mg bid<br>FVC [mL]<br>change from<br>baseline at<br>Week 52 <sup>1</sup> | 9 mg bid<br>FVC [mL]<br>change from<br>baseline at<br>Week 52 <sup>1</sup> | 18 mg bid<br>time-to resp<br>hosp. or<br>exac. or<br>death <sup>2</sup> | 9 mg bid<br>time-to resp<br>hosp. or<br>exac. or<br>death <sup>2</sup> |
|---|---|---|---|---|
| Scenario #1<br>(both doses achieve<br>target effect) | 74 | 74 | 0.6 | 0.6 |
| Probability of rejecting each hypothesis | 90% | 87% | 75% | 63% |
| Probability of rejecting at least one dose primary endpoint | 94% | | | |
| Scenario #2<br>(low dose approx. 70%<br>of high dose) | 74 | 52 | 0.60 | 0.72 |
| Probability of rejecting each hypothesis | 90% | 60% | 71% | 30% |

**Clinical Trial Protocol** 

c39145241-04  Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 18 mg bid<br>FVC [mL]<br>change from<br>baseline at<br>Week 52 <sup>1</sup> | 9 mg bid<br>FVC [mL]<br>change from<br>baseline at<br>Week 52 <sup>1</sup> | 18 mg bid<br>time-to resp<br>hosp. or<br>exac. or<br>death <sup>2</sup> | 9 mg bid<br>time-to resp<br>hosp. or<br>exac. or<br>death <sup>2</sup> |
|---|---|---|---|---|
| Probability of rejecting at least one dose primary endpoint | 90% | | | |
| Scenario #3<br>(low dose approx. 50%<br>of high dose) | 74 | 37 | 0.60 | 0.80 |
| Probability of rejecting each hypothesis | 89% | 35% | 69% | 11% |
| Probability of rejecting at least one dose primary endpoint | 90% | | | |
| Scenario #4<br>(low dose no effect) | 74 | 0 | 0.60 | 1 |
| Probability of rejecting each hypothesis | 89% | 3.5% | 65% | 0.2% |
| Probability of rejecting at least one dose primary endpoint | 89% | , | | |
| Scenario #5<br>(null effect) | 0 | 0 | 1 | 1 |
| Probability of rejecting each hypothesis | 4.1% | 1.3% | 0.1% | <0.1% |
| Probability of rejecting at least one dose primary endpoint | 4.8% | | | |

Probability calculated based on 50 000 simulation iterations. Total alpha-level = 0.05 (two-sided), 1:1:1 randomization ratio with 310 patients per arm.

Calculations were performed using "rpact" package version 3.0.4 in R version 4.0.2.

<sup>[1]</sup> For FVC change from baseline at Week 52, SD assumed to be 280 mL.

<sup>[2]</sup> For composite endpoint: placebo event rate at 52 weeks = 17.5%, accrual period = 15 months, no dropout, correlation between endpoints for each dose = 0.4.

BI Trial No.: 1305-0014 c39145241-04

**Clinical Trial Protocol** 


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Based on the proportions of early treatment discontinuation, patients with missing data and missing data patterns as observed in our Phase II trial 1305-0013 and INBUILD trial, we project 20% patients will prematurely terminate treatment in our Phase III trial. Since BI will take every measure to collect all data at planned visits from early dropout, we anticipate 75% of these dropouts will have efficacy outcome collected after treatment termination and can be used for analysis. Based on these estimations, we assume a 5% rate for missing data. Furthermore, an information content of 0.34 estimated from pivotal INPULSIS trials, which provides average amount of information by a non-completing patient is assumed. Based on these estimations, we apply a 3.3% correction for missing data in sample size calculation for this Phase III trial. This gives the total number of 963 randomized patients, with 321 randomized patients in each treatment arm.

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU directive 2001/20/EC/EU regulation 536/2014, the Japanese GCP regulations (Ministry of Health and Welfare Ordinance No. 28, March 27, 1997) and other relevant regulations. Investigators and site staff must adhere to these principles. Deviation from the protocol, the principles of ICH GCP or applicable regulations as will be treated as "protocol deviation". Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains the responsibility of the treating physician of the patient.

The investigator will inform the sponsor or delegate immediately of any urgent safety measures taken to protect the trial patients against any immediate hazard, as well as of any serious breaches of the protocol or of ICH GCP.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. The rights of the investigator and of the Sponsor with regard to publication of the results of this trial are described in the investigator contract. As a rule, no trial results should be published prior to finalisation of the Clinical Trial Report.

The certificate of insurance cover is made available to the investigator and the patients and is stored in the ISF.

### 8.1 TRIAL APPROVAL, PATIENT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB)/Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations). The same applies for the implementation of changes introduced by amendments. Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The investigator or delegate must give a full explanation to trial patients based on the patient information form. A language understandable to the patient should be chosen, technical terms and expressions avoided, if possible.

The patient must be given sufficient time to consider participation in the trial. The investigator or delegate obtains written consent of the patient's own free will with the informed consent form after confirming that the patient understands the contents. The investigator or delegate must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent. Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

The consent and re-consenting process should be properly documented in the source documentation.

### 8.2 DATA QUALITY ASSURANCE

A risk-based approach is used for trial quality management. It is initiated by the assessment of critical data and processes for trial subject protection and reliability of the results as well as identification and assessment of associated risks. An Integrated Quality and Risk Management Plan or alternative plan, in line with the guidance provided by ICH Q9 and ICH-GCP E6, for fully outsourced trials, documents the rationale and strategies for risk management during trial conduct including monitoring approaches, vendor management and other processes focusing on areas of greatest risk.

Continuous risk review and assessment may lead to adjustments in trial conduct, trial design or monitoring approaches.

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB/IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

### 8.3 RECORDS

CRFs for individual patients will be provided by the sponsor. See Section <u>4.1.5.2</u> for rules about emergency code breaks. For drug accountability, refer to Section <u>4.1.8</u>.

### **8.3.1** Source documents

For adverse events, an end date may not always be available (e.g. due to hospital discharge and later recovery, or change in treating physician), but should be recorded in the source if known.

For eCRF all data need to be derived from source documents, which need to be available onsite (this could be for example physician's notes in patient files, printouts, patient diaries).

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In accordance with regulatory requirements, the investigator should prepare and maintain adequate and accurate source documents and trial records that include all observations and other data pertinent to the investigation on each trial patient. Source data as well as reported data should follow the "ALCOA principles" and be attributable, legible, contemporaneous, original and accurate. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

The current medical history of the patient may not be sufficient to confirm eligibility for the trial and the investigator may need to request previous medical histories and evidence of any diagnostic tests. In this case, the investigator must make at least one documented attempt to retrieve previous medical records. If this fails, a verbal history from the patient, documented in their medical records, would be acceptable.

Copies of source documents necessary for evaluation of adverse events will be provided to the adjudication committee members or the pharmacovigilance department. Before sending or uploading those copies, the investigator must ensure that all patient identifiers (e.g. patient's name, initials, address, phone number, social security number) have properly been removed or redacted from any copy of the patients' source documents.

If the patient is not compliant with the protocol, any corrective action e.g. re-training must be documented in the patient file.

For the CRF, data must be derived from source documents, for example:

- Patient identification: gender, year of birth (in accordance with local laws and regulations)
- Patient participation in the trial (substance, trial number, patient number, date patient was informed)
- Dates of patient's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- Medication history
- Adverse events and and outcome events (onset date (mandatory), and end date (if available))
- Serious adverse events (onset date (mandatory), and end date (if available))
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results and other imaging or testing results, i.e. chest HRCT or biopsy reports, DLCO report with proper documented medical evaluation (in validated electronic format, if available)
- Patient-reported outcome forms and C-SSRS questionnaire if done on paper
- Completion of patient's participation in the trial" (end date; in case of premature discontinuation document the reason for it).
- Prior to allocation of a patient to a treatment into a clinical trial, there must be documented evidence in the source data (e.g. medical records) that the trial participant meets all inclusion criteria and does not meet any exclusion criteria. The absence of records (either medical records, verbal documented feedback of the patient or testing conducted specific for a protocol) to support inclusion / exclusion criteria does not make the patient eligible for the clinical trial.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For the spirometry, electronic patient-reported outcomes and C-SSRS questionnaire data will be transferred to the data base from the respective vendor and the electronic records are regarded as source documents.

### 8.3.2 Direct access to source data and documents

The investigator / institution will allow site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents / data, including progress notes, copies of laboratory and medical test results, which must always be available for review by the CRA, auditor and regulatory inspector (e.g. FDA). They may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor or delegate will also monitor compliance with the protocol and GCP.

### 8.3.3 Storage period of records

### Trial sites:

The trial sites must retain the source and essential documents (including ISF) according to contract or the local requirements valid at the time of the end of the trial (whatever is longer).

### Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal and regulatory reporting obligation in accordance with regulatory requirements.

### 8.5 STATEMENT OF CONFIDENTIALITY AND PATIENT PRIVACY

Data protection and data security measures are implemented for the collection, storage and processing of trial participant data in accordance with the principles 7 and 12 of the WHO GCP handbook.

To ensure confidentiality of records and personal data, only pseudonymised data will be transferred to the sponsor by using a patient identification number instead of the patient's name. The code is only available at the site and must not be forwarded to the sponsor. In case patient's records will be forwarded e.g. for SAE processing or adjudication committees, personal data that can identify the patient will be redacted by the site prior to forwarding. Access to the patient files and clinical data is strictly limited: personalised treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated at the site as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

A potential data security breach will be assessed regarding the implications for rights and privacy of the affected person(s). Immediate actions as well as corrective and preventive actions will be implemented. Respective regulatory authorities, IRBs / IECs and patients will be informed as appropriate.

c39145241-04  Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, biobanking and future use of biological samples and clinical data, in particular

- Sample and data usage have to be in accordance with the separate biobanking informed consent
- The BI-internal facilities storing biological samples from clinical trial participants as well as the external banking facility are qualified for the storage of biological samples collected in clinical trials
- An appropriate sample and data management system, incl. audit trail for clinical data and samples to identify and destroy such samples according to ICF is in place
- A fit for the purpose documentation (biomarker proposal, analysis plan and report) ensures compliant usage
- A fit for purpose approach will be used for assay/equipment validation depending on the intended use of the biomarker data
- Samples and / or data may be transferred to third parties and other countries as specified in the biobanking ICF

### 8.6 TRIAL MILESTONES

The **start of the trial** is defined as the date when the first patient in the whole trial signs informed consent.

The end of the trial is defined as the date of the last visit of the last patient in the whole trial ("Last Patient Completed").

The "Last Patient Last Treatment" (LPLT) date is defined as the date on which the last patient in the whole trial is administered the last dose of trial treatment (as scheduled per protocol or prematurely). Individual investigators will be notified of SUSARs occurring with the trial medication until 30 days after LPLT at their site. Early termination of the trial is defined as the premature termination of the trial due to any reason before the end of the trial as specified in this protocol.

**Temporary halt of the trial** is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

Suspension of the trial is defined as an interruption of the trial based on a Health Authority

The IEC / competent authority in each participating EU member state will be notified about the trial milestones according to the respective laws.

A final report of the clinical trial data will be written only after all patients have completed the trial in all countries (EU or non-EU) to incorporate and consider all data in the report. The sponsor will submit to the EU database a summary of the final trial results within one year from the end of a clinical trial as a whole, regardless of the country of the last patient (EU or non-EU).

### 8.7 ADMINISTRATIVE STRUCTURE OF THE TRIAL

The trial is sponsored by Boehringer Ingelheim (BI).

### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

A Coordinating Investigator is responsible to coordinate investigators at the different sites participating in this trial. Tasks and responsibilities are defined in a contract.

A Steering Committee (SC) consisting of independent experts and sponsor representatives will be established to support the Coordinating Investigator who will be the chair of the SC. The composition of the SC will be documented in the TMF. The tasks and responsibilities will be agreed in contracts between the SC members and the sponsor and summarised in a SC charter.

A DMC will be established. Members of the DMC are independent of BI, they are physicians experienced in the treatment of the disease under investigation and a statistician. The DMC will evaluate safety data on a regular basis and perform the interim analysis. While DMC members may be unblinded, measures are in place to ensure the blinding for everyone else involved in the trial. Regular DMC meetings will be held at specified intervals. The DMC will recommend continuation, modification or termination of the trial as detailed in the DMC charter. DMC recommendations as well as the final BI decision will be reported to the appropriate Regulatory Authorities (RAs)/Health Authorities (HAs), IRBs/ECs, and to investigators as requested by local law. The tasks and responsibilities of the DMC are specified in a charter.

An independent adjudication committee will review all fatal cases and adjudicate all deaths due to cardiac or respiratory causes. The adjudication committee will a will also review all adverse events categorized as major adverse cardiovascular events (MACE). A separate independent adjudication committee will review all events suspicious for vasculitis.

Relevant documentation on the participating (Principal) Investigators (e.g. their curricula vitae) will be filed in the ISF.

The investigators will have access to the BI web portal Clinergize to access documents provided by the sponsor.

BI has appointed a Clinical Trial Leader responsible for coordinating all required activities, in order to

- manage the trial in accordance with applicable regulations and internal SOPs,
- direct the clinical trial team in the preparation, conduct, and reporting of the trial,
- ensure appropriate training and information of Clinical Trial Managers (CT Managers), Clinical Research Associates (CRAs), and investigators of participating countries.

Data Management and Statistical Evaluation will be done by BI according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

A central laboratory service, a central images service, a central ePRO service, a central spirometry service, a central patient and site engagement service and an IRT vendor will be used in this trial. Details will be provided in the respective vendor specific instruction manuals as applicable, in the ISF.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9. REFERENCES

### 9.1 PUBLISHED REFERENCES

- P11-07084 Raghu G, et al. ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med 2011;183(6):788-824.
- P12-03241 King TE, Pardo A, Selman M. Idiopathic pulmonary fibrosis. Lancet 2011;378(9807):1949-1961.
- P15-07362 Raghu G, et al. ATS, ERS, JRS, and ALAT. An official ATS/ERS/JRS/ALAT clinical practice guideline: treatment of idiopathic pulmonary fibrosis: executive summary: an update of the 2011 clinical practice guideline. Am J Respir Crit Care Med 2015;192(2):238-248.
- P16-06899 Collard HR, Ryerson CJ, Corte TJ, et al. Acute exacerbation of idiopathic pulmonary fibrosis: an international working group report. American Journal of Respiratory and Critical Care Medicine, Article in press, published on 14-June-2016, doi: 10.1164/rccm.201604-0801CI; 2016. p. 265-275.
- P22-03204 Raghu G, Remy-Jardin M, Richeldi L, et al. American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, Asociacion Latinoamericana de Torax. Idiopathic pulmonary fibrosis (an update) and progressive pulmonary fibrosis in adults: an official ATS/ERS/JRS/ALAT clinical practice guideline. Am J Respir Crit Care Med 2022;205(9):e18-e47.
- R06-0638 Wang SK, Tsiatis AA. Approximately optimal one-parameter boundaries for group sequential trials. Biometrics 1987;43,193-199.
- R06-2002 Macintyre N, Crapo RO, Viegi G, et al. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J 2005;26(4):720-735.
- R10-1559 Giembycz MA. Life after PDE4: overcoming adverse events with dual-specificity phosphodiesterase inhibitors. Curr Opin Pharmacol 2005;5:238-244.
- R12-1920 Herdman M, Gudex C, Lloyd A, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res 2011;20:1727-1736.
- R16-4473 Bretz, F., Maurer, W., Brannath, W. and Posch, M. A graphical approach to sequentially rejective multiple test procedures. Statistics in Medicine (2009). 28, 586–604.
- R17-2617 Winthrop KL, Novosad SA, Baddley JW, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance. Ann Rheum Dis 2015;74:2107-2116.
- R17-2947 Maurer W, Bretz F. Multiple testing in group sequential trials using graphical approaches. Stat Biopharm Res 2013;5(4):311-320.

Boehringer Ingelheim BI Trial No.: 1305-0014

c39145241-04

20 Sep 2023

### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- R17-4075 Lynch DA, Sverzellati N, Travis WD, et al. Diagnostic criteria for idiopathic pulmonary fibrosis: a Fleischner Society White Paper. Lancet Respiratory Medicine, Published online November 15, 2017, doi: 10.1016/S2213-2600(17)30433-2; 2017.
- R18-2794 Raghu G, Remy-Jardin M, Myers JL, et al. American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, Latin American Thoracic Society. Diagnosis of idiopathic pulmonary fibrosis: an official ATS/ERS/JRS/ALAT clinical practice guideline. Am J Respir Crit Care Med 2018;198(5):e44-e68.
- R20-2419 Graham BL, Steenbruggen I, Miller MR, et al. American Thoracic Society, European Respiratory Society. Standardization of spirometry 2019 update: an official American Thoracic Society and European Respiratory Society technical statement. Am J Respir Crit Care Med 2019;200(8):e70-e88.
- R22-1856 Stern, A. F. The Hospital Anxiety and Depression Scale. Occup Med-c 64 2014, 393–394.
- R22-1857 Aronson, K. I. et al. Patient-centered Outcomes Research in Interstitial Lung Disease: An Official American Thoracic Society Research Statement. Am J Resp Crit Care 204 2021, e3–e23.
- R96-2382 EuroQol a new facility for the measurement of health-related quality of life. Health Policy 1990;16:199-208.

### 9.2 UNPUBLISHED REFERENCES

- c02094779 Investigator's Brochure 1305.P03. BI 1015550.
- c37065416 A randomised, double-blind, placebo-controlled parallel group study in IPF patients over 12 weeks evaluating efficacy, safety and tolerability of BI 1015550 taken orally. 1305-0013.
- c37934954 Population Pharmacodynamic Model for Forced Vital Capacity during BI 1015550 Treatment in Patients with Idiopathic Pulmonary Fibrosis.

c39145241-04 Clinical Trial Protocol


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10. APPENDICES

## 10.1 SPIROMETRY: BRONCHODILATOR WASHOUT RECOMMENDATIONS

Based on ATS/ERS 2019 guidelines [R20-2419] for the conduct of spirometry, the following washout of bronchodilators is recommended before spirometry (see Table 10.1: 1). According to the ongoing treatment, the investigator should advise the patient on the washout on/before the days of the onsite spirometry and document it in the source documents.

Table 10.1: 1 Minimal washout timeframes for bronchodilators before spirometry

| Bronchodilator Medication | Withholding Time |
|---|---|
| SABA (e.g., albuterol or salbutamol) | 4-6 hours |
| SAMA (e.g., ipratropium bromide) | 12 hours |
| LABA (e.g., formoterol or salmeterol) | 24 hours |
| Ultra-LABA (e.g., indacaterol, vilanterol, or olodaterol) | 36 hours |
| LAMA (e.g., tiotropium, umeclidinium, aclidinium, or glycopyrronium) | 36-48 hours |

c39145241-04 Clinical Trial Protocol


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.2 PATIENT-REPORTED OUTCOMES

### 10.2.1 Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (LPF)

### Instructions for Completing the Living with Pulmonary Fibrosis (L-PF) Symptoms Questionnaire

Complete this questionnaire to assess the symptoms you may have experienced from Pulmonary Fibrosis (PF) over the last 24 hours.

### Keep in mind:

- · you are not being asked to compare yourself to anyone else
- you are not being asked to compare how you are now with any time in the past

Items 1-12: The first 12 items ask about your symptoms in relation to physical activities, some of which you may not have done in the last 24 hours. If you did not perform an activity, we would like to know whether it was because you did not have the opportunity to do it (for example, maybe your home doesn't have stairs, so you did not walk up a flight of stairs), or whether you avoided the activity because it was too difficult.

If you did the stated activity, then reflect on the last 24 hours, and consider whether, on average, doing the activity at your usual pace or intensity level made you short of breath—and if so, how much.

If you normally use oxygen when you perform a given activity, then consider your response as if you were using supplemental oxygen.

Please select the box that best describes your experience.

| Did you get dressed in the last 24 hours? | |
|---|---|
| Yes | How short of breath did getting dressed make you? |
| | Not at all 0 1 2 3 4 Extremely |
| No | No I did not get dressed in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform | |
| B Not applicable, because I did not want or have the opportunity to do it | |

| 2. Did you walk up one flight of stairs in the last 24 hours? |
|---|
| How short of breath did walking up one flight of stairs make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not walk up one flight of stairs in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |
| <ol> <li>Over the last 24 hours, how short of breath have you been while sitting down, relaxing, reading, or<br/>watching TV?</li> </ol> |
| Not at all 0 1 2 3 4 Extremely |
| 4. Did you walk up a short, gradual incline (like a wheelchair ramp into a building) in the last 24 hours? |
| Yes How short of breath did walking up a short, gradual incline make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not walk up a short, gradual incline in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |
| 5. Did you perform a grooming activity (e.g., brush teeth, shave, fix hair) in the last 24 hours? |
| Yes How short of breath did grooming make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not perform a grooming activity in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |

| 6. Did you walk outside on a level surface (approximately 150 feet/45 meters, or the distance of half a typical city block) in the last 24 hours? |
|---|
| Yes How short of breath did walking outside on a level surface make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not walk outside on a level surface in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |
| 7. Did you walk from room to room inside your home in the last 24 hours? |
| Yes How short of breath did walking from room to room inside your home make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not walk from room to room inside my home in the last 24 hours because: |
| A I avoided this activity because it was too difficult to perform |
| B Not applicable, because I did not want or have the opportunity to do it |
| 8. Did you leave your home in the last 24 hours? |
| Yes How short of breath did getting ready to leave your home (e.g., find keys, put on coat, lock doors) make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not leave my home in the last 24 hours because: |
| A I avoided this activity because it was too difficult to perform |
| B Not applicable, because I did not want or have the opportunity to do it |

| 9. Did you bathe or shower in the last 24 hours? |
|---|
| Yes How short of breath did bathing or showering make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not bathe or shower in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |
| 10. Did you do light cleaning around the house in the last 24 hours? |
| Yes How short of breath did doing light cleaning around the house make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not do light cleaning around the house in the last 24 hours because: |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |
| 11. Over the last 24 hours, how short of breath were you after eating a meal or snacks? |
| Not at all 0 1 2 3 4 Extremely |
| Not at all 0 1 2 0 4 Extremely |
| 12. Did you lift and carry a light load (e.g., less than 10 lbs) a short distance (e.g., from one room to<br>another) in the last 24 hours? |
| Yes How short of breath did lifting and carrying a light load a short distance make you? |
| Not at all 0 1 2 3 4 Extremely |
| No I did not lift or carry a light load a short distance in the last 24 hours because: |
| Total not me of sany a ngirt load a short distance in the last 24 hours seconds. |
| I avoided this activity because it was too difficult to perform |
| Not applicable, because I did not want or have the opportunity to do it |

### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Items 13-18: Each item focuses on cough. Again, reflect on the last 24 hours as you

| consider where you are on | consider where you are on the scale between the two statements. | | | | |
|---|---|---|---|---|---|
| 13. Over the last 24 hours, how | v often did | you cougl | n? | | |
| Not at all | 0 1 | 1 2 | 3 | 4 | Constantly |
| If you chose "O | )", please s | skip to Ite | m 19. | | |
| 14. Over the last 24 hours, how | v often did | you coug | n when | you to | ok a deep breath? |
| Not at all | 0 | 1 2 | 3 | 4 | Constantly |
| 15. Over the last 24 hours, how | v often did | you cougl | when | you w | ere breathing hard or fast? |
| Not at all | 0 1 | 2 | 3 | 4 | Constantly |
| 16. Over the last 24 hours, how | v often did | you cough | when | you ov | er-exerted yourself? |
| Not at all | 0 1 | 2 | 3 | 4 | Constantly |
| 17. Over the last 24 hours, how | v often did | coughing | make y | ou sho | rt of breath? |
| Not at all | 0 1 | 2 | 3 | 4 | Constantly |
| 18. Over the last 24 hours, how | 18. Over the last 24 hours, how often did you feel an annoying tickle in your throat? | | | | |
| Not at all | 0 1 | 2 | 3 | 4 | Constantly |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

19-23: These items primarily focus on your energy level. Again, reflect on the last 24 hours as you consider where you are on the scale between the two statements.

| 19. Over the last 24 hours, how was your energy level? |
|---|
| Extremely low 0 1 2 3 4 Excellent |
| 20. Over the last 24 hours, of all that you wanted to get done, how much did you actually get done? Nothing 0 1 2 3 4 Everything |
| 21. Over the last 24 hours, how much energy did you have to do all the things you like to do? No energy 0 1 2 3 4 A lot |
| 22. Over the last 24 hours, how much did coughing have a negative effect on your energy? |
| No effect at all 0 1 2 3 4 A lot |
| 23. Did you become short of breath in the last 24 hours? Yes How long did it take you to recover when you became short of breath? No time at all 0 1 2 3 4 An extremely long time No Please continue to the next page. |

### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Finally, we would like to ask you 5 questions about your supplemental oxygen use.

| Oxygen Question 1. Do you ever use supplemental oxygen? (Place an "X" in one box) |
|---|
| yes → → proceed to Oxygen Question #2. |
| No → → skip Oxygen Questions 2-5 |
| Oxygen Question 2. I use supplemental oxygen (Place an "X" in one box) |
| only when I sleep (answer Oxygen Question #3) → only when I perform a physical activity (such as getting dressed or walking) (answer Oxygen Question #4) |
| ⇒ → when I sleep or perform a physical activity (such as getting dressed or walking) but not at rest (answer Oxygen Questions #3 and #4) |
| 4 → → all the time (answer Oxygen Questions #3-5) |
| Oxygen Question 3. When I sleep, I most often use an oxygen flow rate ofL/min. (Place an "X" in one box) |
| 0.5 1.0 1.5 2.0 2.5 3.0 3.5 4.0 4.5 5 6 7 8 9 10 11 12 >12 |
| Oxygen Question 4. When I perform a physical activity (such as getting dressed or walking), I most often use an oxygen flow rate ofL/min. (Place an "X" in one box) |
| 0.5 1.0 1.5 2.0 2.5 3.0 3.5 4.0 4.5 5 6 7 8 9 10 11 12 >12 |
| Oxygen Question 5. At <u>rest</u> , I most often use an oxygen flow rate ofL/min. (Place an "X" in one box) |
| 0.5 1.0 1.5 2.0 2.5 3.0 3.5 4.0 4.5 5 6 7 8 9 10 11 12 >12 |
| Thank you for taking the time to complete the L-PF Symptoms Questionnaire. |

c39145241-04 Clinical Trial Protocol


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Instructions for Completing the Living with Pulmonary Fibrosis (L-PF) Impacts Questionnaire

The goal of this questionnaire is to determine how Pulmonary Fibrosis affects your quality of life.

Quality of life refers to your perceptions of your overall position in life in relation to:

- · your goals and expectations
- · your standards and values
- · your concerns and judgments

Among other things, quality of life encompasses:

- your physical health (conditions/diseases, symptoms, therapies)
- · your psychological state (outlook, emotional well-being)
- · your level of independence
- the relationships you have with pertinent features of your environment

Reflect on your life: has Pulmonary Fibrosis affected your quality of life? As you respond to the items, reflect on your physical health, how you have been functioning, your psychological state, how you have been feeling, your level of independence, what you have done, and where you have gone over the last 7 days.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Items 1-16:** For these items, reflect on the **last 7 days** as you consider where you are on the scale between the two statements.

| Oı | average, over the last 7 | days | 98 | | | | |
|---|---|---|---|---|---|---|---|
| 1. | How much did shortness of b | reath p | revent | you fr | om doi | ng thin | gs you wanted to do? |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 2. | . How much did fear of becoming too short of breath limit your physical exertion? | | | | | | |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 3. | 3. How was your stamina when you exerted physically? | | | | | | |
| | Extremely poor | 0 | 1 | 2 | 3 | 4 | Excellent |
| 4. | How frustrated were you by | the tim | e it too | k you t | o com | plete a | physical activity? |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 5. | How frustrated were you by | the spe | ed it to | ook you | to con | nplete | a physical activity? |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 6. | How frustrated were you by | your ne | eed to r | est du | ing or | after c | ompleting a physical activity? |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 7. | How much did coughing emb | arrass | you? | | | | |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 8. | How much did coughing frust | trate yo | ou? | | | | |
| | Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

On average, over the last 7 days...

| 9. How much did coughing inter | rupt y | our con | versati | ons (in | persor | or on the phone)? |
|---|---|---|---|---|---|---|
| Never | 0 | 1 | 2 | 3 | 4 | All of the time |
| 10. How frightening was your coughing to you? | | | | | | |
| Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 11. How much was your cough a | proble | m for y | ou? | | | |
| Not at all | 0 | 1 | 2 | 3 | 4 | Extremely |
| 12. How much hassle or inconver | nience | has pul | monar | y fibros | is caus | ed you in your day-to-day life? |
| None | 0 | 1 | 2 | 3 | 4 | Alot |
| 13. How much did you have to re | est in th | e midd | lle of d | oing a s | imple | chore inside the house? |
| Not at all | 0 | 1 | 2 | 3 | 4 | A lot |
| 14. How much did you have to p | ace you | rself to | make | it thro | ugh the | day? |
| Not at all | 0 | 1 | 2 | 3 | 4 | A lot |
| 15. How much did it take to get yourself ready to leave the house? | | | | | | |
| Very little<br>time | 0 | 1 | 2 | 3 | 4 | Extremely long time |
| 16. How much were you forced t | o depe | nd on o | other p | eople t | o do th | ings for you? |
| Not at all | 0 | 1 | 2 | 3 | 4 | A lot |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Only five more...

For Items 17-19: Think broadly about your shortness of breath, cough and energy level over the last 7 days. Have these symptoms affected how you have felt physically? Psychologically? Have they disrupted your life? Or limited you in terms of what you would like to do or how you would like to do it? Now, please respond to Items 17-19.

### On average, over the last 7 days...

| 17. How has shortness of breath affected your quality of life? | | | | | |
|---|---|---|---|---|---|
| Made my quality of life extremely poor | 0 | 1 2 | 3 | 4 | No negative effect |
| 18. How much has your cough affected your quality of life? | | | | | |
| Made my quality of life extremely poor | 0 | 1 2 | 3 | 4 | No negative effect |
| 19. How much has your energy level affected your quality of life? | | | | | |
| Made my quality of life 0 1 2 3 4 No negative effect extremely poor | | | | | |

For these last two Items: Think broadly again about whether Pulmonary Fibrosis has affected you and your quality of life over the last 7 days. Reflect on your symptoms and other aspects of your physical health, how you have been functioning, your psychological state, how you have been feeling, your level of independence, what you have done, and where you have gone over the last 7 days.

### On average, over the last 7 days...

| 20. How have you felt in terms of physic | al heal | lth? | | | |
|---|---|---|---|---|---|
| Extremely poor 0 | 1 | 2 | 3 | 4 | Excellent |
| 21. How has your quality of life been? | | | | | |

The end.

Thank you for taking the time to complete the L-PF Impacts Questionnaire.

### 10.2.2 EuroQol 5-Dimensional quality of life Questionnaire (EQ-5D)

This trial uses the English version for the United Kingdom [R12-1920].

20 Sep 2023

**Clinical Trial Protocol** 


| Under each heading, please check the ONE box that best describ | es your health TODAY. |
|---|---|
| MOBILITY | |
| I have no problems walking | |
| I have slight problems walking | |
| I have moderate problems walking | |
| I have severe problems walking | |
| I am unable to walk | |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | |
| I have extreme pain or discomfort | |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- · We would like to know how good or bad your health is TODAY.
- . This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- . Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =




Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.2.3 Hospital Anxiety and Depression Scale (HADS)

| | | Name: | Date: | | |
|---|---|---|---|---|---|
| | FOLD HERE | Clinicians are aware that emotions play an important these feelings he or she will be able to help you more. This questionnaire is designed to help your clinician underline the reply which comes closest to how yo numbers printed at the edge of the questionnaire. Don't take too long over your replies, your immedian accurate than a long, thought-out response. | to know how you feel. Read each item below and<br>u have been feeling in the past week. Ignore the | FOLD HERE | |
| A | D | | | A | ] |
| 3<br>2<br>1<br>0 | | I feel tense or "wound up" Most of the time A lot of the time From time to time, occasionally Never | I feel as if I am slowed down<br>Nearly all the time<br>Very often<br>Sometimes<br>Never | | |
| | 0<br>1<br>2<br>3 | I enjoy the things I used to enjoy<br>Definitely<br>Not quite so much<br>Only a little<br>Hardly at all | I get a sort of anxious feeling like<br>"butterflies" in the stomach<br>Never<br>Occasionally<br>Often<br>Very often | 0<br>1<br>2<br>3 | |
| 3<br>2<br>1<br>0 | | I get a sort of frightened feeling as if<br>something awful is about to happen<br>Very definitely and fairly badly<br>Yes, but not too badly<br>Sometimes, but it doesn't worry me<br>Never | I have lost interest in my appearance<br>Definitely<br>Often I don't take as much care as I should<br>Sometimes I don't take as much care as I should<br>I take just as much care as ever | | |
| | 0<br>1<br>2<br>3 | I can laugh and see the funny side of things<br>As much as I always could<br>Not quite so much now<br>Definitely not so much now<br>Never | I feel restless as if I have to be on the move<br>Definitely<br>Quite a lot<br>Not very much<br>Never | 3<br>2<br>1<br>0 | |
| 3<br>2<br>1<br>0 | | Worrying thoughts go through my mind<br>A great deal of the time<br>A lot of the time<br>Not too often<br>Almost never | I look forward with enjoyment to things<br>As much as I ever have<br>Somewhat less than I used to<br>Much less than I used to<br>Rarely | | |
| | 3<br>2<br>1<br>0 | I feel cheerful Never Not often Sometimes Most of the time | I get sudden feelings of panic<br>Very often<br>Often<br>Not very often<br>Never | 3<br>2<br>1<br>0 | |
| 0 1 2 3 | | I can sit at ease and feel relaxed<br>Always<br>Usually<br>Not often<br>Never | I can enjoy a good book, radio or<br>television program<br>Often<br>Sometimes<br>Not often<br>Very seldom | | |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10.2.4 Patient's Global Impression of Severity (PGIS) for Cough, Shortness of Breath, and Fatigue

### Cough

| Please think about cough and reflect on the last 7 days: call to mind whether you have had a cough and |
|---|
| if so, how frequently it has occurred, how severe it has been, and whether cough has affected how you |
| feel and how you function in your daily life. |

| Considering all these, | please rate the severity | of your cough over | the last 7 days by | placing a tic in the |
|---|---|---|---|---|
| one box correspondir | ng to your response: | | | |

| □ <sub>(0)</sub> | (1) | □ <sub>(2)</sub> | □ <sub>(3)</sub> | □ <sub>(4)</sub> | □ <sub>(5)</sub> |
|---|---|---|---|---|---|
| Not present | Very mild | Mild | Moderate | Severe | Very severe |

### Shortness of breath

Please think about <u>shortness of breath</u> and reflect on the last 7 days: call to mind how severe it has been and whether shortness of breath has affected how you feel and how you function in your daily life.

Considering all these, please rate the severity of your shortness of breath over the last 7 days by placing a tic in the one box corresponding to your response:

| (o) | <b></b> (1) | □ <sub>(2)</sub> | □(3) | <b>(4)</b> | □ <sub>(5)</sub> |
|---|---|---|---|---|---|
| Not present | Very mild | Mild | Moderate | Severe | Very severe |

### **Fatigue**

Please choose the response below that best describes the overall severity of your fatigue over the past 24 hours.

(Select one response)

| No symptoms | Mild | Moderate | Severe | Very severe |
|-------------|------|----------|--------|-------------|

### 10.3 COLUMBIA SUICIDAL SEVERITY RATING SCALE (C-SSRS)

The C-SSRS is a brief measure which is designed to assess severity and change of suicidality by integrating both, behavior and ideation. The C-SSRS was designed to address the need for a summary measure to track change in the severity of suicidality across both clinical settings and treatment trials.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The C-SSRS interview may be administered by any type of physician, psychologist, clinical social worker, mental health counsel, nurse, or coordinator with C-SSRS training. It has a typical duration of five minutes and causes only a low burden on patients. At a minimum, the interview consists of 2 screening questions related to suicidal ideation and 4 related to suicidal behavior and may be expanded to up to 17 items in case of positive responses. Free text entries are allowed for; the investigator has to directly evaluate the scale and write a report.

The investigator is to review all positive and negative reports for plausibility and clinical relevance. Doubtful reports may be validated by a consulting psychiatrist. If there is a confirmed positive report of suicidal behavior or suicidal ideation type 4 or 5 after start of trial, the investigator is to immediately interview the patient during the clinic visit and/or is to consult a psychiatrist. If the positive report is confirmed, appropriate actions for the patient's safety have to be initiated.

At screening, C-SSRS (screening/baseline version) will be used with the aim to exclude patients with suicidal ideation type 4 to 5 within the preceding 3 months or at Visit 1 or any suicidal behaviour in the past 2 years.

Subsequently, the C-SSRS "since last visit" will be performed at the time points given in the flow chart.

All positive reports during trial treatment are treatment-emergent adverse events (AEs). The results of further medical, including psychiatric examinations, should be documented as adverse events where appropriate.

The original Columbia Suicidal Severity Rating scales used in this trial are attached in the following appendix sections.

c39145241-04  Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.3.1 **Visit 1 – Screening/baseline version**

# **COLUMBIA-SUICIDE SEVERITY RATING SCALE** (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

| Definitions of behavioral suicidal events in this developed by | scale are based on those used in <u>The Columbia Suicide History Form</u> , Conte Center for the Neuroscience of Mental Disorders |
|---|---|
| , , | e, 1051 Riverside Drive, New York, NY, 10032. |
| the property of the contract o | icidal behavior: utility and limitations of research instruments. In M.B. First |
| Ed.] Standardized Evaluation in Clinical Pra | |
| For reprints of the C-SSRS contact | New York State Psychiatric Institute, 1051 Riverside Drive, New |
| York, New York, 10032; inquiries and training | |
| © 2008 The Re | search Foundation for Mental Hygiene, Inc. |

#### c39145241-04

| SUICIDAL IDEATION | | | | | | |
|---|---|---|---|---|---|---|
| Ask questions 1 and 2. If both are negative, question 2 is "yes", ask questions 3, 4 and 3 "Intensity of Ideation" section below. | | | He/S | ne: Time<br>She Felt<br>Suicidal | Past<br>Mon | |
| Wish to be Dead Subject endorses thoughts about a wish to be dead or n Have you wished you were dead or wished you could; | | | Yes | No | Yes | No |
| If yes, describe: | | | | | | |
| 2. Non-Specific Active Suicidal Thoughts<br>General non-specific thoughts of wanting to end one's<br>ways to kill oneself'associated methods, intent, or plan<br>Have you actually had any thoughts of killing yoursel | during the assessment pe | , "I've thought about killing myself") without thoughts of eriod. | Yes | No | Yes | No |
| If yes, describe: | | | | | | |
| plan with time, place or method details worked out (e.g | f at least one method dur<br>t, thought of method to k<br>ade a specific plan as to | out Intent to Act ring the assessment period. This is different than a specific cill self but not a specific plan). Includes person who would when, where or how I would actually do tt and I would | Yes | No | Yes | No |
| If yes, describe: | | | | | | |
| 4. Active Suicidal Ideation with Some Inter<br>Active suicidal thoughts of killing oneself and subject to<br>but I definitely will not do anything about them."<br>Have you had these thoughts and had some intention | reports having some inter | pecific Plan nt to act on such thoughts, as opposed to "I have the thoughts | Yes | No | Yes | No |
| If yes, describe: | | | | | | |
| 5. Active Suicidal Ideation with Specific Pla<br>Thoughts of killing oneself with details of plan fully or<br>Have you started to work out or worked out the detail. | partially worked out and | | Yes | No | Yes | No |
| If yes, describe: | | | " | П | | |
| INTENSITY OF IDEATION | | | | | | |
| The following features should be rated with resp.<br>the least severe and 5 being the most severe). As | | type of ideation (i.e.,1-5 from above, with 1 being as feeling the most suicidal. | | | | |
| <u>Lifetime</u> - Most Severe Ideation: | Type # (1-5) | Description of Ideation | Mos | t Severe | | ost<br>vere |
| Past X Months - Most Severe Ideation: | Type # (1-5) | Description of Ideation | | | | |
| Frequency How many times have you had these thought (1) Less than once a week (2) Once a week | s? | 2 500000782 St 197000 St 18 12 | | _ | _ | _3 |
| Duration When you have the thoughts how long do the (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | ry last? | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | ) | _ | _ | _== |
| Controllability | 16 | | | | 1 | |
| Could/can you stop thinking about killing you<br>(1) Easily able to control thoughts<br>(2) Can control thoughts with little difficulty<br>(3) Can control thoughts with some difficulty | urself or wanting to | (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | 8 | _ | - | _ |
| Deterrents Are there things - anyone or anything (e.g., facting on thoughts of committing suicide? (1) Deterrents definitely stopped you from atte (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | 2 ST ST | of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | Accept | | - | _ |
| Reasons for Ideation | | | | | | |
| | you couldn't go on | die or killing yourself? Was it to end the pain or<br>living with this pain or how you were feeling) or<br>h? | | | | |
| (1) Completely to get attention, revenge or a reacti (2) Mostly to get attention, revenge or a reacti (3) Equally to get attention, revenge or a reacti end/stop the pain | eaction from others<br>on from others | (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (0) Does not apply | | _ | _ | |


| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | | Life | time | Past<br>Yea | |
|---|---|---|---|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as no neself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger wh mouth but gun is broken so no injury results, this is considered an attempt. Inferring Intent. Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fir a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be infer thave you made a suicide attempt? Have you done anything to harm yourself? | a actual suicide<br>ile gun is in<br>. For example,<br>om window of | Yes | No | Yes | No |
| Have you done anything dangerous where you could have died? What did you do? Did you as a way to end your life? Did you want to die (even a little) when you ? | | | l # of<br>mpts | Total<br>Atten | |
| Were you trying to end your life when you? Or did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | , feel better, | Yes | No | Yes | No. |
| | | 163 | | 165 | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual would have occurred). | ıl attempt | Yes | N₀ | Yes | No |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather tha attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulli Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopp before you actually did anything? If yes, describe: | ng trigger.<br>down from | | l#of<br>rupted | Total<br>intern | |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in a destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being something else. | ny self-<br>stopped by | Yes | No | Yes | No |
| Has there been a time when you started to do something to try to end your life but you stopped yourself b actually did anything? If yes, describe: | efore you | | l # of<br>orted | Total<br>abor | |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting a gun, giving valuables away or writing a suicide note)? If yes, describe: | way, writing a | Yes | No | Yes | No |
| Suicidal Behavior: | | Yes | No | Yes | No |
| Suicidal behavior was present during the assessment period? | | | | | |
| Answer for Actual Attempts Only | Most Recent<br>Attempt<br>Date: | Most L<br>Attemp<br>Date: | | Initial/Fi<br>Attempt<br>Date: | |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | Enter Code | Enter | Code | Enter ( | Code |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury | | Enter | Code | Enter ( | Code |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | 79 | 14 | |


c39145241-04

**Clinical Trial Protocol** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.3.2 C-SSRS – since last visit

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

| Definitions of behavioral | suicidal events in this scale | e are based on those used in <b>The Columbia Suicide History For</b> |
|---|---|---|
| developed by | and | Conte Center for the Neuroscience of Mental Disorders |
| (CCNMD), New York St | ate Psychiatric Institute, 10 | 051 Riverside Drive, New York, NY, 10032. |
| | Risk factors for suicida | of behavior: utility and limitations of research instruments. In M.B. First |
| [Ed.] Standardized Eval | uation in Clinical Practic | е, рр. 103 -130, 2003.) |
| For reprints of the C-SSF | S contact | New York State Psychiatric Institute, 1051 Riverside Drive, New |
| | inquiries and training requ | |

© 2008 The Research Foundation for Mental Hygiene, Inc.

#### c39145241-04

| SUICIDAL IDEATION | | et e | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suic ask questions 3, 4 and 5. If the answer to question 1 and/or 2 | | Since<br>Vi | |
| <ol> <li>Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or a Have you wished you were dead or wished you could go to sleep and not w </li> </ol> | | Yes | No |
| If yes, describe: | | 00000 | (22) |
| 2. Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit suicide ( onesell'associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | e.g., "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| If yes, describe: | | | |
| | during the assessment period. This is different than a specific plan with time, not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Active suicidal thoughts of killing oneself and subject reports having some iwill not do anything about them". Have you had these thoughts and had some intention of acting on them? | t Specific Plan intent to act on such thoughts, as opposed to "I have the thoughts but I definitely intent to act on such thoughts," as opposed to "I have the thoughts but I definitely intent to act on such thoughts, as opposed to "I have the thoughts but I definitely intent to act on such thoughts," as opposed to "I have the thoughts but I definitely intent to act on such thoughts, as opposed to "I have the thoughts but I definitely intent to act on such thoughts," as opposed to "I have the thoughts but I definitely intent to act on such thoughts, as opposed to "I have the thoughts but I definitely intent to act on such thoughts," as opposed to "I have the thoughts but I definitely intent to act on such thoughts, as opposed to "I have the thoughts but I definitely intent to act on such thoughts," as opposed to "I have the thoughts but I definitely intent to act on such thoughts, as opposed to "I have the thoughts," as opposed to "I have the theological the " | Yes | No |
| If yes, describe: | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent<br>Thoughts of killing oneself with details of plan fully or partially worked out<br>Have you started to work out or worked out the details of how to kill yours | | Yes | No |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | | | |
| The following features should be rated with respect to the most severand 5 being the most severe). | ere type of ideation (i.e.,1-5 from above, with 1 being the least severe | Mo | ost |
| Most Severe Ideation: | 2 200 2 | Sev | ere |
| Type # (1-5) | Description of Ideation | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week | (4) Daily or almost daily (5) Many times each day | - | _ ;: |
| Duration When you have the thoughts how long do they last? | | | |
| (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | _ | - :: |
| Controllability Could/can you stop thinking about killing yourself or wanting (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | - | - |
| Deterrents | | | 123 |
| Are there things - anyone or anything (e.g., family, religion, per<br>thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide | nin of death) - that stopped you from wanting to die or acting on (4) Deterrents most likely did not stop you | | |
| (2) Deterrents probably stopped you<br>(3) Uncertain that deterrents stopped you | (5) Deterrents definitely did not stop you<br>(0) Does not apply | - | |
| Reasons for Ideation | | | |
| What sort of reasons did you have for thinking about wanting<br>you were feeling (in other words you couldn't go on living with | to die or killing yourself? Was it to end the pain or stop the way | | |
| revenge or a reaction from others? Or both? | inis pain or non you were feeling or was it to get attention, | | |
| (1) Completely to get attention, revenge or a reaction from others (2) Mostly to get attention, revenge or a reaction from others (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain | (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (0) Does not apply | ·- | - 22 |

c39145241-04

#### **Clinical Trial Protocol**


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Actual Attempt: Appennially self-impirous act committed with at least some wish to die, at a result of act. Behavior was in part thought of as method to kill one-self. Intent does not have to be 100%. If there is any intent/estimate to die associated with the act, then it can be considered an actual suicide stempt. There does not have to be 100%. If there is an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but nucide can be inferred et [e.g., gunshot to bead, jumping from window of a high floor/story). Alto, of someone denies ment to die, but they though that what they did could be lehal, intent may be inferred. Have you done anything dangerous where you could have died? What did you do? Did you made a suicide attempt? Have you done anything dangerous where you could have died? What did you do? Did you think it was possible you could have died from? Or Did you think it was possible you could have died from? Or did you do 1 purely for other reasons' without aNY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal ment) liye, describe. Yes 2 Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act iff not for that, acnual attempt would have occurred. Overdose Person has juit point and the strength of the potentially self-injurious act iff not for that, acnual attempt would have occurred. Overdose Person has pills in hand but it stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. When they may also the stempt strength and the potentially self-injurious act iff not for that, acnual attempt would have occurred. Overdose Person has puls pointed toward self, mis i | UICIDAL BEHAVIOR Theck all that apply, so long as these are separate events; must ask about all types) | Sir<br>Last | |
|---|---|---|---|
| If the you done anything to harm yourself? What did you do? Did you as a way to end your life? Did you want to die (even a little) when you? Or Did you think it was possible you could have died from? Or Did you think it was possible you could have died from? Or Did you think it was possible you could have died from? Or Did you think it was possible you could have died from? Or Did you think it was possible you could have died from? Or did you do it purely for other reasons / without AVY intention of killing yourself (like to relieve stress, feel better, get yangathy, or get something else to happen)? (Self-lajunious Behavior without suicidal intent) Yes 2 Gas subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act if/not for that, actual attempt would have controlled by the self-injurious and the down from heigh. Stangang Ferron has purely pointed own delf, gut is that sea way by onecone cle, or is somebow percented from polling miger. Once they pull the trigger, self-but has not yet started to hang, is stopped from doing to. If the there been at time when you started to do something to end your life but someone or something stopped you before you circumsly did anything? Yes, describe: When person begans to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Yes 1. Yes 2. Total # . Total # | potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent es not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual suicide attempt. There does not | 11.000 | No |
| Mixed did you do? Did you want to die (even a little) when you Per you triping to end your life when you Per you triping to end your life when you Per your triping to end your life when you Per your triping to end your life when you Per your triping to end your life when you Per your triping to end you could have died from Per your triping to end you could have died from Per your triping to end you could have died from Per your triping to end you could have died from Per did you do it purch for other reasons' without AV' Intention of killing yourself (like to relieve stress, feel better, get younguls), or get something else to happen)? (Self-Injurious Behavior? Interrupted Attempt: Wes 2 Interrupted Attempt: Wes 2 Interrupted Attempt: Wes 2 Interrupted Attempt: Wes 3 Interrupted by an outside circumstance) from starting the potentially self-injurious act if not for that, actual attempt would have corrected. Yes 2 Interrupted Attempt: Wes 3 Interrupted by an outside circumstance) from starting the potentially self-injurious act if not for that, actual attempt would have corrected from pulling trigger. Once they pull the trigger to the steps that a trigger to the steps to the steps to variety to the trigger to the steps to the steps to variety they are trigger to the trigger. Once they pull the trigger to the | ave you done anything to harm yourself? | T | |
| Did you want to die (ever a little) when you? Were you traing to end you riff when you? Or Did you think it was possible you could have died from? Pet did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get rempathy, or get something else to happen)? (Self-injurious Behavior without suicidal intent) Yes | | 100 | |
| Wes you trying to end your life when you? Or Did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) (yes, describe- life the person is interrupted thempt: Interrupted Attempt: Men the person is interrupted by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have coursed). Ves your fiften the person is interrupted by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have coursed). Ves your fiften the person is interrupted thempt. Person is interrupted attempt, the started to hang it is slaped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, the total to the intervious of the injurity is probled and then down from ledge. Hanging: Person has part to the total to this, it is attempt at the time of the injurity is probled and then down from ledge. Hanging: Person has to use to the total thange is slopped from doing to the three bears of the major is a three when you started to do something to end your life but someone or something stopped you before you cannot full did anything? Yes, describe. Whorted Attempt: Untered Attempt: Untered Attempt: Untered Attempt: Untered Attempt: Untered Attempt: Unter Attempt: Unter Description of the injurity of the injurit | | | |
| The fill you do it purely for other reasons / without AVN intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-injurious Behavior without suicidal intent) Yes Satisfact engaged in Non-Suicidal Self-Injurious Behavior without suicidal intention of the self-Injurious act (if not for that, actual attempt would have courseld) Yes Satisfact engaged in Injurious act in Injurious act (if not for that, actual attempt would have courseld) Yes Satisfact engaged in Injurious Behavior without suicidal injurious act (if not for that, actual attempt would have courseld. Injurious act (if not for that, actual attempt would have care of the season and the part of the season and the part of the season actually actual that with the part of the season actually actual that with the season actual behavior. Yes Satisfact the part of the season actual that in the individual stops him/bertelf instead of being stopped yourself before you actually did not part of the season actual that the individual stops him/bertelf instead of being stopped your | 500000 10000 LONG 10000 100000 10000 100000 10000 100000 10000 100 | _ | |
| In as subject engaged in Non-Suicidal Self-Injurious Behavior without suicidal intent) Yes, describe: Yes Sa subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: In the the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have verdous; Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, oncome person has pill in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, even if the gun fails to fire, it is an attempt. Jumping: Person is pointed to jump, is grabbed and taken down from ledge. Hanging: Person has noose around each but has not yet started to hang: its stopped from ong so. Its sthere been a time when you started to do something to end your life but someone or something stopped you before you cannot be a subject to the steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. It is at there been a time when you started to do something to try to end your life but you stopped yourself before you actually did my will have a subject to the steps toward making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a certification of preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, purchasing a gun) or preparing for one's death by suicide (e.g., griming things wany, writing a suicide note)? Yes of the proparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, preparing to kill yourself (such as collecting pills, getting a gun, preparing to kill yourself (such as collecting pills, getting a gun, preparing to kill yourself (such as collecting pills, getting as gun, or preparing | Or Did you think it was possible you could have died from? | | |
| As subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: Then the perion is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have verdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, becomes: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, becomes the but has not yet started to hang; as topped from doing so. It is there been a time when you started to do something to end your life but someone or something stopped you before you can be the steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Stangles are similar to interrupted attempts, except that the individual stops himberself; instead of being stopped by something else. It is also there been a time when you started to do something to try to end your life but you stopped yourself before you actually did your you do not not a time when you started to do something to try to end your life but you stopped yourself before you actually did your you to preparation towards immamently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a certification towards immamently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gran, pring valuables away or writing a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gran, pring valuables away or writing a suicide antempt or preparing to kill yourself (such as collecting pills, getting a gran, pring valuables away or writing a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gran, pring valuables away or writing a suicide attempt on the preparing to kill yourself (such as collecting pills, gettin | impathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | | |
| therrupted Attempt: The person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have coursed). The person has pulls in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, theoring. Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, are if the gun fails to fire, it is an attempt. Jumping Person is a possed to jump, is grabbed and taken down from ledge. Hanging: Person has no around esk but has not yet started to hang - is stopped from doing so. It is there been at time when you started to do something to end your life but someone or something stopped you before you cutually did anything? Yes, describe: The person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior, samples are similar to interrupted attempt, except that the individual stops him/herself, instead of being stopped yourself before you actually did nything? Yes, describe. Teparatory Acts or Behavior: test or preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, pills yes, describe. Teparatory Acts or Behavior: test or preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, pills yes, describe. Teparatory Acts or Behavior: test or preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, pills yes, describe. Test or perparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, pills, yes, describe. Test or perparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a g | yes, describe. | Yes | No |
| Ves Content Ves Conten | as subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| recurred. verdose. Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, thooting. Person has gua pointed toward self, gun is taken away by someone clee, or is somehow prevented from pulling trigger. Once they pull the trigger, are if the gun fails to fire, it is an attempt. Jumping. Person sha store around each but has not yet started to hang - is stopped from doing so. It is there been at time when you started to do something to end your life but someone or something stopped you before you cutually did anything? It is there been a time when you started to do something to end your life but someone or something stopped you before you can be give, describe. Ves. 2 Total # interrupted attempt: The person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. It is there been a time when you started to do something to try to end your life but you stopped yourself before you actually did nything? Tyes, describe: **Reparatory Acts or Behavior:** tel or preparatory Acts or Behavior: tel or preparatory Acts or Behavior: act or preparation towards immineently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a earlied nearly you take any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun), withing valuables away or writing a suicide note)? **Yes 2** **Wes 2** **Wes 3** **Wes 4** **Answer for Actual Attempts Only** **Nextual Lethality/Medical Damage:** **Wes 4** **Moderate physical damage were you minor physical damage (e.g., surface scratches). **Monor physical damage well and attempt not preceded (e.g., consolose without reflexes; third-degree bums; bleeding of major vessel). **Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose without reflexes; third- | | Ves | No |
| Itola # interruptic citically did anything? Total # interruptic citically did anything? Total # interruptic citically did anything? Total # interruptic citically did anything? Total # interruptic citically did anything? Total # interruptic citically did anything a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. A samples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Interruptic citically for the properties of the part of the properties of the part of the properties of the properties of the part of the properties of the properties of the part of the properties of the properties of the part of the properties of the part of the properties of the properties of the part of the properties of the properties of the part of the properties of the part of | curred). rerdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, tooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, en if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around | | |
| District Attempt: Then person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Namples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Total #: aborted inviting? New Actual Lethality: Only Answer if Ac | as there been a time when you started to do something to end your life but someone or something stopped you before you<br>tually did anything? | | |
| then person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. At samples are similar to interrupted attempts, except that the individual stops him/berself, instead of being stopped by something else. It is there been a time when you started to do something to try to end your life but you stopped yourself before you actually did nything? It is on preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a pecific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). It is alway you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, iving valuables away or writing a suicide note)? It is alway you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, iving valuables away or writing a suicide note)? Yes alway you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, iving valuables away or writing a suicide note)? Yes a limited behavior was present during the assessment period? Answer for Actual Attempts Only Actual Lethality/Medical Damage: Answer for Actual Attempts Only Most Leth Attempt Actual Lethality/Medical Damage (e.g., surface scratches). Monor physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree bums; bleeding of major vessel). Moderately severe physical damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree bums over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the follow | yes, describe: | 100 | - 1 |
| Total # Actual Lethality/Medical Damage: Answer for Actual Lethality Medical attempts Only | | Yes | No |
| reparatory Acts or Behavior: cts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a becific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Idave you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, iving valuables away or writing a suicide note)? In the second of | tamples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. as there been a time when you started to do something to try to end your life but you stopped yourself before you actually did | Total | |
| Yes Peparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a pecific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). | yes, describe: | n_ | |
| Districted Second Process Second P | ets or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a ecific method (e.g., biving pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). are you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, wing valuables away or writing a suicide note)? | 1,000 | No |
| Actual Lethality/Medical Damage: Actual Lethality/Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious ethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away sefore run over). | | Yes | No |
| Answer for Actual Attempts Only Most Leth Attempt Date: Actual Lethality/Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderately severe physical damage; medical nospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Doeath Cotential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious ethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away efore run over). | - 1 | _ | |
| Answer for Actual Attempts Only Most Leth Attempt Date: No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Potential Lethality: Only Answer if Actual Lethality=0 inkely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious thality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away efore run over). | aicide: | | No |
| No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Potential Lethality: Only Answer if Actual Lethality=0 likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious thality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away efore run over). | Inswer for Actual Attempts Only | Most L<br>Attemp | ethal |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious ethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). | | Code |
| 1 = Behavior likely to result in injury but not likely to cause death | otential Lethality: Only Answer if Actual Lethality=0 kely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious thality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away fore run over). = Behavior not likely to result in injury | Enter | Code |

#### 10.4 RESTRICTED MEDICATIONS TABLES

Lists of medication can be found in the sections below. The lists are not exhaustive and will not be updated during the course of the trial.

Investigators are advised to verify product labelling information.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.4.1 Strong CYP3A4 inhibitors

#### **Strong CYP3A4 inhibitors:**

- boceprevir
- ceritinib
- clarithromycin
- cobicistat
- conivaptan
- diltiazem
- idelalisib
- indinavir
- itraconazole
- ketoconazole oral administration
- LCL161
- mifepristone
- mibefradil
- nefazodone
- nelfinafir
- posaconazole
- ribociclib
- ritonavir
- saquinavir
- telaprevir
- telithromycin
- troleandomycin
- VIEKIRA PAK2
- voriconazole

#### **Combinations of CYP3A4 inhibitors:**

- danoprevir/ritonavir
- elvitegravir/ritonavir
- indinavir/ritonavir
- lopinavir/ritonavir
- paritaprevir/ritonavir/ombitasvir/dasbuvir
- saquinavir/ritonavir
- tipranavir/ritonavir

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.4.2 Equivalent doses of corticosteroids

Table 10.4.2: 1 Equivalent Doses of Corticosteroids

| Drug | Equivalent dose (mg) | Conversion factor |
|---------------------------|----------------------|-------------------|
| Prednisone | 5 | x 1 |
| Prednisolone | 5 | x 1 |
| Triamcinolone | 4 | x 1.25 |
| 6-Methylprednisolone | 4 | x 1.25 |
| Dexamethasone | 1 | x 5 |
| Betamethasone | 0.75 | x 6.7 |
| 16-Methylprednisolone | 6 | x 0.8 |
| Fluocortalon | 5 | x 1 |
| Cloprednol | 3.75-5 | x 1.0-1.5 |
| Deflazacort | 6 | x 0.8 |
| Cortisol (hydrocortisone) | 20 | x 0.25 |
| Cortisone | 25 | x 0.20 |

#### **10.4.3** Restricted PDE inhibitors

| Compound | Indication |
|---|---|
| Non-selective | |
| Theophylline (Theolair, Slo-Bid, Theo 24) | Asthma and bronchoconstriction |
| Aminophylline (Phyllocontin) | Asthma and bronchoconstriction |
| Oxtriphylline (Choledyl) | Asthma and bronchoconstriction |
| Dyphylline (inhibits PDE3, 4, 7, adenosine 2 receptors) (Dilor, Lufyllin) | Asthma and bronchoconstriction |
| Pentoxifylline (inhibits PDE4, 5, adenosine 2 receptors) (Trental, Pentoxil) | Intermittent claudication |
| Ibudilast (highest affinity for PDE10A, 4, 11, 3) | Asthma and dizziness related to cerebral infarction |
| (Ketas, Pinatos, Eyevinal) | Allergic conjunctivitis |
| Tofisopam (highest affinity for PDE4, 10, 3, 2) (Emandaxin, Grandaxin) | Anxiety |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Compound | Indication |
|---|---|
| Dipyridamole (highest affinity for PDE8, 1, 3, 2, adenosine deaminase and ENT1) (Persantine) | Post-operative thromboembolism |
| PDE3 with potential PDE4-cross reactivity | |
| Milrinone (Primacor, Corotrope) | Congestive heart failure |
| Amrinone (Inamrinone, Inocor) | Congestive heart failure |
| Enoximone (Perfan) | Congestive heart failure |
| Pimobendan (Acardi) | Heart failure |
| PDE4 | |
| Roflumilast (Daliresp, Daxas) | Chronic obstructive pulmonary disease |
| Apremilast (Otezla) | Psoriasis and psoriatic disorders |
| Crisaborole (Eucrisa) | Moderate atopic dermatitis (patients >2 years old) |
| Drotaverine (also inhibits L-type voltage-<br>operated calcium channel) (No-Spa, Doverin) | Functional bowel disorders; pain caused by smooth muscle spasm |

#### 10.5 OPPORTUNISTIC INFECTIONS

These include *Pneumocystis jirovecii*, BK virus disease including polyomavirus-associated nephropathy (PVAN), *Cytomegalovirus* (CMV), post-transplant lymphoproliferative disorder (Epstein–Barr virus [EBV]), progressive multifocal leucoencephalopathy, bartonellosis (disseminated only), blastomycosis, toxoplasmosis, coccidioidomycosis, histoplasmosis, aspergillosis (invasive only), candidiasis (invasive or pharyngeal), cryptococcosis, other invasive fungi (mucormycosis (zygomycosis, rhizopus, mucor, lichtheimia), *Scedosporium/Pseudallescheria boydii*, fusarium), legionellosis, *Listeria monocytogenes* (invasive only), tuberculosis, nocardiosis, non-tuberculous mycobacterium, salmonellosis (invasive only), HBV reactivation, herpes simplex (invasive only), herpes zoster, strongyloides (hyperinfection syndrome and disseminated forms only), paracoccidioides, *Penicillium marneffei*, *Sporothrix schenckii*, cryptosporidium species (chronic only), microsporidiosis, leishmaniasis (visceral only), *Trypanosoma cruzi* infection (Chagas' disease) (disseminated only), campylobacteriosis (invasive only), shigellosis (invasive only), vibriosis (invasive due to vibrio vulnificus), HCV progression [R17-2617].

#### 10.6 ELIGIBILITY CONFIRMATION OF IPF DIAGNOSIS

Eligible are Patients with a clinical diagnosis of IPF based on the 2022 guideline *Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline* as confirmed by the investigator based on chest HRCT scan taken within 12 month of Visit 1 and, if available, surgical lung biopsy or


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

transbronchial lung cryobiopsy (TBLC), as well as a "UIP" or "Probable UIP" HRCT pattern consistent with the clinical diagnosis of IPF, as confirmed by central review prior to Visit 2. If the HRCT finding is "Indeterminate", the clinical diagnosis of IPF may be confirmed locally by (historical) surgical lung biopsy or TBLC demonstrating a "UIP" or "Probable UIP" histopathology pattern. If the HRCT findings are "suggestive of an alternative diagnosis", the clinical diagnosis of IPF may be confirmed locally by (historical) surgical lung biopsy or TBLC demonstrating a "UIP" histopathology pattern.

All chest HRCTs will be sent for central review by an experienced expert based on the recent ATS/ERS/JRS/ALAT guideline on the diagnosis of IPF [P22-03204].

Patients with a centrally reviewed HRCT pattern qualifying as UIP or Probable UIP are eligible for participation and are not required to have a surgical lung biopsy in the appropriate clinical context for the diagnosis of IPF.

Patients clinically suspected to have IPF with an HRCT pattern of "Indeterminate for UIP" require historical (i.e., not taken for the purpose of this trial) surgical lung biopsy or TBLC, which will be reviewed locally (by the investigator/local histopathologist). In these patients, specific combinations of HRCT patterns and histopathology patterns may still allow a diagnosis of IPF based on the 2022 ATS/ERS/JRS/ALAT Guideline, i.e., an HRCT pattern of "indeterminate for UIP" in combination with a surgical lung biopsy or TBLC with a histopathologic pattern of "UIP or probable UIP" could qualify for inclusion.

Patients clinically suspected to have IPF with an HRCT pattern "suggestive of an alternative diagnosis" require historical (i.e., not taken for the purpose of this trial) surgical lung biopsy or TBLC which will be reviewed locally (by the investigator/local histopathologist). In these patients, specific combinations of HRCT patterns and histopathology patterns may still allow a diagnosis of IPF based on the 2022 ATS/ERS/JRS/ALAT Guideline, i.e., an HRCT pattern of "alternative diagnosis" in combination with a surgical lung biopsy or TBLC with a histopathology pattern of "UIP" could qualify for inclusion.

Appropriate documentation at site for these cases is required. Copies of the original, histopathological assessments and resulting diagnosis are required in patient files.

In case the HRCT does not meet eligibility criteria of 1305-0014, patient is allowed to be rescreened in the 1305-0023 trial if an alternative clinical ILD diagnosis is reached and the patient fulfils the respective inclusion & exclusion criteria.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 10.6: 1 Idiopathic Pulmonary Fibrosis diagnosis based upon chest HRCT and biopsy patterns

| IPF | suspected <sup>1</sup> | Histopathology pattern | | | |
|---|---|---|---|---|---|
| | | UIP | Probable UIP | Indeterminate<br>for UIP or<br>biopsy not<br>performed | Alternative diagnosis |
| HRCT | UIP | IPF | IPF | IPF | Non-IPF dx |
| pattern | <b>Probable UIP</b> | IPF | IPF | IPF (Likely) <sup>2</sup> | Non-IPF dx |
| | Indeterminate | IPF | IPF (Likely) <sup>2</sup> | Indeterminate <sup>3</sup> | Non-IPF dx |
| | Alternative diagnosis | IPF(Likely) <sup>2</sup> | Indeterminate <sup>3</sup> | Non-IPF dx | Non-IPF dx |

dx = diagnosis; HRCT = high-resolution computed tomography; IPF = idiopathic pulmonary fibrosis; UIP = usual interstitial pneumonia. (adapted from Figure 9 in [P22-03204])

<sup>2</sup> IPF is the likely diagnosis when any of the following features are present:

- Moderate-to-severe traction bronchiectasis and/or bronchiolectasis (defined as mild traction bronchiectasis and/or bronchiolectasis in four or more lobes including the lingual as a lobe, or moderate to severe traction bronchiectasis in two or more lobes) in a man over age 50 years or in a woman over age 60 years
- Extensive (30%) reticulation on HRCT and an age >70 years
- Increased neutrophils and/or absence of lymphocytosis in BAL fluid
- Multidisciplinary discussion reaches a confident diagnosis of IPF.

• Without an adequate biopsy remains indeterminate

With an adequate biopsy may be reclassified to a more specific diagnosis after multidisciplinary discussion and/or additional consultation.

#### 10.7 TRIAL PARTICIPANT FEEDBACK

Optional Trial Participant Feedback Questionnaires:

This trial will include an option for participants to complete anonymized questionnaires, 'Trial Participant Feedback Questionnaire', to provide feedback on their clinical trial experience. Individual participant level responses will not be reviewed by investigators. Responses will be used by the sponsor to understand where improvements can be made in the clinical trial process. These questionnaires will not collect data about the participant's disease, symptoms, treatment effect, or AEs and therefore will not be part of the trial data or clinical trial report. The questionnaires will be implemented after local regulatory approval and after consent of the trial participant. Providing feedback is optional and not required for participation in the trial.

<sup>&</sup>lt;sup>1</sup> "Clinically suspected of having IPF" = unexplained symptomatic or asymptomatic patterns of bilateral pulmonary fibrosis on a chest radiograph or chest computed tomography, bibasilar inspiratory crackles, and age greater than 60 years. (Middle-aged adults [40 yr and 60 yr], especially patients with risks for familial pulmonary fibrosis, can rarely present with the otherwise same clinical scenario as the typical patient older than 60 years.)

<sup>&</sup>lt;sup>3</sup> Indeterminate for IPF

Boehringer Ingelheim BI Trial No.: 1305-0014

c39145241-04

Clinical Trial Protocol


20 Sep 2023

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Optional Caregiver Feedback Questionnaires:

If applicable, this trial will include an option for caregivers to complete anonymized questionnaires, 'Caregiver Feedback Questionnaire', to provide feedback on the clinical trial experience. Individual caregiver level responses will not be reviewed by investigators. Responses will be used by the sponsor to understand where improvements can be made in the clinical trial process. These questionnaires will not collect data about the participant's disease, symptoms, treatment effect, or AEs and therefore will not be part of the trial data or clinical trial report. The questionnaires will be implemented after local regulatory approval and after consent of the caregiver. Providing feedback is optional and not required for participation in the trial.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. DESCRIPTION OF GLOBAL AMENDMENT(S)

#### 11.1 GLOBAL AMENDMENT 1

| Date of amendment | 26 Jul 2022 | |
|---|---|---|
| EudraCT No. | 2022-001091-34 | |
| BI Trial No. | 1305-0014 | |
| BI Investigational<br>Medicinal Product | BI 1015550 | |
| Title of protocol | A double blind, randomized, placebo-controlled trial evaluating the efficacy and safety of BI 1015550 over at least 52 weeks in patients with Idiopathic Pulmonary Fibrosis (IPF) | |
| Global Amendment due t | o urgent safety reasons | |
| Global Amendment (non- | -substantial changes) | X |
| | - | |
| Section to be changed | Flow chart (number of days for visit assignment | <u>(</u> ) |
| Description of change | The number of days for Visit 4 was changed from 35 to 43. The number of days for Visit 7 was changed from 169 to 183. | |
| Rationale for change | Changed to correct the calculated number of days for visit assignments based on the conversion of trial weeks into days. | |
| Section to be abanged | Flow short (factness ** on ESD collection) | |
| Description of change | Flow chart (footnote ** on ESR collection) Updated wording in footnote: Central laboratory not provide the material for ESR collection to so countries. Instead, material from local site has to perform the test locally. ESR should also be rease of potential vasculitis. | ome<br>to be used |
| Rationale for change | Clarification that material for ESR collection may be provided to some countries by central laboratory. | |
| Section to be changed | Flow chart (footnote 11) | |
| Description of change | Addition of sentence: More frequent pregnancy testing may be done if required. | |
| Rationale for change | Clarification on pregnancy tests. | |

| Section to be changed | Section 1.4.2 Risks |
|---|---|
| Description of change | Addition of <b>Psychiatric disorders</b> to Table 1.4.2: 1 |
| | Overview of trial related risks. |
| Rationale for change | Correction as this row was unintentionally missing in this |
| | table to maintain consistency with information in the IB. |
| Section to be changed | |
| Description of change | |
| Rationale for change | |
| Section to be changed | Section 3.2 Discussion of trial design including the choice |
| | of control group(s) |
| Description of change | Deleted information on continuing, adding, or changing |
| | treatment with immunosuppressive and immunomodulatory |
| | drugs. |
| Rationale for change | Correction as immunosuppressive drugs are not indicated |
| | for treatment of IPF, where no other underlying disease is |
| | present as per definition. |
| Cartan to be about a | Section 3.3.4.1 Discontinuation of trial treatment |
| Section to be changed | |
| Description of change | Deleted last part of the sentence: Ideally, the patient should |
| | attend all remaining visits after treatment discontinuation. For those patients who are unable to complete the scheduled |
| | visits, at least phone contacts should occur at the scheduled |
| | visit sine points and FVC measurement at Week 52 should |
| | be collected. |
| Rationale for change | Clarification as in case of a phone contact, FVC |
| Turionare for enange | measurements cannot be performed. |
| | 1 |
| Section to be changed | Section 5.1.1 FVC |
| Description of change | Deletion of phone call: During the treatment phase, the |
| | iSpiro device and respective phone with the App will be |
| | provided to the patient upon decision of the investigator in |
| | order to perform an assisted (via phone or video call) home |
| | spirometry either at unscheduled visits or as a fallback |
| | solution if the patient is unable to get to the site for the |
| | scheduled visit. |
| Rationale for change | Clarification as the provided device does not offer the |
| | facility to have a phone call without video connection. |

| Г | |
|---|---|
| Section to be changed | Section 5.3.1 Assessment of pharmacokinetics |
| Description of change | Updated wording: PK sampling will be performed at the |
| D ( ) L C 1 | time points indicated in the flow chart. Visits 4, 5, and 7. |
| Rationale for change | Clarification to keep text consistent with the flow chart |
| Section to be changed | Section 6.2.2.2 Conduct of a fallback visit (remote/home visit) |
| Description of change | Added sentence: Trial medication may be shipped from |
| | the site directly to the patient (if acceptable according to |
| | local laws and regulations). |
| Rationale for change | Clarification on the fallback visit |
| Kationale for change | Clarification on the famour visit |
| | 0 1 (000 0 1 1 0 0 111 1 1 1 1 1 1 1 |
| Section to be changed | Section 6.2.2.2 Conduct of a fallback visit (remote/home |
| | visit) |
| Description of change | Added bullet point to assessments that can be done |
| | remotely: |
| | • Urine dipstick pregnancy test performed by the |
| | patient at home |
| Rationale for change | The possibility of urine pregnancy testing done during |
| Trationale for change | remote visits was missing. |
| | Temote visits was missing. |
| | S-4: (222 S-1-4-f-f-f-1111:-://4/l |
| Section to be changed | Section 6.2.2.2 Conduct of a fallback visit (remote/home |
| | visit) |
| Description of change | Updated wording: If blood and urine sampling for central |
| | lab at the patient's home is not possible, safety lab analyses |
| | including the routine safety lab tasks as per Table 5.2.3.1: 1 |
| | should be performed at a local lab. |
| Rationale for change | Clarification on safety lab analyses during home visits. |
| 9 | , , , |
| Section to be changed | Section 7.5 Determination of sample size |
| Description of change | Deletion of asterisks for 2 footnotes in Table 7.5: 2: |
| Description of change | *—Probability calculated based on 50,000 simulation |
| | iterations. Total alpha-level = 0.05 (two-sided), 1:1:1 |
| | randomization ratio with 336 patients per arm |
| | ** multiplicity adjusted for interim analysis using group |
| | sequential design with Wang-Tsiatis alpha spending |
| | function (delta = 0.25) |
| Rationale for change | Clarification as these notes refer to the whole table. |
| Section to be changed | Section 10.6 Eligibility confirmation of IPF diagnosis |
| Description of change | Reference related to HRCT scans changed |
| Rationale for change | Corrected to reference number of updated |
| | ATS/ERS/JRS/ALAT guideline |
| <u> </u> | TITO DICO VICO I IDEI I SUIGOIIIIC |
| Section to be shared | Throughout the CTD |
| Section to be changed | Throughout the CTP |
| Description of change | Typographical errors and minor formatting issues amended |
| Rationale for change | To increase readability |


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.2 GLOBAL AMENDMENT 2

| Date of amendment | 10 May 2023 | |
|---|---|---|
| EudraCT No. | 2022-001091-34 | |
| BI Trial No. | 1305-0014 | |
| BI Investigational | BI 1015550 | |
| Medicinal Product | | |
| Title of protocol | A double blind, randomized, placebo-controlled | trial |
| | evaluating the efficacy and safety of BI 1015550 | |
| | least 52 weeks in patients with Idiopathic Pulmo | onary |
| | Fibrosis (IPF) | |
| Clabal Assaulance described | | |
| Global Amendment due to | | |
| Global Amendment (subs | tantial changes) | X |
| Section to be changed | Flow Chart (screening period) | |
| Description of change | The minimum period for screening was reduced | to 1 week |
| Rationale for change | Provide more flexibility for randomizations | |
| Section to be changed | Flow Chart (lab tests) | |
| <b>Description of change</b> | The erythrocyte sedimentation rate (ESR) test w | |
| Rationale for change | Local workup is crucial for the reliability of the | |
| | sites are not familiar with the sample handling a | |
| | procedures. Therefore test results are often incompared to the second of | nclusive. |
| Section to be changed | Flow Chart (temporary discontinuation of trial t | reatment) |
| Description of change | Footnote #2 was modified as follows: | |
| Description of change | In case of premature discontinuation of trial | medication. |
| | the End of Treatment (EOT) visit should only b | |
| | cases of premature trial medication if the discor | |
| | permanent, and with a Follow-up (FU) visit is | |
| | performed 7 days (+3 days) after end of treatme | |
| | patient discontinued the trial medication mor | |
| | week prior to the EOT visit, this FU visit is n | - |
| | A scheduled visit may be missed if EOT or FUe | - |
| | visit occurs within 4 weeks prior to scheduled v | |
| | the premature EOT, every effort should be made data until the end of the trial. | e to collect |
| Dationals for shares | | · NG |
| Rationale for change | Clarification of procedures in case of temporary permanent discontinuation of trial treatment. | vs. |
| | permanent discontinuation of trial treatment. | |
| Section to be changed | Flow Chart (patient-reported outcomes) | |
| Section to be changed | 1 10 w Chart (patient-reported outcomes) | |


| Description of change | Addition to Footnote #3: |
|---|---|
| | At the latest, the patients' questionnaires must be |
| | completed prior to the pulmonary function tests. |
| Rationale for change | Clarification of the timing of the patients' questionnaires |
| | (consistent with the change in Section 6.2) |
| Section to be changed | Flow Chart (pregnancy tests) |
| Description of change | Footnote #11 was modified as follows: |
| | Women of childbearing potential only. Serum pregnancy |
| | test to be performed at V1; urine dipstick pregnancy test |
| | to be performed at V2 and following visits (if positive, |
| | urine dipstick test to be followed by serum test for |
| | <b>confirmation).</b> More frequent pregnancy testing may be |
| | done if required. |
| Rationale for change | The type and timing of the pregnancy tests were clarified. |
| Section to be changed | Flow Chart (design of the extension trial) |
| Description of change | Footnote #17 was updated to remove the design of the |
| | extension trial ("open-label") and clarify when a follow-up |
| | visit is needed. |
| Rationale for change | The extension trial design is not finalized and might also |
| | contain a double-blind start until the decision about the final |
| | intended marketed dose. |
| | The follow-up visit can be skipped if the following regular |
| | visit after the end of treatment is planned at 7-21 days after |
| | the last dose was administered. |
| | C (' 12D C1 |
| Section to be changed | Section 1.2 Drug profile |
| Description of change | Sentence added to the drug-drug interaction subsection: |
| | In a clinical drug-drug interaction study with |
| | midazolam (sensitive CYP3A4 substrate), BI 1015550 |
| | was not shown to have a clinically relevant CYP3A induction. |
| | muucuon. |
| | Subsection on the data from non-clinical toxicology studies |
| | updated to reflect the fact that the toxicology summary |
| | remained applicable when considering the data from the |
| | 39-week study in monkeys and sentence added: |
| | A sporadic menstrual cycle prolongation was observed |
| | in the 39-week study in female monkeys receiving |
| | ≥10 mg/kg/day, i.e., at approximately 4-fold human |
| | exposure at 18 mg bid. |
| Rationale for change | Addition of data from a recent drug-drug interaction study |
| | with midazolam |
| <u>, </u> | <u> </u> |

c39145241-04

| | Addition of data from a recent 39-week oral (gavage) |
|---|---|
| | toxicity and toxicokinetic study in Cynomolgus monkeys |
| | with a 8-week recovery period |
| Section to be changed | Section 1.4.2 Risks (Table 1.4.2: 1, PK interaction with |
| Section to be changed | strong CYP34A inhibitors) |
| Description of change | Mitigation strategy updated as follows: |
| | This is also applicable for Paxlovid in the treatment of |
| | Covid-19: iIf short-term treatment with Paxlovid potent |
| | <b>CYP3A4 inhibitor</b> is needed, trial medication needs to be |
| D 4' 1 C 1 | paused |
| Rationale for change | Application of the mitigation strategy to all potent CYP3A4 inhibitors, not just Paxlovid. |
| Seation to be abouted | Castian 1 4 2 Diales (Table 1 4 2, 1 Massaylitis) |
| Section to be changed Description of change | Section 1.4.2 Risks (Table 1.4.2: 1, Vasculitis) Summary of data updated to reflect the fact that vasculitis |
| Description of change | was not observed following oral administration of |
| | BI 1015550 in 13- or 39-week studies in monkeys |
| Rationale for change | Addition of data from a recent 39-week oral (gavage) |
| | toxicity and toxicokinetic study in Cynomolgus monkeys |
| | with a 8-week recovery period |
| Section to be abouged | Section 1.4.2 Risks (Table 1.4.2: 1, Severe infections) |
| Section to be changed Description of change | Patients with <b>active</b> tuberculosis are excluded from the trial. |
| Description of change | rations with active tuberculosis are excluded from the trial. |
| Rationale for change | Mitigation strategy updated to reflect the change in EC23 |
| | (Section 3.3.3) |
| | G ( 142 B) 1 ( T 11 142 1 B 1 1 ( 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| Section to be changed | Section 1.4.2 Risks (Table 1.4.2: 1, Reproductive toxicity) |
| Description of change | Summary of data updated as follows: |
| | • In monkeys, a sporadic prolongation in menstrual cycles was observed at approximately ≥4-fold human |
| | exposure at 18 mg BI 1015550 bid. |
| | • Efficacy of oral hormonal contraceptives can be |
| | impacted by potential BI 1015550 related CYP3A |
| | induction |
| | Mitigation strategy on reproductive toxicity updated as follows: |
| | <ul> <li>Women of childbearing potential (WOCBP) need to use</li> </ul> |
| | a highly effective method of contraception. Of note, oral |
| | hormonal contraceptives are not considered a highly |
| | effective method due to potential drug interactions. |
| | WOCBP taking oral contraceptives (OCs) also have |
| | to ensure the use of one barrier method during sexual |
| | intercourse with their partner, e.g., condom to |


| Rationale for change | <ul> <li>account for the risk of potentially reduced efficacy of the OCs in the event of severe vomiting and diarrhea</li> <li>In case of vomiting or diarrhea, instructions in the label of the OC should be followed</li> <li>In case of prolonged (&gt;48h) or repeated vomiting/diarrhea, the use of an alternative highly effective contraceptive measure should be considered</li> <li>The potentially reduced efficacy of OCs from potential CYP3A induction by BI 1015550 was ruled out by a drugdrug interaction trial on the PK of midazolam, a recommended substrate of CYP3A4.</li> <li>Based on these results, OCs are now allowed as highly effective measure of contraception in WOCBP, associated with one barrier method to prevent the risk of potentially reduced efficacy of the OCs in case of severe vomiting and</li> </ul> |
|---|---|
| | diarrhea. |
| Section to be changed | Section 3.2 Discussion of trial design (participants and caregivers questionnaires) |
| Description of change | The following paragraph was added: This trial will include an option for participants and participant caregivers to complete anonymized questionnaires to provide feedback on their clinical trial experience. Providing this feedback is not required for trial participation, and information collected from these questionnaires will not be analyzed as part of the clinical data for the trial (see Section 10.7). |
| Rationale for change | To identify where improvements can be made in the clinical trial process, the sponsor wants to collect the participants' and caregivers' feedback on their clinical trial experience. |
| Section to be changed | Section 3.3.1 Main diagnosis for trial entry |
| Description of change | Eligibilty criteria for patients with an "alternative diagnosis" HRCT finding added: Patients with an "Alternative diagnosis" HRCT finding are eligible if a clinical diagnosis of IPF can be confirmed locally based on (historical) surgical lung biopsy or cryobiopsy demonstrating a "UIP" histopathology pattern Cross references to Table 10.6: 1 were also added in this section. |
| Rationale for change | Patients with an "alternative diagnosis" HRCT finding are considered for eligibility (also see Section 10.6). |
| Section to be changed Description of change | Section 3.3.2 Inclusion criteria (IC6, also in synopsis) Inclusion criterion 6 was updated as follows: |


| | DLCO corrected for Hemoglobin (Hb) [Visit 1] >25% and |
|---|---|
| | <90% of predicted of normal corrected for hemoglobin |
| | (Hb) at Visit 1. |
| Rationale for change | The upper limit for DLCO was deleted since it is not |
| | relevant as an exclusion criterion. Exclusion criteria |
| | regarding lung function are sufficiently covered by the |
| | criteria based on FVC (EC5). |
| | The wording regarding the correction for Hb of predicted |
| | value of DLCO was clarified. |
| Section to be changed | Section 3.3.2 Inclusion criteria (IC7) |
| Description of change | Inclusion criterion 7 was updated as follows: |
| Description of enunge | Women of childbearing potential (WOCBP) must be ready |
| | and able to use highly effective methods of birth control. Of |
| | note, oral hormonal contraceptives are not considered a |
| | highly effective method due to potential drug-drug |
| | interactions WOCBP taking oral contraceptives (OCs) |
| | also have to use one barrier method; please refer to |
| | Section 4.2.2.3. |
| Rationale for change | Based on the results of a drug-drug interaction trial on the |
| Tuestoniase for ename | PK of midazolam, OCs are now allowed as highly effective |
| | measure of contraception in WOCBP, associated with one |
| | barrier method to prevent the risk of potentially reduced |
| | efficacy of the OCs in case of severe vomiting and diarrhea |
| | (also see change to Section 1.4.2). |
| | (undo dee change to decide 11112). |
| Section to be changed | Section 3.3.3 Exclusion criteria (EC1, also in synopsis) |
| Description of change | Exclusion criterion 1 was updated as follows: |
| | Relevant airways obstruction (pPrebronchodilator |
| | FEV1/FVC <0.7) at Visit 1 |
| Rationale for change | Any FEV/FVC ratio <0.7 should be avoided as the risk of |
| | emphysema and obstruction is high and would influence |
| | efficacy endpoint measurements. This criterion was |
| | therefore simplified. |
| Section to be changed | Section 3.3.3 Exclusion criteria (EC10) |
| Description of change | Exclusion criterion 10 was updated as follows: |
| | Patients with underlying chronic liver disease cirrhosis |
| | (Child Pugh A, B, or C hepatic impairment). |
| Rationale for change | Clarification following a question from a site (as Child Pugh |
| | only refers to liver cirrhosis, not chronic liver disease). |
| Section to be abouted | Section 2.2.2 Evaluation emitaria (EC22) |
| Section to be changed | Section 3.3.3 Exclusion criteria (EC23) |
| Description of change | Exclusion criterion 23 was updated as follows: |
| | Patients with positive active tuberculosis (TB) test at Visit |
| | 1 unless they have completed treatment for active or latent |
| | tuberculosis in line with local guidelines. |


| Rationale for change | No negative effect of BI 1015550 on latent tuberculosis is |
|---|---|
| Tationale for change | expected based on new preclinical data (immunophenotype |
| | in a 39-week monkey study). The TB diagnosis was |
| | simplified, relying on the site's expertise. |
| | simplified, relying on the site's expertise. |
| | G (: 222 F 1 : '/ (FC27 |
| Section to be changed | Section 3.3.3 Exclusion criteria (EC27 - new) |
| Description of change | Exclusion criterion 27 was added: |
| | History of stem cell therapy for the treatment of |
| | pulmonary fibrosis. |
| Rationale for change | The effect on the lung of such treatment in the longer term |
| | is currently unknown. |
| Section to be changed | Section 3.3.4.1 Discontinuation of trial treatment |
| Description of change | The following paragraph was updated as follows: |
| | All patients who prematurely discontinue trial medication |
| | will need to complete an End of Treatment (EOT) visit at |
| | the time of discontinuation, and The End of Treatment |
| | (EOT) visit activities will be performed when a patient |
| | discontinues trial medication permanently. |
| | aA premature Follow-up (FU) visit is to be performed |
| | 7 days (+3 days) 1 week later after end of treatment. If |
| | the patient discontinued the trial medication more than |
| | a week prior to the EOT visit, this FU visit is not |
| | required. Patients who prematurely discontinue trial |
| | medication will be asked to remain in the trial and to return |
| | to all regularly scheduled visits until the end of the trial. |
| | Ideally, the patients who permanently discontinue trial |
| | <b>medication</b> should attend all remaining visits after treatment discontinuation. |
| D-4: | |
| Rationale for change | The procedures in case of temporary vs. permanent |
| | discontinuation of trial treatment were clarified. |
| Section to be changed | Section 4.1.4 Drug assignment and administration |
| | (supervision and timing) |
| Description of change | The need for supervision during administration was |
| | clarified: |
| | The patient will receive either active treatment at a dose of 9 |
| | mg, 18 mg, or placebo. The first dose of BI 1015550 or |
| | placebo will be administered to the patient at the end of |
| | Visit 2 (Day 1) under direct supervision of the |
| | investigator or designee. On the day of any further clinic |
| | visits, supervision of administration is not required but |
| | the treatment will <b>preferably</b> be administered to the patient |
| | during the visit. |
| | The timing of administration was clarified to say that the |
| | trial medication should be taken at the same time every day |

| | (±30 mins), ideally between 6:00 and 11:00 in the morning and between 18:00 and 23:00 in the evening, and that if taken around the same time (approximately within an hour), pPatients on nintedanib background should take trial medication first, followed by the antifibrotic background medication after some minutes. |
|---|---|
| Rationale for change | Supervision remains mandatory during the first administration but is not mandatory for any of the following administrations including further clinic visits. Simplified for facilitation of scheduling the visits. |
| | The timing of administration was clarified due to questions on the timeframe, e.g. when a baseline patient visit ends at 12:00. |
| | The order of administration would only have an influence in case intake of antifibrotic and BI 1015550 is close to each other timewise (potential effect of side effects like vomiting). |
| Section to be changed | Section 4.1.5.1 Blinding and procedures for unblinding |
| Description of change | The following sentence was added: If the 9 mg dose is considered futile based on the respective interim analysis (see Section 7.2.8), the patients will be re-assigned to the 18 mg dose in a blinded manner and the 18 mg dose will be given at the next scheduled visit. |
| Rationale for change | The management and handling of patients and data in case the dose of 9 mg bid is considered as futile were clarified. |
| Section to be changed | Section 4.2.2.1 Restrictions regarding concomitant treatment (Table 4.2.2.1: 1, about prednisone) |
| Description of change | The restrictions regarding prednisone prior to the study were updated from not permitted to permitted. As indicated in the footnote of the table, this is referring to 'historical episodes of intake' (i.e. treatment should not be ongoing at Visit 1). It was clarified in the text that prednisone >15 mg/day or equivalent should not be started for respiratory indications during the screening or treatment period. However, prednisone >15 mg/day or equivalent can be prescribed during the treatment period in case of |
| Rationale for change | (suspected) acute IPF exacerbation. Clarification of restrictions regarding historical episodes of |
| 8 | intake, and introduction in case of exacerbations |
| Section to be changed | Section 4.2.2.1 Restrictions regarding concomitant treatment (CYP3A4 inhibitors) |

| Description of change | Restrictions regarding potent CYP3A4 inhibitors were |
|---|---|
| Description of change | updated to clarify that, if any short-term treatment with |
| | potent CYP3A4 inhibitor is needed, IMP should be |
| | 1 |
| | temporarily discontinued and a cross-reference to |
| | Section 3.3.4.1 was added about the conditions to |
| | re-introduce the IMP. |
| | A footnote was also added to Table 4.2.2.1. |
| Rationale for change | The sentence was added to be consistent with Table 1.4.2: 1 |
| | (about trial-related risks) and with Section 3.3.4.1 (about |
| | temporary discontinuation of trial treatment). |
| Section to be changed | Section 4.2.2.1 Restrictions regarding concomitant |
| | treatment (including Table 4.2.2.1: 1, about stem cell |
| | therapy) |
| Description of change | The following restriction was added: |
| | Stem cell therapy for the treatment of pulmonary |
| | fibrosis is not allowed. |
| Rationale for change | The effect on the lung of such treatment in the longer term |
| | is currently unknown (also see addition of EC 27). |
| · | |
| Section to be changed | Section 4.2.2.2 Restrictions on diet and lifestyle |
| Description of change | The restriction regarding the consumption of |
| | methylxanthine-containing drinks or food was lifted: |
| | Patients should refrain from consuming Methylxanthine- |
| | containing drinks or foods (such as coffee, tea, cola, energy |
| | drinks, and chocolate) in the 24 h preceding each on site |
| | visit. Patients should also refrain <b>from</b> drinking grapefruit |
| | juice during the duration of the trial. |
| Rationale for change | Caffeine, theobromine, and theophylline are the most well- |
| | known compounds of the family of methylxanthines. They |
| | are predominantly metabolized by CYP1A2. Since |
| | BI 1015550 is not a CYP1A2 substrate and also does not |
| | modulate CYP1A2, an interaction between BI 1015550 and |
| | methylxanthine-containing drinks or food is not expected. |
| | mean, maintaine commining armine or rood is not expected. |
| Section to be changed | Section 4.2.2.3 Contraception requirements |
| Section to be changed | Section 1.2.2.3 Contraception requirements |


| D : 4: 6.1 | T1 C 11 ' 4 1 1 4 1 |
|---|---|
| <b>Description of change</b> | The following sentence was deleted: |
| | Of note, oral hormonal contraceptives are not considered |
| | highly effective due to a potential CYP3A4 drug interaction |
| | of BI 1015550 in the gastrointestinal tract. Non-oral |
| | hormonal contraception is permissible as described below. |
| | And the following was added to the list of acceptable highly |
| | effective methods of contraception: |
| | • Oral hormonal contraceptives together with one |
| | 2 9 |
| | barrier method (e.g. condom) to account for the risk of |
| | potentially reduced efficacy of the OCs in the event of |
| | severe vomiting and diarrhea. In case of vomiting or |
| | diarrhea, instructions in the label of the OC should be |
| | followed in addition. In case of prolonged (>48h) or |
| | repeated vomiting/diarrhea, the use of an alternative |
| | highly effective contraceptive measure should be |
| | considered |
| Rationale for change | Based on the results of a drug-drug interaction trial on the |
| g- | PK of midazolam, OCs are now allowed as highly effective |
| | measure of contraception in WOCBP, associated with one |
| | barrier method to prevent the risk of potentially reduced |
| | 1 1 |
| | efficacy of the OCs in case of severe vomiting and diarrhea |
| | (also see change to Section 1.4.2). |
| Section to be changed | Section 5.1.1 FVC |
| Description of change | Addition of the following sentence: |
| | In case unacceptable results for FVC/FEV1 at V1 or |
| | FVC at V10 are obtained after the review, the patient |
| | must be reassessed. |
| Rationale for change | These instructions are in the spirometry guidance document |
| g- | but it was considered important to emphasize to the sites. |
| | out it was constanted important to emphasize to the steel. |
| Section to be changed | Section 5.1.5.3 Patient's Global Impression of Severity |
| Section to be changed | (PGIS) of Cough, Shortness of Breath, and Fatigue (also |
| D 1 11 4 1 | Section 5.1.5) |
| <b>Description of change</b> | The description of the questionnaire assessing the severity |
| | of the patient's fatigue was added (the actual questionnaire |
| | was added in Appendix 10.2.4). |
| Rationale for change | The assessment of fatigue severity will be implemented in |
| | all countries where the setup is completed and translated |
| | questionnaire available. |
| 1 | • |
| Section to be changed | Section 5.1.6 DLCO |
| Description of change | The section was updated to clarify that the correction for Hb |
| Description of change | |
| | was applied to <b>predicted</b> DLCO values. It was also clarified |
| | that the site has to enter the unadjusted <b>predicted</b> DLCO |
| | result without Hb correction in the eCRF. |


| | The first formula (one for each gender) was for predicted |
|---|---|
| | DLCO corrected for Hb (and not percent predicted DLCO |
| | corrected for Hb) and the unit of Hb was clarified (g·dL-1) |
| | A second formula was added for percent predicted DLCO |
| | corrected for Hb: |
| | Percent predicted DLCO corrected for Hb = (Mean |
| | value of two DLCO measurements, expressed in |
| | mmol/min/kPa) / Predicted DLCO corrected for Hb) * |
| | 100 |
| | DLCO should always must be performed after spirometry |
| | on the same day. |
| Rationale for change | Clarification of the correction of predicted DLCO for Hb |
| | and revision/addition of formulas to calculate 1) predicted |
| | DLCO corrected for Hb, and 2) percent predicted DLCO |
| | corrected for Hb. |
| | Clarification of the timing of DLCO relative to spirometry. |
| Section to be changed | Section 5.2.3 Safety laboratory parameters |
| Description of change | The ESR test was removed from the routine safety lab test |
| | panel (Section 5.2.3.1) and the test for cryoglobulins was |
| | removed from the vasculitis lab test panel (Section 5.2.3.3). |
| | Note: the mention of ESR test in Section 5.2.6.1.4 (Adverse |
| | Events of Special Interest) was also removed. |
| Rationale for change | Local workup is crucial for the reliability of the results, but |
| | sites are not familiar with the sample handling and |
| | procedures. Therefore test results are often inconclusive. |
| Section to be changed | Section 5.2.3.1 Routine safety lab tests (Table 5.2.3.1: 1) |
| <b>Description of change</b> | The type and timing of the pregnancy tests were clarified. |
| | At screening (V1), a serum pregnancy test is to be |
| | performed (no IMP taken at that time) whereas at V2 (and |
| | following visits), urine dipstick pregnancy test is to be |
| | performed (if positive, urine dipstick test should be |
| | followed by serum test for confirmation). |
| Rationale for change | The use of "Day -1" in the table was confusing; visit |
| | numbers were used instead. |
| - | |
| Section to be changed | Section 5.2.3.2 Infection serology |
| Description of change | Wording was updated as follows: |
| | In case of positive <b>TB test</b> Screening Test, further |
| | diagnostic work up to confirm/exclude the diagnosis of |
| | latent or active is needed (documentation on respective |
| | eCRF page). |
| Rationale for change | Clarification that further diagnostic work up to |
| | confirm/exclude the diagnosis of latent or active TB is to be |
| | done for any positive TB test (not just at screening) |
| | many position is the very more are belowing) |


| Section to be changed | Section 5.2.3.3 Immunological vasculitis markers |
|---|---|
| <b>Description of change</b> | Addition of the following paragraph: |
| | Due to stability matter during storage, ANCA markers |
| | (MPO-ANCA and PR3-ANCA) from Visit 2 and Visit 10 |
| | are analyzed upon receipt, but investigators will not |
| | receive these results as it could influence their |
| | judgement regarding a suspected vasculitis. The rest of |
| | the analysis of immunological vasculitis markers is |
| | performed if an unscheduled "Vasculitis event" is |
| | collected. In this situation, the site will receive the result |
| | for all vasculitis markers previously performed (from |
| | V2 and V10 if already done) and from the unscheduled |
| | "Vasculitis event" kit. These results are shared by the |
| | trial team to the site via the CRA. |
| Rationale for change | The timing and conditions of analysis of ANCA markers |
| | and communication of results to the site were clarified due |
| | to stability matter during storage. |
| | , |
| Section to be changed | Section 5.2.6.3 Independent safety monitoring and adverse |
| | events with additional information collection |
| Description of change | Wording was updated as follows: |
| | Additional details (on top of standard AE and SAE |
| | reporting) will be collected in the eCRF for the adverse |
| | event 'Diarrhea/gastrointestinal events', the adverse events |
| | in the Standard MedDRA Query (SMQ) 'vasculitis' and in |
| | case of positive TB tests tuberculosis screening (see |
| | Section 5.2.3.2). |
| Rationale for change | Clarifications that additional details should be collected in |
| | the eCRF for any positive TB test (not just at screening). |
| | g d f (1 of LID on ) |
| Section to be changed | Section 5.6.1 Chest HRCT assessment (repetition of HRCT) |
| <b>Description of change</b> | The following sentence was deleted: |
| | HRCT should not be repeated for eligibility if previous scan |
| | was taken within the past 3 months. |
| Rationale for change | The possibility to repeat the HRCT for eligibility and the |
| | allowed timeframe between scans will be left up to the |
| | investigator's decision, based on local guidance. |
| Section to be abanged | Section 6.1 Visit Schedule |
| Section to be changed Description of change | The following sentence was amended: |
| <b>Description of change</b> | The following sentence was amended. The patient will be randomized at Visit 2 if all inclusion |
| | • |
| | criteria (including positive HRCT review and acceptable |
| | spirometry measurements) and none of the exclusion |
| | criteria (lab exclusion criteria referring to Visit 1 results) are |
| | fulfilled. |


| Rationale for change | The conditions for randomization were clarified (also see |
|---|---|
| rationale for enange | the change in Section 5.1.1) |
| <u>l</u> | the change in Section 3.1.1) |
| Section to be changed | Section 6.2 Details of trial procedures at selected visits |
| Description of change | The following edits were made: |
| Description of change | |
| | Regarding patients' questionnaire: At the latest, the |
| | patients' questionnaires must be completed prior to the |
| | pulmonary function tests |
| | Regarding the pulmonary function tests: FVC (spirometry) |
| | should must be performed before DLCO |
| | Regarding IRT call and IMP dosing/dispensing: IRT call |
| | and IMP dosing/dispensing should always be done as the |
| | last procedure after all visit assessments, except at Visit 1 |
| | where the IRT call may be done earlier during the |
| | patient's visit. |
| Rationale for change | The order of procedures was clarified. |
| Section to be changed | Section 6.2.1 Screening period |
| Description of change | Sentence amended: |
| r r | If a patient is re-screened and there are valid screening |
| | determinations from patient's previous participation in the |
| | trial, like for example safety labs, performed within 28 days |
| | 8 weeks prior to randomization (Visit 2), these do not need |
| | to be repeated. |
| Rationale for change | This is to align the timeframe with the regular allowed |
| Rationale for change | screening phase of 8 weeks without repetition of V1 |
| | laboratory tests. |
| Casting to be about 1 | Section 6221 Conduct of a nearly site visit |
| Section to be changed | Section 6.2.2.1 Conduct of a regular site visit |
| <b>Description of change</b> | The need for supervision during administration was |
| | clarified: |
| | Each patient will receive the first dose of BI 1015550 or |
| | placebo at the end of Visit 2 (Day 1) under direct |
| | supervision of the investigator or designee. Patients will |
| | take trial medication twice daily (bid) orally from that |
| | timepoint onwards. On the day of any further At clinic |
| | visits, supervision of administration is not required but |
| | trial medication will <b>preferably</b> be administered to the |
| | patient during the visit (as the last procedure, see |
| | Section 6.2) taken under direct supervision of the |
| | investigator or designee. |
| Rationale for change | Supervision remains mandatory during the first |
| 9 | administration but is not mandatory for any of the following |
| | administrations including further clinic visits. Simplified for |
| | facilitation of scheduling the visits. |
| Section to be changed | Section 6.2.3 Follow-up period and trial completion |
| Section to be changed | Section 0.2.3 Pollow-up period and that completion |

| Description of change | Specification about the design of the extension trial ("open- |
|---|---|
| | label") was removed (also applied in Section 3.1). |
| | The procedures in case of temporary vs. permanent |
| | discontinuation of trial treatment were aligned with the |
| | changes made in Section 3.3.4.1. |
| | It was clarified that the abnormal values to monitor are |
| | those collected at the last study visit (EOS). |
| Rationale for change | The extension trial design is not finalized and might also |
| 1g | contain a double-blind start until the decision about the dose |
| | that could be given as an open-label treatment is taken. |
| | Alignment of procedures in case of temporary vs. |
| | permanent discontinuation of trial treatment with |
| | Section 3.3.4.1. |
| | occuon 3.3.7.1. |
| Section to be changed | Section 7.2.1 General considerations (and Sections 7.2.3 |
| Section to be changed | · · |
| Description of shapes | and 7.2.4) Addition of the Full Analysis Set (EAS) as the primary |
| Description of change | Addition of the Full Analysis Set (FAS) as the primary |
| | population for the efficacy analysis, and modification of the |
| | definition of the Treated Set (TS), which will be the primary |
| | population for the safety analysis (but not the efficacy |
| | analysis). |
| | Inclusion of the analysis strategy in the definition of the |
| | analysis sets. |
| | Deletion of the following sentence: For efficacy and safety |
| | analyses, patients will be analysed according to their |
| | planned treatment group. |
| | Deletion of the Per Protocol Set (PPS). |
| | Sections 7.2.3 and 7.2.4 were updated to reflect the fact that |
| | the FAS will be the efficacy set. |
| Rationale for change | Efficacy and safety analyses will be conducted with |
| | different analysis strategy. Patients will be analyzed as |
| | randomized in the efficacy analysis, whereas they will be |
| | analyzed as treated in the safety analysis. |
| | The PPS was deleted as post-randomization events will be |
| | handled via estimands (based on ICH E9 addendum), as |
| | described in the TSAP. |
| | desertion in the 15/11. |
| Section to be changed | Section 7.2.1 General considerations (important protocol |
| Section to be changed | deviations) |
| Description of shapes | , |
| Description of change | The sentence was updated as follows: |


| | Specifications for Definitions and handlings of important protocol deviations (IPDs) leading to exclusion from PPS will be provided in the trial Integrated Quality and Risk Management Plan (IQRMP) included in the DV domain specifications and will be stored within the trial master file (TMF) in the electronic document management system (EDMS). All potential important protocol deviations will be discussed during trial oversight meetings and report planning meetings. and aAll final decisions concerning IPDs will be made before un-blinding. |
|---|---|
| Rationale for change | Clarification on handling, documentation and review of IPDs. |
| Section to be changed | Section 7.2.3.1 Sensitivity analyses Section 7.2.4.1 Analysis of key secondary endpoint |
| Description of change | Sentence amended: On-treatment-analyses, while-compliant-to-protocol analyses in the PerProtocol Set and models with modified sets of covariates will be conducted as further sensitivity analyses |
| Rationale for change | Deletion of the PPS. |
| Section to be changed | Section 7.2.4.1 Analysis of key secondary endpoint Section 7.2.4.2 Analysis of other secondary endpoints |
| Description of change | For all time-to-event endpoints, the start date considered when calculating the time to event of interest (and the time to censoring) was changed from 'randomization date' to 'first drug intake date'. |
| Rationale for change | There may be a few days gap between the randomization date and the first drug intake date. For the purpose of time-to-event analyses, the actual time at risk starts with the first drug intake. |
| Section to be abanged | Section 7.2.9 Interior analyses (and symposis) |
| Description of change | Section 7.2.8 Interim analyses (and synopsis) The following sentences were added: If the 9 mg dose is considered futile, the patients on that treatment arm will be re-assigned to the 18 mg dose in a blinded manner (see Section 4.1.5.1) at their next scheduled visit. A shorter version of this new paragraph was added to the synopsis. |
| Rationale for change | The management and handling of patients and data in case the dose of 9 mg bid is considered as futile were clarified. |
| Section to be changed | Section 7.2.8 Interim analyses (and synopsis) |
| Description of change | The description of the interim analysis to detect early signs of substantial efficacy was adjusted: |

c39145241-04 Clinical Trial Protocol 

| | | | | | | | | - |
|---|---|---|---|---|---|---|---|---|
| Proprieta | ry confidentia | al information © 20 | 23 Boehringe | er Ingelheim | International | GmbH or one or more of | of its affiliated comp | anies |

| | [] an interim analysis for efficacy will may be performed |
|---|---|
| | by the DMC. |
| | This interim analysis is planned to may be conducted when |
| | a minimum of 450 patients (150 patients per arm) have |
| | reached the Week 52 FVC assessment approximately |
| | 52 weeks after 450 patients (150 patients per arm) have |
| | started treatment and 26 weeks after the last patient has |
| | started treatment. |
| Rationale for change | The previous wording excluded patients who died or who |
| | were lost to follow-up from the count of 450 because these |
| | patients would not reach the Week 52 FVC assessment. The |
| | new wording does include the patients who died or who |
| | were lost to follow-up in the count of 450. |
| | The exact timing of this analysis remains to be confirmed. |
| | The exact uning of this analysis remains to be confillined. |
| Section to be abouted | Section 7.4 Dandomization (fatility analysis) |
| Section to be changed | Section 7.4 Randomization (futility analysis) |
| Description of change | The following sentence was added: |
| | For patients to be enrolled and randomized after a |
| | potential futility stop of the low dose level (9 mg; see |
| | Section 7.2.8), the randomization ratio will be 1:1 |
| | (BI 1015550 18 mg bid vs. Placebo). |
| Rationale for change | The randomization ratio in case the dose of 9 mg bid is |
| | considered as futile were clarified. |
| Section to be changed | Section 7.5 Determination of sample size |
| Description of change | Sentence deleted: This leads to the same overall treatment |
| | effect of 74 mL overall. |
| Rationale for change | The treatment effect is already stated further below in that |
| | section. |
| · | • |
| Section to be changed | Section 10.1 Spirometry: Bronchodilator Washout |
| | Recommendations |
| Description of change | The title of table was amended to clarify that the washout |
| _ compain or change | timeframes presented were <b>minimal</b> timeframes |
| Rationale for change | Washout timeframes for bronchodilators before spirometry |
| Tadonale for change | may be longer than those presented in the table. |
| | may be longer than those presented in the table. |
| Section to be changed | Section 10.2.4 Patient's Global Impression of Severity |
| Section to be changed | <u> </u> |
| Description of shares | (PGIS) for Cough, Shortness of Breath, and Fatigue |
| Description of change | Addition of the questionnaire on fatigue severity |
| Rationale for change | See change to Section 5.1.5.3 |
| Section to be changed | Section 10.6 Eligibility confirmation of IPF diagnosis |
| Description of change | Eligibilty criteria for patients with an "alternative diagnosis" |
| | HRCT finding were clarified with the following: |
| | If the HRCT findings are "suggestive of an alternative |
| | diagnosis", the clinical diagnosis of IPF may be |

c39145241-04 Clinical Trial Protocol 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | confirmed locally by (historical) surgical lung biopsy or TBLC demonstrating a "UIP" histopathology pattern. [] Patients clinically suspected to have IPF with an HRCT pattern "suggestive of an alternative diagnosis" require historical (i.e., not taken for the purpose of this trial) surgical lung biopsy or TBLC which will be reviewed locally (by the investigator/local histopathologist). In these patients, specific combinations of HRCT patterns and histopathology patterns may still allow a diagnosis of IPF based on the 2022 ATS/ERS/JRS/ALAT Guideline, i.e., an HRCT pattern of "alternative diagnosis" in combination with a surgical lung biopsy or TBLC with a histopathology pattern of "UIP" could qualify for inclusion. |
|---|---|
| Rationale for change | Patients with an "alternative diagnosis" HRCT finding are considered for eligibility (also see Section 3.3.1). |
| Section to be changed | Section 10.7 Trial participant feedback |
| Description of change | This new section describes the conditions of implementation of the optional participant and caregiver feedback questionnaires. |
| Rationale for change | To identify where improvements can be made in the clinical trial process, the sponsor wants to collect the participants' and caregivers' feedback on their clinical trial experience. |
| Section to be changed | Throughout the CTP |
| Description of change | Typographical errors and minor formatting issues amended |
| Rationale for change | To increase readability |

#### 11.3 GLOBAL AMENDMENT 3

| Date of amendment | 20 September 2023 | |
|---|---|---|
| EudraCT number | 2022-001091-34 | |
| BI Trial number | 1305-0014 | |
| BI Investigational | BI 1015550 | |
| Medicinal Product | | |
| Title of protocol | evaluating the efficacy and | A double blind, randomized, placebo-controlled trial evaluating the efficacy and safety of BI 1015550 over at least 52 weeks in patients with Idiopathic Pulmonary Fibrosis (IPF) |
| Global Amendment due | to urgent safety reasons | |
| Global Amendment (sub | stantial changes) | X |
| Section to be changed | Synopsis | |


| Description of change | A paragraph was deleted, and a new paragraph added to the |
|---|---|
| Description of change | statistical methods: |
| | statistical methods. |
| | An interim analysis for a potentially earlier regulatory |
| | submission may be conducted approximately 52 weeks after |
| | 450 patients (150 patients per arm) have started treatment |
| | and 26 weeks after the last patient has started treatment in |
| | order to detect early signs of substantial efficacy. The |
| | interim analysis will be implemented within a group |
| | sequential design with the aim to decide whether or not |
| | efficacy of BI 1015550 can be claimed early on in a |
| | confirmatory manner. Once the last randomized patient |
| | completes the Week-52 assessment, the main analysis of |
| | the trial will be carried out by the sponsor, who will be unblinded to assess the benefit-risk of the two doses of |
| | BI 1015550 compared with placebo. Patients will remain |
| | on their randomized blinded treatment until the sponsor |
| | has reviewed the efficacy and safety data from the main |
| | analysis and communicated the end of the trial. Once |
| | this trial ends, a final analysis based on all data will be |
| | carried out. |
| Rationale for change | 1) To reflect that the efficacy interim analysis will not be |
| | conducted, which was decided by the sponsor before the |
| | futility analysis. The sponsor's decision was based on |
| | Health Authority feedback and shifting trial timelines with fast recruitment, which make the time advantage in |
| | conducting the interim analysis limited |
| | 2) To specify the main analysis and the final analysis |
| | - |
| Section to be changed | Flow chart |
| Description of change | The following footnotes were revised: |
| | (1) Following completion of V10 patients will continue to |
| | have study visits every 12 weeks until <b>the start of EoT</b> |
| | visits is announced. The global study will be completed |
| | after all patients have performed the EoT visit and the |
| | EoS visit (if not continuing in the separate extension |
| | trial)the last patient randomized has reached Week 52. If |
| | the patient will complete EOT at 52 weeks (study |
| | completion phase), V10 is replaced by the EOT visit. |
| | (8) Assisted home spirometry will be offered at selected |
| | centres where every patient should have a training and |
| | measurement with the device <b>ideally</b> at Visits 2 or 3. <b>If the</b> |
| | requirement to use the iSpiro appears later in the trial, |
| | then this timepoint can be shifted. Remote measurement |


| | can be performed as per investigator's judgement but |
|---|---|
| | should not replace the on-site FVC measurement. |
| Rationale for change | 1) Clarification 2) To allow flexibility in training of iSpiro |
| Section to be changed | Section 3.1 Overall trial design |
| Description of change | The following paragraphs were added or revised: |
| | The main analysis of this study will be performed once the last randomized patient reaches the Week-52 visit (Visit 10 at the end of Part A). At that time, a first database lock (DBL1; Figure 3.1: 1) will occur and all data will be unblinded to the sponsor. Efficacy and safety analyses will be performed on the data from Part A of the trial to assess the benefit-risk of BI 1015550 over 52 weeks. In addition, data collected in Part B of the trial (after 52 weeks) and available at the time of data cut-off for the main analysis will be reported together with data from Part A (i.e. over the whole trial). |
| | Trial 1305-0014 Part B, will continue until all patients have completed the EOT visit and the EOS visit as applicable. A final database lock (DBL2; Figure 3.1: 1) will then occur and a final analysis based on the data over the whole trial will be carried out. |
| | Depending on the results of the evaluation based on DBL1 and determination of the BI 1015550 dose with the more favorable benefit-risk profile, patients receiving trial medication until the end of Part B will be eligible for open-label treatment with BI 1015550 in a separate extension trial. |
| | Around the time the last randomized patient reaches 52 weeks of treatment, After review of the efficacy and safety data available at DBL1, the sponsor will communicate the end of the trial and all patients still on blinded study treatment will perform an End of Treatment (EOT) visit and an End of Study (EOS) visit if applicable. The trial ends when all patients complete these visits. Details on follow-up and rollover to the extension trial are given in Section 6.2.3. |
| | "Figure 3.1: 1 Trial design overview at patient level (upper panel) and trial level (lower panel)" was updated according to the revised text. |
| Rationale for change | To specify the main analysis and the final analysis |

| Section to be changed | Section 3.2 Discussion of trial design, including the choice |
|---|---|
| _ | of control group(s) |
| Description of change | The following sentences were added: |
| | The additional data collected while patients remain on blinded treatment beyond 52 weeks will provide supportive long-term efficacy and safety data on the effect of BI 1015550 in a controlled manner. Due to the varying length of follow-up in Part B of the trial, the efficacy analyses incorporating data from Part A and Part B will focus on time-to-event endpoints. |
| Rationale for change | To add the rationale on conducting Part B |
| | · |
| Section to be changed | Section 4.1.5.1 Blinding |
| Description of change | The following paragraphs were added or revised: |
| | At the main analysis database lock (DBL1; see Section 3.1), the sponsor will be unblinded to assess the benefitrisk of both doses of BI 1015550 vs placebo and select the dose with the more favorable benefit-risk profile for the open-label extension trial. Patients, investigators, and other site personnel will remain blinded to the randomized treatment assignment until the end of the trial. |
| | The trial medication is identified by a medication code number and packaging is identical. The color, size, and shape of the respective 9 mg and 18 mg BI 1015550 and the matching placebo tablets will be indistinguishable. The access to the randomization code will be kept restricted until its release for analysis at DBL1. Further details regarding the timepoint of unblinding the database for analysis is documented in the TSAP. |
| | The randomization codes will be provided to bioanalytics before the last patient completed the trial <b>DBL1</b> to exclude placebo or comparator samples from the PK analysis. Bioanalytics will not disclose the randomization code or the results of their measurements until the database lock <b>DBL1</b> . |
| | A dedicated database snapshot (not a partial DBL) will be generated prior to DBL1, after all patients have completed the last PK visit (i.e. Week-26 visit), to allow for development and refinement of the population PK model (for "fast-track" PK analysis). Details of the analysis will be defined in the PK/PD analysis plan. In addition, the data will be used for front-loading of descriptive analysis for PK. Only personnel involved in the population PK and descriptive analyses will be |


| | granted access to the unblinded PK data before DBL1, whereas the trial team and all other functions not involved in the population PK and PK descriptive analyses will remain blinded (details will be provided in a separate logistics and access plan). The analysis plan for the population PK analysis will be finalized and signed prior to this dedicated database snapshot. No formal interim report will be generated for the population PK analysis. The final PK and PK/PD analyses will be reported separately from the clinical |
|---|---|
| | trial report (CTR) after DBL1. The external DMC will review unblinded data upon request and for the futility interim analyses analysis as described in Section 7.2.8, and only under conditions that ensure that patients, investigators, everyone involved in trial conduct or analysis, and anyone with any other participation in this double-blind trial will remain blinded. |
| | In case the interim analyses result in the recommendation for a preliminary report preparation, a respective team ("shadow team") independent of the main trial team will be formed to conduct the necessary data cleaning, analysis, and reporting steps and ensure to maintain the blind and restrict access to the randomization codes from the main trial team. Details of data transfer, timelines and involved trial functions during this process will be described in a separate logistics plan which will also specify details on data access. |
| Rationale for change | 1) To explain that unblinding of the sponsor will occur at the main analysis (DBL1); 2) To add that to front-load, personnel involved in the PK analyses will use unblinded PK data before DBL1; 3) To reflect that the efficacy interim analysis will not be conducted |
| Section to be changed | Section 4.2.2.1 Restrictions regarding concomitant |
| Description of change | treatment The following sentence was revised: |
| Description of change | Treatment with non-selective PDE inhibitors as well as PDE1, PDE3, PDE4, and PDE10 inhibitors is not allowed. "Table 4.2.2.1: 1 Restrictions regarding concomitant treatment" was updated according to the revised text. |
| Rationale for change | To narrow restricted PDE inhibitors down to those that specifically interfere with PDE4 |


| Section to be changed | Section 5.1.1 FVC |
|---|---|
| <b>Description of change</b> | The following sentence was revised: |
| | Training of the patients on the use of the iSpiro device and |
| | App should can be done at any visit, ideally at Visit 2 or |
| | Visit 3 together with a first recording. |
| Rationale for change | To allow flexibility in training of iSpiro |
| Turionale for enange | To wife it from the first |
| Section to be changed | Section 5.2.6.1.1 Adverse event |
| Description of change | The following paragraph was added: |
| | Adverse event report for depression and anxiety |
| | AE reporting based on the Hospital Anxiety and Depression Scale (HADS): new onset of moderate depression, defined as HADS subscore of >10, has to be reported as AE; new onset of moderate anxiety, defined as HADS subscore of >10, has to be reported as AE. HADS subscore of ≤10 should only be reported as an AE if clinically relevant. See Section 5.2.6.1.4 for reporting of AESI based on HADS. |
| Rationale for change | To clarify AE reporting based on HADS |
| 8 | |
| Section to be changed | Section 6.2.2.3 End of treatment visit |
| Description of change | The following sentence was revised: |
| | As described in Section 3.1, around the time the last randomized patient reaches 52 weeks of treatment (Visit 10) after the confirmation of the benefit-risk evaluation for a potential start of the extension trial based on the main analysis, all patients still on blinded study treatment will perform an EOT visit. It will occur either at the regular timepoint of Visit 10 (52 weeks) if it falls within this timeframe (e.g. if patient is still in Treatment Period A) or at a convenient timepoint in this timeframe if the patient already had performed Visit 10 previously (e.g. if the patient had already started Treatment Period B). |
| | The start of these EOT visits will be communicated when the last patient is randomized and thus, the timepoint of the anticipated last patient at 52 weeks visit is known. |
| Rationale for change | Clarification |
| Section to be changed | Section 7.1 Null and alternative hypotheses |
| <b>Description of change</b> | A paragraph was added: |

| | The hypothesis testing of the key secondary endpoint is based on data collected up to the main analysis (all data up to DBL1; see Figure 3.1: 1). A supplementary analysis of the key secondary endpoint using all data collected over the whole trial will be performed after DBL2. The following sentence was deleted: The tests for the primary endpoint comparing each dose vs. placebo within the graphical testing procedure will include one interim analysis for potential efficacy claim using a group sequential design. The alpha level at interim analysis and final analysis will be adjusted accordingly, see Section 7.2.8: |
|---|---|
| Rationale for change | 1) To clarify that the hypothesis testing of the key secondary endpoint will be done at the main analysis; 2) To reflect that the efficacy interim analysis will not be conducted |
| Section to be changed | Section 7.2.1 General considerations |
| Description of change | A paragraph was added: |
| | All planned efficacy and safety analyses, including for the primary and key secondary endpoints will be carried out at DBL1 (Figure 3.1: 1) and the statistical hypotheses described in Section 7.1 will be tested. After DBL2, analyses of the efficacy endpoints defined as "over the duration of the trial" and all safety analyses will be repeated to include all data collected until the end of the trial. |
| Rationale for change | To describe at a high level what will be analyzed at the |
| | main and the final analysis |
| Section to be changed | Section 7.2.3.3 Supplementary Analyses |
| Description of change | The following sentence was revised: |
| | Further details will be specified in the TSAPNot applicable for this trial. |
| Rationale for change | Clarification |
| Section to be changed | Section 7.2.8 Interim analyses |
| Description of change | The following paragraphs were deleted: |
| | To allow for the early initiation of marketing authorization applications in the case of a positive efficacy finding combined with a favorable safety profile which are |

c39145241-04

**Clinical Trial Protocol** 


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

considered sufficient to conclude for a clearly positive benefit-risk balance, an interim analysis for efficacy may be performed by the DMC. This interim analysis will be implemented within a group sequential design with the aim to decide whether or not efficacy of BI 1015550 can be claimed early on in a confirmatory manner. This interim analysis may be conducted approximately 52 weeks after 450 patients (150 patients per arm) have started treatment and 26 weeks after the last patient has started treatment. A Wang-Tsiatis type alpha spending approach [R06-0638] with a delta parameter of 0.25 will be used for the tests H 01 and H 02 of the primary endpoint comparing the 18 mg bid and 9 mg bid dose vs. placebo, respectively. It is expected that at the time of the interim analysis around 70% of the events for the key secondary endpoint have been observed. The graphical testing procedure as defined in Section 7.1 will be followed with an extension to group sequential designs [R17-2947]. The secondary endpoint will not be tested at this interim analysis for either of the doses and all alpha propagated to secondary endpoint will be reserved for the final analysis as the trial will not be stopped.

In order to conclude that the trial met its primary endpoint for at least one dose, the following criteria must be met: The p-value for the primary endpoint meets the required cut-offs for one dose based on the Wang-Tsiatis type alpha spending approach with a delta parameter of 0.25, e.g. for an interim at approximately 450 patients complete 52 week follow-up, planned at two-sided,  $\alpha_{ia}=0.0103$  for H\_01 or  $\alpha_{ia}=0.0016$  for H\_02.

If the interim analysis meets the primary endpoint, the DMC will take into account the totality of the data for the recommendation to the sponsor to unblind the trial by a team independent of the trial team with the task to prepare regulatory submission documents.

The interim analysis is expected to occur approximately 6 months before the final analysis. Independent of the results the patients will be followed up until the planned End of Study.

The trial team, patients and investigators will remain blinded until the final data base lock. All measures taken will be directed to maintain the trial integrity. Details regarding the safeguards to keep patients, investigators and the trial team blinded will be provided in a logistics plan (Section 4.1.5).


| D di l C l | T 0 44 44 00 14 1 11 41 |
|---|---|
| Rationale for change | To reflect that the efficacy interim analysis will not be |
| | conducted |
| Section to be changed | Section 7.3.1 Efficacy endpoints |
| Description of change | The following table reference was corrected: |
| | In the primary analysis of primary endpoint, missing data will not be imputed except for death, where a poor outcome will be assigned, see <b>Table 7.3.1:</b> 1-Table 7.5: 1. |
| Rationale for change | Correction |
| Section to be changed | Section 7.5 Determination of sample size |
| Description of change | The following paragraphs were revised: |
| | An effective sample size of 310 patients per group, will detect a treatment effect of 74 mL with 9091% power under two-stage group sequential design with Wang-Tsiatis alpha spending function (delta=0.25) and cumulative two-sided alpha of 5% for one active BI 1015550 dose arm vs. placebo. With 310 patients per arm and a two-sided type I error rate of 0.05, a treatment effect size of 90, 65, 55, and 45 can be detected for each of the primary endpoint with 98%, 8182%, 6769%, and 5052% power respectively. |
| | Simulation results as presented in Table 7.5: 2 suggest that with 310 effective sample size per arm, there is at least 93% power to detect an effect size of 74 mL in FVC change from baseline at Week 52 for at least one dose is significant (Scenario #1). Regardless of effect size of the 9 mg bid arm, probability of detecting a significant FVC effect of 74 mL in the 18 mg bid arm is between 8889% to 90%. Furthermore, if 18 mg bid arm has an effect of 74 mL in primary endpoint and HR of 0.6 in key secondary endpoint, the probability of rejecting both H_01 and H_03 is between 65% to 74% depending on relative effect size of the 9 mg bid arm. The simulation results also show a well controlled type-I error under the null hypothesis (Scenario #5) with the proposed testing strategy. |
| | "Table 7.5: 2 Multiplicity adjusted probabilities of success for each hypothesis,— and positive study and interim success under different scenarios of effect sizes from simulations" was revised to update the numbers without the efficacy interim analysis, to delete 5 lines with "probability of rejecting at least one dose primary endpoint at interim", and to delete a footnote "Multiplicity adjusted for interim |

## Boehringer Ingelheim BI Trial No.: 1305-0014

c39145241-04 Clinical Trial Protocol


| T | |
|---|---|
| | analysis using group sequential design with Wang-Tsiatis |
| | alpha spending function (delta = 0.25).". |
| Rationale for change | To reflect that the efficacy interim analysis will not be |
| | conducted |
| Section to be changed | Appendix 10.4.3 Restricted PDE inhibitors |
| Description of change | The table was revised to delete the lines of the following |
| | PDE inhibitors: |
| | PDE1 |
| | Vinpocetine (Cavinton) |
| | PDE3 |
| | Cilostazol (Pletal, Ekistol) |
| | Olprinone (Coretec) |
| | Anagrelide (also inhibits phospholipase A2) (Agrylin, |
| | Xagrid) |
| | PDE10A |
| | Papaverine (Pavabid, Pavagen) |
| Rationale for change | To narrow restricted PDE inhibitors down to those that |
| | specifically interfere with PDE4 |



#### APPROVAL / SIGNATURE PAGE

Document Number: c39145241 Technical Version Number: 4.0

**Document Name:** clinical-trial-protocol-1305-0014-version-04

**Title:** A double blind, randomized, placebo-controlled trial evaluating the efficacy and safety of BI 1015550 over at least 52 weeks in patients with Idiopathic Pulmonary Fibrosis (IPF)

### **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval-Clinical Program | | 21 Sep 2023 13:29 CEST |
| Approval-Biostatistics | | 21 Sep 2023 13:29 CEST |
| Approval-Clinical Trial Leader | | 21 Sep 2023 15:20 CEST |
| Verification-Paper Signature<br>Completion | | 25 Sep 2023 11:31 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c39145241Technical Version Number: 4.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|